#### Protocol for

# Official Title of Study

A PHASE 3, MULTICENTER, OPEN-LABEL,
RANDOMIZED STUDY TO EVALUATE THE EFFICACY
AND SAFETY OF FEDRATINIB COMPARED TO BEST
AVAILABLE THERAPY IN SUBJECTS WITH DIPSSINTERMEDIATE
OR HIGH-RISK PRIMARY
MYELOFIBROSIS, POST-POLYCYTHEMIA VERA
MYELOFIBROSIS, OR POST-ESSENTIAL
THROMBOCYTHEMIA MYELOFIBROSIS AND
PREVIOUSLY TREATED WITH RUXOLITINIB
NCT03952039

April 23, 2021

# A PHASE 3, MULTICENTER, OPEN-LABEL, RANDOMIZED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF FEDRATINIB COMPARED TO BEST AVAILABLE THERAPY IN SUBJECTS WITH DIPSSINTERMEDIATE OR HIGH-RISK PRIMARY MYELOFIBROSIS, POST-POLYCYTHEMIA VERA MYELOFIBROSIS, OR POST-ESSENTIAL THROMBOCYTHEMIA MYELOFIBROSIS AND PREVIOUSLY TREATED WITH RUXOLITINIB

#### The "FREEDOM 2" trial

 PROTOCOL NUMBER:
 FEDR-MF-002

 DATE FINAL:
 26-Sep-2018

 AMENDMENT No. 1 DATE:
 01-Feb-2019

 AMENDMENT No. 2 DATE:
 08 Oct 2019

 AMENDMENT No. 3 DATE:
 15 Jan 2021

 AMENDMENT No. 4 DATE:
 23 Apr 2021

 EudraCT NUMBER:
 2018-003411-21

IND NUMBER: 078286

**SPONSOR NAME/ ADDRESS:** Impact Biomedicines, Inc., a Wholly Owned

Subsidiary of Celgene Corporation (hereafter

referred to as Celgene-Impact)

#### **CONFIDENTIAL**

This protocol is provided to you as an Investigator, potential Investigator, or consultant for review by you, your staff, and ethics committee/institutional review board. The information contained in this document is regarded as confidential and, except to the extent necessary to obtain informed consent, may not be disclosed to another party unless such disclosure is required by law or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# MEDICAL MONITOR / EMERGENCY CONTACT INFORMATION

| Contact Information: |
|----------------------|
| Name: |
| Title: |
| Address: |
| Phone: |
| E-mail: |

Note: The back-up 24-hour global emergency contact call center should only be used if you are not able to reach the Clinical Research Physician(s) or Medical Monitor or designee for emergency calls.

# CELGENE THERAPEUTIC AREA HEAD SIGNATURE PAGE

| See appended electronic signature page | |
|--------------------------------------------|-------------|
| Signature of Celgene Therapeutic Area Head | dd mmm yyyy |

Printed Name of Celgene Therapeutic Area Head and Title

By my signature, I indicate I have reviewed this protocol and find its content to be acceptable.

# SITE PRINCIPAL INVESTIGATOR SIGNATURE PAGE

| Signature of Site Principal Investigator | dd mmm yyyy |
|---|---|
| Printed Name of Site Principal Investigator | |
| Institution Name: | |
| By my signature, I agree to personally supervise the conduct of the site and to ensure its conduct is in compliance with the protocol, Institutional Review Board (IRB)/Ethics Committee (EC) proced Celgene-Impact representatives, the Declaration of Helsinki, Intel Harmonisation (ICH) Good Clinical Practices Guidelines, and longoverning the conduct of clinical studies. | informed consent,<br>dures, instructions from<br>ernational Council for |

# COORDINATING PRINCIPAL INVESTIGATOR SIGNATURE PAGE

| Signature of Coordinating Principal Investigator | dd mmm yyyy |
|---|---|
| Printed Name of Coordinating Principal Investigator | |
| Institution Name: | |
| By my signature, I agree the protocol has been written to comply with ICH Good Clinical Practices guidelines and agree to offer guidance throughout the study as needed. | |

# PROTOCOL SUMMARY

#### **Study Title**

A Phase 3, multicenter, open-label, randomized study to evaluate the efficacy and safety of fedratinib compared to best available therapy (BAT) in subjects with DIPSS (Dynamic International Prognostic Scoring System)-intermediate or high-risk primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (post-PV MF), or post-essential thrombocythemia myelofibrosis (post-ET MF) and previously treated with ruxolitinib.

# **Objectives**

The primary objective of the study is to evaluate the percentage of subjects with at least 35% spleen volume reduction in the fedratinib and the BAT arms.

The secondary objectives are:

- To evaluate the percentage of subjects with at least 50% reduction in myelofibrosis (MF)-associated symptoms as measured by the Myelofibrosis Symptom Assessment Form (MFSAF)
- To evaluate the percentage of subjects with at least 25% spleen volume reduction (SVR)
- To evaluate the safety of fedratinib
- To evaluate the reduction of spleen size by palpation
- To evaluate durability of spleen response by magnetic resonance imaging (MRI) / computed tomography (CT) and by palpation
- To evaluate the durability of symptoms response
- To evaluate spleen and disease progression free survival
- To assess the effectiveness of the risk mitigation strategy for gastrointestinal events and Encephalopathy, including Wernicke's
- To evaluate Health-Related Quality of Life (HRQoL) as measured by the European Organization for Research and Treatment of Cancer Quality of Life C30 (EORTC QLQ-C30)
- To evaluate Patient-Reported Outcomes (PRO) as measured by the EQ-5D-5L questionnaire
- To evaluate Overall Survival (OS)





# Study Population and Design

This Phase 3, multicenter, randomized, two-arm, open-label study will include subjects with intermediate-2 or high-risk (as per the DIPSS score) primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (post-PV MF), or post-essential thrombocythemia myelofibrosis (post-ET MF). This study will be conducted in compliance with International Council for Harmonisation (ICH) Good Clinical Practices (GCPs).

Study design includes:

- A 28-day Screening Period
- 2:1 Randomization to fedratinib or best available therapy (BAT)
- Stratification at Randomization according to:
  - Spleen size by palpation: < 15 cm below left costal margin (LCM) versus ≥ 15 cm below LCM
  - Platelets  $\geq 50$  to  $\leq 100 \times 10^9/L$  versus platelets  $\geq 100 \times 10^9/L$
  - Refractory or relapsed to ruxolitinib treatment versus intolerance to ruxolitinib treatment
- Study Treatment Period (time on study drug plus 30 days after last dose)
- Subjects are allowed to crossover from BAT to the fedratinib arm after the Cycle 6 response assessment or before the Cycle 6 response assessment in the event of a confirmed progression of splenomegaly by MRI/CT scan
- A Survival Follow-up Period for progression and survival

Refer to the eligibility criteria below for more information.

#### Length of Study

The expected duration of entire study is approximately 5 years, which includes approximately 24 months to fully enroll, and at least 36 months for treatment and follow-up. The actual duration of the trial will be dependent upon the median treatment duration for subjects.

The End of Trial is defined as the date of the last visit of the last subject to complete the Survival Follow-up or the date of receipt of the last data point from the last subject that is required for primary, secondary analysis, as prespecified in the protocol, whichever is the later date. End of trial is expected approximately 3 years after the last subject is randomized. Refer to Section 3.3 for more information.

#### **Study Treatments**

Subjects satisfying the eligibility criteria will be randomized 2:1 to one of these two arms:

- Arm 1 (Fedratinib) will include up to 128 subjects receiving fedratinib 400 mg
   OR
- Arm 2 (BAT) will include up to 64 subjects receiving best available therapy

Fedratinib will be orally self-administered on an outpatient basis, once daily preferably together with food during an evening meal at the same time each day in consecutive 4-week (28-day) cycles. Fedratinib may be taken with or without regard to food.

The most common adverse events associated with fedratinib are hematological and gastrointestinal. Hematological adverse events associated with Janus kinase (JAK) inhibitors are dose dependent, mechanism-based and managed through dose reductions, dose interruptions and transfusions.

The fedratinib dose in this study is 400 mg/day. If a subject experiences a drug toxicity as specified in the Fedratinib Dose Modification Schedule table (Table 4), the dosing should be interrupted and the dose may need to be modified (Section 7).

If a subject does not tolerate fedratinib therapy after 2 dose level reductions from the starting dose, he/she must be withdrawn from the study treatment. If the toxicity does not resolve in the time period as specified in the Fedratinib Dose Modification Schedule table (Table 4), subjects must be withdrawn from the study treatment. Reescalation of doses is possible in certain cases as defined in the Fedratinib Dose Modification Schedule table (Table 4). The daily dose of fedratinib cannot exceed 400 mg/day.

Subjects may continue treatment with fedratinib or BAT until unacceptable toxicity, lack of therapeutic effect, progression of disease according to the IWG-MRT 2013 criteria or until a subject is not compliant with treatment or withdraws consent.

Best available therapy (BAT) regimen may include any Investigator-selected treatment. Investigational agents, fedratinib (if approved during the course of the study) and hematopoietic stem cell transplantation are not regarded to be BAT.

# **Overview of Key Efficacy Assessments**

# **Assessment of Spleen Size**

Spleen volume will be assessed at the study site (MRI or CT Scan if MRI is contraindicated) during screening and at the end of cycle 3, 6, 12, 18, 24, every sixth (6<sup>th</sup>) cycle after Cycle 24 and at End of Treatment Visit. MRI/CT scans will be reviewed centrally. The central review will be blinded for arm assignment and treatment.

Spleen size will also be assessed by palpation at screening and on Day 1 of each treatment cycle, at the End of Treatment visit and at the 30-day follow-up visit after last dose of study treatment.

# Assessment of MF-associated symptoms

The MF-related symptoms evaluation will be performed using the MFSAF version 4.0 using a 7-day recall period (Gwaltney, 2017).

# Overview of Key Safety Assessments

Safety of fedratinib is evaluated based on the incidence of treatment-emergent adverse events (TEAEs) and changes in clinical laboratory parameters, Eastern Cooperative Oncology Group (ECOG) Performance Status (PS), electrocardiogram (ECG), and vital signs.

Safety assessments will comprise:

- Record of adverse events (AEs) and serious adverse events (SAEs) at each study visit
- Physical examination including assessment of abnormal eye movements, cerebellar abnormalities, body weight
- Vital signs
- Cognitive assessment: Mini-Mental State Examination (MMSE)
- Laboratory assessments: hematology, serum chemistry, thiamine level, coagulation, urinalysis, serum/urine pregnancy tests
- Electrocardiogram (ECG)



# **Overview of Other Patient-Reported Outcomes**

The HRQoL/PRO evaluations will be performed using the following tools:

- HRQoL and its various domains will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life C30 (EORTC QLQ-C30) questionnaire version 3 (Aaronson, 1993).
- Health utilities will be assessed using EQ-5D-5L classifier for 5 levels. The
  instrument contains 5 items that assess mobility, self-care, usual activities,
  pain/discomfort, and anxiety/depression and a visual analog scale (VAS) for global
  health.



All HRQoL/PRO evaluations will be performed on an electronic tablet at the site on Day 1 of each treatment cycle, at the End of Treatment (EOT) and the 30-day follow-up visit after last dose of study treatment. All these QoL-related assessments should be performed before any other assessments are performed by the Investigator or designee during the visit.

# **TABLE OF CONTENTS**

| TITLE F | PAGE | 1 |
|---|---|---|
| PROTO | COL SUMMARY | 6 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Background | 18 |
| 1.1.1. | Myeloproliferative Neoplasm (MPN) Associated Myelofibrosis | 18 |
| 1.1.2. | Treatment Options for MPN-Associated Myelofibrosis | 19 |
| 1.1.3. | Approved Therapies | 19 |
| 1.1.4. | Medical Need | 20 |
| 1.2. | Fedratinib | 21 |
| 1.3. | Wernicke Encephalopathy (WE) in Patients Treated with Fedratinib | 23 |
| 1.4. | Rationale | 24 |
| 1.4.1. | Study Rationale and Purpose | 24 |
| 1.4.2. | Rationale for the Study Design | 24 |
| 1.4.3. | Rationale for Dose, Schedule and Regimen Selection | 25 |
| 1.4.4. | Rationale for Patient-Reported Outcomes | 26 |
| 1.4.5. | | 27 |
| 1.4.6. | | 27 |
| 2. | STUDY OBJECTIVES AND ENDPOINTS | 29 |
| 3. | OVERALL STUDY DESIGN | 34 |
| 3.1. | Study Design | 34 |
| 3.2. | Study Duration for Subjects | 35 |
| 3.3. | End of Trial | 36 |
| 4. | STUDY POPULATION | 37 |
| 4.1. | Number of Subjects | 37 |
| 4.2. | Inclusion Criteria | 37 |
| 4.3. | Exclusion Criteria | 39 |
| 5. | TABLE OF EVENTS | 41 |
| 6. | PROCEDURES | 44 |
| 6.1. | Screening Period. | 44 |
| 6.2. | Randomization of a Subject to the Study. | 48 |
| 6.3 | Treatment Period | 10 |

# Impact Biomedicines, Inc., a Wholly Owned Subsidiary of Celgene Corporation

| 6.3.1. | Symptoms Response Assessment using MFSAF version 4.0 | 50 |
|---|---|---|
| 6.3.2. | Health-related Quality of Life Assessments and Patient-Reported Outcomes | 51 |
| 6.3.2.1. | EORTC QLQ-C30 questionnaire | 51 |
| 6.3.2.2. | EQ-5D-5L | 51 |
| 6.3.2.3. | | 52 |
| 6.3.3. | | 53 |
| 6.4. | Response Assessment | 54 |
| 6.5. | Crossover | 54 |
| 6.6. | End of Treatment Visit | 55 |
| 6.7. | 30-Day Follow-up After Last Dose Visit | 57 |
| 6.8. | Survival Follow-up | 57 |
| 6.9. | Unscheduled Assessments or Visits | 58 |
| 7. | DESCRIPTION OF STUDY TREATMENT | 59 |
| 7.1. | Description of Investigational Product | 59 |
| 7.2. | Best Available Therapy Regimens | 59 |
| 7.3. | Treatment Administration and Schedule | 59 |
| 7.3.1. | Dose Modification for Toxicity | 59 |
| 7.3.2. | Dose Adjustment for Co-administration of Fedratinib with Strong CYP3A4 Inhibitors | 62 |
| 7.3.3. | Dose Adjustment for Renal Impairment | 63 |
| 7.4. | Overview on Management of Gastrointestinal Adverse Events | 63 |
| 7.4.1. | Management of Nausea and Vomiting | 63 |
| 7.4.2. | Management of Diarrhea | 64 |
| 7.5. | Management of Encephalopathy, including Wernicke's | 64 |
| 7.5.1. | Clinical and Cognitive Assessment | 64 |
| 7.5.2. | Management of Encephalopathy, including Wernicke's | 65 |
| 7.5.3. | Thiamine, Supplementation, Monitoring and Correction | 65 |
| 7.6. | Method of Treatment Assignment | 66 |
| 7.7. | Packaging and Labeling | 66 |
| 7.8. | Investigational Product Accountability and Disposal | 67 |
| 7.9. | Investigational Product Compliance | 67 |
| 8. | CONCOMITANT MEDICATIONS AND PROCEDURES | 68 |
| 8.1. | Permitted Concomitant Medications and Procedures | 68 |

# Impact Biomedicines, Inc., a Wholly Owned Subsidiary of Celgene Corporation

| 8.2. | Prohibited Concomitant Medications | 69 |
|---|---|---|
| 8.3. | Clinically Relevant Cytochrome P450 Inducers, Inhibitors, Substrates, and | |
| 0 | Transporter Substrates | |
| 9. | STATISTICAL CONSIDERATIONS | |
| 9.1. | Overview | |
| 9.2. | Study Population Definitions | 71 |
| 9.3. | Sample Size Consideration | |
| 9.4. | Background and Demographic Characteristics | 73 |
| 9.4.1. | Demographic and Baseline Characteristics. | 73 |
| 9.4.2. | Prior or Concomitant Medications | 73 |
| 9.5. | Subject Disposition | 73 |
| 9.6. | Extent of Study Treatment Exposure and Compliance | 73 |
| 9.7. | Efficacy Analysis | 74 |
| 9.7.1. | Spleen Volume Response Rate (35%) by MRI / CT (RR) | 74 |
| 9.7.2. | Symptom Response Rate (SRR) | 74 |
| 9.7.3. | Spleen Volume Response Rate (25%) by MRI / CT (RR25) | 75 |
| 9.7.4. | Spleen Response Rate by Palpation (RRP) | 75 |
| 9.7.5. | Durability of Spleen Volume Response by MRI/CT (DR) | 75 |
| 9.7.6. | Spleen and Disease Progression Free Survival (SDPFS) | 76 |
| 9.7.7. | Durability of Spleen Response by Palpation (DRP) | 76 |
| 9.7.8. | Overall Survival | 76 |
| 9.7.9. | Crossover Efficacy Analysis | 76 |
| 9.8. | Safety Analysis | 77 |
| 9.8.1. | Adverse Events | 77 |
| 9.8.2. | Assessment of Risk Mitigation Strategy for Gastrointestinal Adverse Events and Encephalopathy, including Wernicke's | 77 |
| 9.8.3. | Laboratory Results | 77 |
| 9.8.4. | Electrocardiograms | 78 |
| 9.8.5. | Vital Signs | 78 |
| 9.9. | Patient-reported Outcomes / Health Economics | 78 |
| 9.9.1. | Symptoms Response Assessment Using MFSAF V.4.0 | 78 |
| 9.9.2. | EORTC QLQ-C30 Version 3.0 | |
| 9.9.3. | EO-5D-5L | 79 |

| 9.10. | | 79 |
|---------|-------------------------------------------------------|----|
| 9.11. | Interim Analysis | 80 |
| 9.12. | Other Topics | 80 |
| 9.12.1. | Steering Committee | 80 |
| 10. | ADVERSE EVENTS | 81 |
| 10.1. | Monitoring, Recording and Reporting of Adverse Events | 81 |
| 10.2. | Evaluation of Adverse Events | 82 |
| 10.2.1. | Seriousness | 82 |
| 10.2.2. | Severity/Intensity | 83 |
| 10.2.3. | Causality | 84 |
| 10.2.4. | Duration | 84 |
| 10.2.5. | Action Taken | 84 |
| 10.2.6. | Outcome | 84 |
| 10.3. | Abnormal Laboratory Values | 84 |
| 10.4. | Pregnancy | 85 |
| 10.4.1. | Females of Childbearing Potential: | 85 |
| 10.4.2. | Male Subjects | 86 |
| 10.5. | Reporting of Serious Adverse Events | 86 |
| 10.5.1. | Safety Queries | 86 |
| 10.6. | Expedited Reporting of Adverse Events | 86 |
| 10.7. | Adverse Events of Special Interest | 87 |
| 11. | DISCONTINUATIONS | 89 |
| 11.1. | Treatment Discontinuation. | 89 |
| 11.2. | Study Discontinuation | 89 |
| 12. | EMERGENCY PROCEDURES | 90 |
| 12.1. | Emergency Contact | 90 |
| 12.2. | Emergency Identification of Investigational Products | 90 |
| 13. | REGULATORY CONSIDERATIONS | 91 |
| 13.1. | Good Clinical Practice | 91 |
| 13.2. | Investigator Responsibilities | 91 |
| 13.3. | Subject Information and Informed Consent | 92 |
| 13.4. | Confidentiality | 92 |
| 13.5. | Protocol Amendments | 92 |

| 13.6. Institutional Review Board/Independent Ethics Committee Review and Approval | 92 |
|---|---|
| 13.7. Ongoing Information for Institutional Review Board/ Ethics Committee | |
| 13.8. Termination of the Study | 93 |
| 14. DATA HANDLING AND RECORDKEEPING | 94 |
| 14.1. Data/Documents | 94 |
| 14.2. Data Management | |
| 14.3. Record Retention | |
| 15. QUALITY CONTROL AND QUALITY ASSURANCE | 96 |
| 15.1. Study Monitoring and Source Data Verification | |
| 15.2. Audits and Inspections | |
| 15.3. Product Quality Complaint | 96 |
| 16. PUBLICATIONS | 98 |
| 17. REFERENCES | 99 |
| 18. APPENDICES | 105 |
| APPENDIX A. TABLE OF ABBREVIATIONS AND SPECIAL TERMS | 105 |
| APPENDIX B. MYELOFIBROSIS SYMPTOM ASSESSMENT FORM (MFSAF) VERSION 4.0 | 109 |
| APPENDIX C. QUALITY OF LIFE ASSESSMENT: EORTC QLQ-C30 QUESTIONNAIRE | 110 |
| APPENDIX D. PATIENT-REPORTED OUTCOMES: EQ-5D-5L QUESTIONNAIRE | 112 |
| APPENDIX E. NATIONAL CANCER INSTITUTE (NCI) COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (CTCAE) | |
| VERSION 5.0 | 114 |
| APPENDIX F. DYNAMIC INTERNATIONAL PROGNOSTIC SCORING SYSTEM (DIPSS) | 115 |
| APPENDIX G. IWG-MRT: INTERNATIONAL WORKING GROUP-<br>MYELOPROLIFERATIVE NEOPLASMS RESEARCH AND<br>TREATMENT (IWG-MRT) | 116 |
| APPENDIX H. 2016 WORLD HEALTH ORGANIZATION (WHO) DIAGNOSTIC CRITERIA FOR PRIMARY MYELOFIBROSIS (PMF) | 117 |
| APPENDIX I. PROPOSED CRITERIA FOR THE DIAGNOSIS OF POST-POLYCYTHEMIA VERA AND POST-ESSENTIAL THROMBOCYTHEMIA MYELOFIBROSIS | 110 |
| APPENDIX J. ECOG PERFORMANCE STATUS SCALE | |

| Fedratinib Protocol FEDR-MF-002 | Impact Biomedicines, Inc., a Wholly Owned Subsidiary of Celgene Corporation |
|---|---|
| | THE GLOMERULAR FILTRATION RATE BY121 |
| | EVANT P450 INDUCERS, INHIBITORS, ANSPORTER SUBSTRATES |
| | T ASSOCIATION CLASSIFICATION FOR<br>AILURE |
| | 125 |
| INTERNATIONAL WOR<br>NEOPLASMS RESEARC | SE CRITERIA FOR MYELOFIBROSIS: KING GROUP-MYELOPROLIFERATIVE H AND TREATMENT (IWG-MRT) AND NET (ELN) CONSENSUS REPORT (2013)126 |
| APPENDIX P. MINI-MENTAL STA | ATE EXAMINATION-2 |

# LIST OF TABLES

| Table 1: | Study Objectives | 29 |
|----------|------------------------------------------|----|
| Table 2: | Study Endpoints | 3 |
| Table 3: | Table of Events | 4 |
| Table 4: | Fedratinib Dose Modification Schedule | 6 |
| Table 5: | PCSA Criteria for Vital Signs and Weight | 78 |

| Fedratinib |
|----------------------|
| Protocol FEDR-MF-002 |

| | Impact Biomedicines | s, Inc., |
|-----------------------|-----------------------|----------|
| a Wholly Owned Subsid | iary of Celgene Corpo | ration |

# LIST OF FIGURES

#### 1. INTRODUCTION

# 1.1. Disease Background

# 1.1.1. Myeloproliferative Neoplasm (MPN) Associated Myelofibrosis

Myeloproliferative neoplasm-associated myelofibrosis (MF) is a serious and life-threatening disease that can present as a de novo or primary myelofibrosis (PMF) or evolve from previous polycythemia vera (post PV-MF) or essential thrombocythemia (post ET-MF) (Swerdlow, 2008). The disease is characterized by clonal myeloproliferation, ineffective erythropoiesis, bone marrow stromal changes, hepatosplenic extramedullary hematopoiesis, and aberrant cytokine expression (Tefferi, 2011). Patients typically present with splenomegaly, constitutional symptoms, moderate to severe anemia, thrombocytopenia, and leukocytosis.

Primary myelofibrosis is a member of a group of Philadelphia chromosome (Ph1)-negative myeloproliferative neoplasms (MPN) which also includes PV and ET (Tefferi, 2007). Almost all patients with PV and about one-half of patients with ET and PMF have a Janus Kinase 2 (JAK2) mutation, typically JAK2V617F. Other mutations in patients with PMF include calreticulin (CALR) and myeloproliferative leukemia virus (MPL). About 20% of patients with PMF have no detectable mutation in JAK2, CALR, or MPL and are termed triple negative (Levine, 2005; Wernig, 2006). Mutations in JAK2, CALR, and MPL result in activation of the JAK/STAT signaling pathway resulting in cell proliferation and inhibiting cell death. The result is clonal expansion (Ihle, 2007). Thus, a JAK2 inhibitor that can down regulate the JAK/STAT pathway is expected to be helpful in reducing cell proliferation.

Polycythemia vera (PV) and essential thrombocythemia (ET) are characterized by increased levels of red blood cells (RBCs) and platelets. However, about 10% of affected patients develop bone marrow fibrosis morphologically indistinguishable from PMF. These conditions are termed post-PV-MF and post-ET-MF (Campbell, 2005), and are clinically named MPN-associated myelofibrosis. Patients with MPN-associated myelofibrosis have similar survival prognoses to that of the PMF and about a 10% cumulative risk of transformation to acute myeloid leukemia (AML).

There are several prognostic scoring systems predicting survival of patients with PMF. The International Prognostic Scoring System (IPSS) is used to predict survival at diagnosis and the Dynamic International Prognostic Scoring System (DIPSS) at any time in the disease course (Cervantes, 2009; Passamonti, 2010). Variables included in the IPSS are age > 65 years, constitutional symptoms, hemoglobin level < 10 g/dL, and white blood cell (WBC) counts. Additional recent prognostic scoring systems include the Dynamic International Prognostic Scoring System Plus (DIPSS Plus) and scoring systems incorporating data from mutation analyses. There is a strong association between overall survival for MF patients and the DIPSS risk category for patients with low, intermediate risk 1, intermediate risk 2, or high risk with median survival of 15.4, 6.5, 2.9, and 1.3 years, respectively (Tefferi, 2016).

Approximately 70% of individuals with MF are in the intermediate-2 or high-risk categories (Gangat, 2011), representing the greatest unmet medical need. Symptomatic enlargement of the spleen and liver, the necessity for RBC transfusions, cachexia, and the other MF-associated symptoms result in greatly compromised quality of life in these patients (Mesa, 2007).

# 1.1.2. Treatment Options for MPN-Associated Myelofibrosis

Allogeneic stem-cell transplantation (SCT) is currently the only treatment that can induce long-term remission in patients with MF. The average age at diagnosis of MF is 65 years; thus, the majority of patients are not eligible for SCT. Therefore, the treatment options are primarily symptom-oriented, to help mitigate the clinical presentation of anemia, splenomegaly, constitutional symptoms and less commonly increased levels of platelets, and WBCs. So far, none of these symptom-oriented treatments have shown an anti-clonal effect, although alleviation in spleen size and splenic discomfort, symptoms, and anemia have been shown (Vannucchi, 2017).

Fortunately, the understanding of MPNs and the molecular mechanisms of the disease have been expanding. In 2005, the JAK2V617F mutation was discovered and observed in approximately 50% to 60% of patients with PMF or ET and 90% to 95% of patients with PV. This discovery, along with the observation of other mutations in patients with MPNs found to activate the JAK/signal transducers and activators of transcription (STAT) pathway (JAK2 exon 12, myeloproliferative leukemia, and adaptor protein LNK) (Oh, 2010; Pikman, 2006; Scott, 2007), has established dysregulation of the JAK signaling pathway as the major contributor to the pathogenesis of MPNs. It has also translated into the development of small-molecule JAK inhibitors.

Until recently, the JAK1/2 inhibitor ruxolitinib was the only approved therapy for MF. On August 16th, 2019, fedratinib was approved by the United States (US) Food and Drug Administration (FDA) for the treatment of MF. Ruxolitinib is indicated for treatment of patients with intermediate or high-risk MPN-associated myelofibrosis (MF), including primary MF, postpolycythemia vera MF and post-essential thrombocythemia MF. The registration of ruxolitinib was based on 2 randomized, controlled studies (COMFORT-I and COMFORT-II) that compared ruxolitinib to placebo and to the best available therapy (BAT), respectively (Harrison, 2012; Verstovsek, 2012). The studies demonstrated benefit, with a higher proportion of subjects in the ruxolitinib arms exhibiting a  $\geq$  35% reduction in spleen volume as measured by magnetic resonance imaging (MRI) at 24 weeks in COMFORT-I (41.9% ruxolitinib versus 0.7% placebo) and at 48 weeks in COMFORT-II (28.5% ruxolitinib versus 0% BAT). In COMFORT-I, there was a > 50% improvement in the Myelofibrosis Symptom Assessment Form (MFSAF) Total Symptom Score (TSS) at 24 weeks in 45.9% of subjects on ruxolitinib compared with 5.3% of subjects on placebo. Improvement of survival in the ruxolitinib arm as compared with BAT was also demonstrated based on the recent 3-year follow-up data from the COMFORT-II study. The Kaplan-Meier estimated probability of survival at 144 weeks was 81% in the ruxolitinib arm and 61% in the BAT arm (Cervantes, 2012). Improvement in bone marrow fibrosis was observed in 15% of subjects receiving ruxolitinib at 24 months compared with 5% of subjects who received BAT; however, the improvements declined by 48 months in the small number of subjects who were available for follow-up. It is unclear if any of the subjects who were included in this study achieved clinical resolution of their spleen and symptoms (Kvasnicka, 2013).

# 1.1.3. Approved Therapies

Ruxolitinib is approved in the United States (US) and in the European Union (EU) for the treatment of MPN-associated myelofibrosis.

In the US, ruxolitinib (Jakafi®) has been approved by the Food and Drug Administration (FDA) in November 2011 for the treatment of patients with intermediate or high-risk myelofibrosis, including primary myelofibrosis, post-polycythemia vera myelofibrosis and post-essential thrombocythemia myelofibrosis. On 16 August 2019, Inrebic® (fedratinib) was approved by the US FDA for the treatment of adult patients with intermediate-2 or high-risk primary or secondary (post-polycythemia vera or post-essential thrombocythemia) myelofibrosis (MF).

In the EU, ruxolitinib (Jakavi®) has been approved by the European Medicines Agency (EMA) in August 2012 for the treatment of disease-related splenomegaly or symptoms in adult patients with primary myelofibrosis (also known as chronic idiopathic myelofibrosis), post polycythemia vera myelofibrosis or post essential thrombocythemia myelofibrosis.

#### 1.1.4. Medical Need

MPN-associated myelofibrosis, particularly intermediate or high-risk disease, is a serious and fatal condition. Until recently, ruxolitinib, a JAK1/2 inhibitor, was the only drug approved for the treatment of patients with intermediate or high-risk MF. While the benefits of ruxolitinib therapy in terms of spleen response and improvement of constitutional symptoms are significant, ruxolitinib is also associated with the risks of treatment-associated anemia (40.4% vs 12.3% for BAT) and thrombocytopenia (44.5% vs 9.65% for BAT) (Harrison, 2012). The 1-, 2-, and 3-year discontinuation rates are 49%, 71% and 86%, respectively. Major reasons for ruxolitinib treatment discontinuation are loss of therapeutic effect, lack of response and drug-induced cytopenias (Tefferi, 2011). Additionally, responses to ruxolitinib are typically observed within the first 3–6 months after therapy initiation (Harrison, 2012; Verstovsek, 2012) and it has been suggested that for patients who have not had a reduction in spleen size or improvement in symptoms after that period, alternative therapies should be considered (Harrison, 2018a; Keohane, 2013). The effect of ruxolitinib on overall survival (OS) continues to be debated and the unclear limited effects on bone marrow fibrosis and driver mutation allele burden suggest that the disease-modifying activity of the drug is likely to be minor. Therefore, the unmet medical need for frontline MF patients remains high, despite the availability of ruxolitinib, especially for patients who have low baseline platelet counts and are susceptible to myelosuppression/thrombocytopenia.

For patients who have been previously treated with a JAK inhibitor, there is no approved therapy and the prognosis is poor (Newberry, 2017). Mechanisms of resistance to ruxolitinib remain unclear. It has been shown preclinically that MF is intrinsically more resistant to JAK2 inhibition than PV or ET and there continues to be a major unmet need for a JAK2 inhibitor that is effective after ruxolitinib treatment failure. Moreover, the median survival of relapsed and refractory patients who discontinued ruxolitinib has been reported to be 6 months (Jabbour, 2013). Notably, after a median follow-up of 10 months from stopping ruxolitinib, only 34% of patients remained alive (Kantarjian, 2013). Only 27% of patients remained on therapy after 5 years in the COMFORT-I trial. Outcomes for patients who discontinue ruxolitinib in this situation are poor.

Two randomized studies assessed the use of JAK inhibitors for subjects with previous ruxolitinib treatment in comparison to BAT that included continuous or retreatment with ruxolitinib.

In the PERSIST-2 study subjects with a platelet count  $100 \times 10^9$ /L or less were randomized to receive either pacritinib 400 mg once daily, 200 mg twice daily or BAT. BAT included

ruxolitinib and ruxolitinib was used in 44/98 (45%) subjects as BAT. In the subgroup of subjects (n=95) with prior ruxolitinib, a spleen volume response of 35% or more at week 24 was achieved at week 24 in 2 subjects (6%) and 4 subjects (13%) and in 1 subject on BAT (3%) respectively (Mascarenhas, 2018).

In the SIMPLIFY-2 study MF subjects (n=156) with previous ruxolitinib treatment for at least 28 days who either required red blood cell transfusions while on ruxolitinib or ruxolitinib dose reduction to less than 20 mg twice a day with at least one of Grade 3 thrombocytopenia, anemia, or bleeding at Grade 3 or worse were randomized 2:1 to receive either momelotinib or BAT including ruxolitinib.

A spleen volume response of 35% or more at week 24 was achieved at week 24 in 7 subjects (7%) and 3 subjects on BAT (6%) (Harrison, 2018b).

Currently, best available therapy (BAT) to treat patients with MF that have been previously treated ruxolitinib is limited. BAT may include retreatment with ruxolitinib, chemotherapy (eg, hydroxyurea), anagrelide, corticosteroids, hematopoietic growth factor, immunomodulating agents, androgens, interferon, and may also include "no treatment" and symptom directed treatment.

Therefore, there remains an unmet need for the patients who have been previously treated with a JAK inhibitor due to the low life expectancy, notably high discontinuation rate with ruxolitinib and the myelosuppression.

# 1.2. Fedratinib

Fedratinib is an oral kinase inhibitor with activity against wild type and mutationally activated Janus Kinase 2 (JAK2) and fibromyalgia syndrome (FMS)-like tyrosine kinase 3 (FLT3). Fedratinib is a JAK2-selective inhibitor with higher potency for JAK2 over family members JAK1, JAK3 and tyrosine kinase 2 (TYK2). In cell models expressing mutationally active JAK2 or FLT3, fedratinib reduced phosphorylation of signal transducer and activator of transcription (STAT3/5) proteins, inhibited cell proliferation, and induced apoptotic cell death. In mouse models of JAK2V617F-driven myeloproliferative disease, fedratinib blocked phosphorylation of STAT3/5, increased survival and improved disease-associated symptoms, including reduction of white blood cells, hematocrit, splenomegaly, and fibrosis.

Eighteen clinical studies were conducted with fedratinib. Fedratinib has been studied extensively in the treatment of patients with MPN-associated myelofibrosis.

Fedratinib demonstrated clinical efficacy in a randomized, placebo-controlled, Phase 3 study (JAKARTA [EFC12153]) in patients with intermediate-2 or high-risk MF who were previously untreated. The primary endpoint was response rate, defined as the proportion of subjects who had a  $\geq$  35% reduction in spleen volume from baseline to the End of Cycle 6 and confirmed 4 weeks later by MRI. Analyses for spleen response were also performed at the end of Cycle 6 (eg, regardless of confirmation), as recommended by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Criteria. Symptom response rate (SRR), based on a patient-reported outcome (PRO) tool, the modified Myelofibrosis Symptom Assessment Form (MFSAF) that assessed 6 key MF-associated symptoms (night sweats, pruritus, abdominal discomfort, early satiety, pain under ribs on left side, and bone or muscle pain) was a key secondary endpoint. The SRR was defined as the

proportion of subjects with a  $\geq$  50% reduction in the Total Symptom Score (TSS) of the modified MFSAF diary from baseline to the end of Cycle 6. Both endpoints are measures for demonstrating clinical benefit in the proposed population. The response rate per primary endpoint was 36.5% and 40.2% at the 400 mg (proposed dose for this study) and 500 mg daily dose respectively vs 1% on the placebo arm. The response rate at Cycle 6 as recommended by IWG-MRT was of 46.9% and 49.5% in patients treated with the 400 mg and 500 mg daily doses respectively. A total of 36.3% and 34.1% of subjects at the dose of 400 mg and 500 mg doses respectively achieved a  $\geq 50\%$  reduction in TSS compared with 7.1% of subjects receiving placebo. Median duration of response (≥35% reduction in spleen volume) was 10.4 months for responders from both active groups (400-mg and 500-mg groups). The most common treatmentemergent adverse events (TEAEs) of all grades reported in the fedratinib 400-mg daily dose group were diarrhea 65.6%, nausea 63.5%, anemia (G3 and G4) 42.7%, vomiting 41.7%, fatigue 15.6%, and peripheral edema 15.6%. The 400-mg dose was confirmed to be better tolerated than the 500-mg dose, in particular with fewer subjects reporting Grade 3 or 4 TEAEs (54.2% and 70.1%, respectively), treatment-emergent serious adverse events (SAEs) (27.1 % and 30.9%, respectively) and TEAEs leading to permanent treatment discontinuation (13.5% and 24.7%, respectively) (Pardanani, 2015).

The single-arm Phase 2 JAKARTA2 study (ARD12181) enrolled patients with intermediate-1 with symptoms, intermediate-2 or high-risk MPN-associated myelofibrosis who have been previously treated with ruxolitinib. The primary endpoint was response rate, which was defined as the proportion of subjects who have  $a \ge 35\%$  reduction from baseline in spleen volume to the End of Cycle 6 in the per protocol defined population.

As in the Phase 3 JAKARTA study, one of the key secondary endpoints was symptom response rate (SRR), defined as the proportion of subjects with  $a \ge 50\%$  reduction in the TSS using the modified MFSAF diary from baseline to the end of Cycle 6.

Resistance to ruxolitinib was defined as any one of the following: a) lack of response: absence of response; b) disease progression: spleen size increase during ruxolitinib treatment; or c) loss of response at any time during ruxolitinib treatment. Intolerance to ruxolitinib was defined as any one of the following: a) hematologic toxicity (anemia, thrombocytopenia, others); b) non-hematologic toxicity.

The overall spleen response rate (proportion of patients with  $\geq$  35% reduction from baseline in spleen volume to the End of Cycle 6) was 55.4%. A total of 25.6% of subjects achieved a  $\geq$  50% reduction in TSS.

All 97 patients had at least 1 TEAE (all grades); Grade 3 or 4 TEAEs were reported by 62.9% patients. The most common nonhematologic TEAEs (reported by  $\geq$  10% of patients) (all grades) were gastrointestinal disorders including diarrhea (61.9%), nausea (55.7%), and vomiting (41.2%). The most common hematologic TEAEs (reported by > 10 patients) (all grades) were anemia (48.5%) and thrombocytopenia (26.8%). Thirty-eight and one-tenth percent experienced Grade 3 or 4 anemia and 21.6% experienced Grade 3 or 4 thrombocytopenia. No Grade 5 hematologic TEAEs were reported. Anti-infectives for systemic use were given to 55.7% patients in the study (Harrison, 2017).

The JAKARTA2 study was initiated shortly after ruxolitinib was approved and at the time, there were no well-established criteria to define resistance or intolerance. Therefore, subjects were

classified as resistant or intolerant to ruxolitinib per the Investigators' assessments and, to be eligible for the study, they were only required to have been treated with ruxolitinib for 14 days at a minimum.

Subsequently, analyses were performed on subjects enrolled in the JAKARTA2 study and determined to be relapsed/refractory or intolerant to ruxolitinib based on more stringent criteria recommended by MF experts. For 79/97 subjects that meet the more stringent definition for relapsed/refractory or intolerant to ruxolitinib, 24 subjects (30.4%) in the intent-to-treat (ITT) population achieved  $\geq$  35% spleen volume reduction at the end of Cycle 6 and 20 out of 74 subjects (27%) in the MFSAF analysis population achieved a  $\geq$  50% reduction in the symptom score relative to baseline.

Please refer to the Investigator's Brochure (IB) for detailed information concerning the available pharmacology, toxicology, drug metabolism, clinical studies, and adverse event profile of fedratinib.

# 1.3. Wernicke Encephalopathy (WE) in Patients Treated with Fedratinib

On 15 November 2013, all clinical studies ongoing at the time in the fedratinib clinical program were placed on clinical hold by the FDA. The hold decision was made based on provided preliminary data on fatal and serious cases of WE and heart failure that occurred in patients treated with fedratinib. Three days later, the fedratinib clinical program was terminated by the previous sponsor and all subjects were permanently discontinued from fedratinib treatment. Supplementation with thiamine (as well as monitoring of thiamine levels) and follow-up for safety for at least 90 days after the last dose of fedratinib were offered to all subjects in the ongoing studies including those who had previously been discontinued. No cases of WE were observed during this period.

No subject has been treated with fedratinib in the clinical trial setting since December 2013.

Independent central review of the data from all patients was performed to assess for potential cases of WE. Ultimately, 8 potential cases of WE were identified among 807 healthy subjects and patients who were enrolled and treated in the fedratinib clinical trials (193 healthy volunteers, 75 patients with solid tumors, and 539 patients with MF). No case of WE was observed at doses of 400 mg or lower. Further analysis of the data surrounding these events suggest that while cases of WE did occur in subjects treated with fedratinib, the subjects had considerable predisposing factors that are known to lead to WE in any population. In addition, preclinical studies demonstrated that fedratinib does not have an effect on the thiamine receptor function (data on file), it does not actively cause WE. Taken together, the possible WE experienced by these patients is likely related to thiamine deficiency due to increased use in a hypermetabolic environment found in malignancies and decreased availability from underlying poor nutrition coupled with gastrointestinal adverse events experienced by these patients.

The FDA removed the clinical hold on 18 August 2017. The agency required that risk mitigation for WE be implemented for further clinical studies.

This study includes routine thiamine monitoring and supplementation in order to mitigate the risk for WE in this study. Additionally, the use of fedratinib 400 mg daily dosing with proactive treatment of nausea, vomiting, and diarrhea will further help to prevent thiamine deficiency in the study patients.

#### 1.4. Rationale

# 1.4.1. Study Rationale and Purpose

MPN-associated myelofibrosis (MF) is a serious and life-threatening disease. The only approved therapy currently available is the JAK1/2 inhibitor ruxolitinib.

For patients who have been previously treated with ruxolitinib and who failed first-line treatment, there is no approved therapy and prognosis for these patients is poor.

Fedratinib is a potent and selective, orally available JAK2 inhibitor.

The single-arm Phase 2 JAKARTA2 study of fedratinib enrolled patients with intermediate-1 with symptoms, intermediate-2 or high-risk MPN-associated myelofibrosis who were previously treated with ruxolitinib. In that study, fedratinib at a starting dose of 400 mg daily, resulted in a reduction in splenomegaly at the end of cycle 6 (last observation carried forward) (response rate 55.4%) and improvement in symptom burden (response rate: 25.6%).

The study was affected by the clinical hold mandated by the US FDA of the fedratinib development program in November 2013 due to reports of Wernicke encephalopathy (WE) and all subjects on treatment with fedratinib were discontinued from treatment.

Based on the presentation of further analyses, the US FDA removed the clinical hold in August 2017 and required that steps be implemented to mitigate the risk for Wernicke encephalopathy for future clinical studies.

The present study is a multicenter, randomized, open-label, Phase 3 study designed with the purpose to assess the efficacy of fedratinib administered at the dose of 400 mg daily orally in successive 28-day cycles as compared to BAT and to further evaluate the safety of fedratinib in subjects previously treated with ruxolitinib and with DIPSS-intermediate-2 or high-risk primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis.

This study will also implement and assess the effectiveness of risk mitigation strategies for Encephalopathy, including Wernicke's, including routine thiamine monitoring and supplementation, monitoring for signs and symptoms of Encephalopathy, including WE, and proactive management of nausea, vomiting, and diarrhea to prevent thiamine deficiency.

The study will also provide additional data to specify population Reported Outcomes and Health-related Quality of Life.

# 1.4.2. Rationale for the Study Design

This is a multicenter, 2:1 randomized, Phase 3 study with spleen volume reduction at the end of Cycle 6 as the primary objective.

The secondary objectives of the study are to further evaluate the safety and to implement and to assess the effectiveness of risk mitigation strategies for Encephalopathy, including Wernicke's and for gastrointestinal (GI) adverse events.

The primary endpoint is the proportion of subjects who have  $a \ge 35\%$  reduction in spleen volume (response rate measured by MRI or computed tomography [CT] scan and assessed by central

blinded review) at the end of Cycle 6. The primary endpoint follows the established response criteria by IWG-MRT (Tefferi, 2013).

With the assumption of a 20% drop-out rate and a true response rate (considering drop-outs) in the BAT arm of 10%, in the fedratinib arm of 28%, 192 subjects will yield approximately 90% power at a one-sided significance level of 0.025. (Refer to Section 9.3).

The assumption of a 28% spleen volume response rate is in line with the results of the JAKARTA-2 study and the assumption of a 10% spleen volume response rate for BAT is derived from similar studies, such as SIMPLIFY-2 and PERSIST-2 (Harrison, 2018b; Mascarenhas, 2018), considering the variability and limited predictably of BAT use in this study.

Considering the potential lack of therapeutic effect of BAT the crossover will allow subjects access to fedratinib and provide additional data on safety and efficacy of fedratinib without affecting assessment of the primary endpoint of the study.

Safety will be assessed by evaluating adverse events and laboratory data. Adverse events and abnormal laboratory value severity will be graded using Version 5.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).

Efficacy in terms of spleen response will be objectively assessed by MRI/CT scans that will be reviewed centrally by an independent reviewer. Spleen response by palpation as well as symptom response will also be assessed.

Symptoms response rate (SRR) will be assessed by the change from baseline to end of cycle 6 of symptoms measured by the MFSAF version 4.0. SRR is a key secondary endpoint because symptoms are an important aspect of the disease, many of which are driven by splenomegaly.

An additional key secondary endpoint is a spleen response rate (RR25) for the subjects who have  $\geq 25\%$  reduction in spleen volume at the end of cycle 6. This addresses the situation in subjects previously treated with ruxolitinib that a 35% reduction of the spleen volume might be only achieved in a small proportion of subjects.

To ensure subjects are evaluable for the key secondary endpoints, the study will randomize subjects with measurable splenomegaly and symptoms score  $\geq 1$  at baseline.

# 1.4.3. Rationale for Dose, Schedule and Regimen Selection

Fedratinib capsules will be administered orally, once-daily at a dose of 400 mg.

Dose finding (study TED12037) and dose ranging (study ARD11936) studies with fedratinib were performed, with the maximum tolerated dose (MTD) being 680 mg for patients with MPN-associated myelofibrosis.

In the JAKARTA study, doses of 400 mg and 500 mg were used in separate study arms, and while the efficacy in terms of spleen response was similar, the 400-mg dose was better tolerated than the 500-mg dose, in particular with fewer subjects reporting Grade 3 or 4 treatment-emergent adverse events (TEAEs) (70.8% and 78.4%, respectively) and TEAEs leading to permanent treatment discontinuation (27.1% and 36.1%, respectively).

Fedratinib dose modifications will be allowed based on observed toxicity to a 300 mg or 200 mg daily dose in this study. Provisions are in place to allow further dose reduction for subjects with co-medication with moderate or strong Cytochrome P450 3A4 (CYP3A4) inhibitors.

Currently there is no established standard of care and no approved treatment option after previous ruxolitinib treatment. Best available therapy has been used as a comparator in studies with subjects previously exposed to ruxolitinib.

# 1.4.4. Rationale for Patient-Reported Outcomes

Beyond the risk of progression to AML and reduced survival, patients with myelofibrosis experience a variety of complications, such as symptomatic enlargement of the spleen and liver, anemia, cachexia, and the other MF-associated symptoms. These symptoms and the need to face the considerable burden from regular transfusions result in greatly compromised quality of life (QoL) in these patients (Mesa, 2007).

In the study protocol, Celgene has identified and prioritized the patient-reported MF-associated symptoms (night sweats, pruritus, abdominal discomfort, early satiety, pain under ribs on left side, bone or muscle pain, and fatigue); they are assessed by a specific PRO measure, the MFSAF version 4.0. The MFSAF is a specific self-administered and validated PRO tool that has been developed to assess MF-associated symptoms and has been used in several prior studies in MF population (Harrison, 2012; Mesa, 2013). The MFSAF version 4.0. is the most recent version developed in collaboration with industry and the FDA, validated and recommended to be used in clinical trials to assess MF symptoms (Gwaltney, 2017).

The European Organization for Research and Treatment of Cancer (EORTC QLQ-C30) version 3.0 is a self-administered, well-known, and validated questionnaire developed to assess the QoL of cancer patients. It is the most commonly used PRO instrument in oncology studies and has been used to assess QoL in MF patients (Mesa, 2013).

Data from the registration trial COMFORT-I assessing ruxolitinib versus BAT indicate that both patient-assessed MF-symptoms using the MFSAF and Health-related Quality of Life (HRQoL) assessed by the EORTC QLQ-C30 are improved in MF patients when clinical improvement in reduction of splenomegaly is achieved (Mesa, 2013).

These data suggest that patient-assessed MF symptoms and HRQoL should be considered as a key endpoint when assessing the efficacy of a novel treatment for this patient population.

The SRR based on the total symptom score of the MFSAF version 4.0 (proportion of subjects with  $\geq 50\%$  reduction in MFSAF TSS at end of cycle 6) is assessed as the key secondary efficacy endpoint. A 50%-reduction in TSS is an accepted endpoint that has already supported label claims in drugs developed MF. The timepoint for its assessment (end of cycle 6) is aligned with the timepoint for assessing the primary endpoint (spleen volume response rate). This timeframe is considered sufficient to assess an effect of treatment on patient-reported MF-associated symptoms and to evaluate the durability of symptom response.

Other PROs assessed by the EORTC QLQ-C30 domains will be considered as secondary endpoints. They will be assessed on Day 1 of each treatment cycle, at the End of Treatment (EOT) and the 30-day follow-up visit after last dose of study treatment, before the subject undergoes any procedure to avoid bias. This schedule would allow to capture any change in subject-reported symptoms, functioning level or HRQoL.





#### 2. STUDY OBJECTIVES AND ENDPOINTS

# **Table 1:** Study Objectives

# **Primary Objective**

The primary objective of the study is:

• To evaluate the percentage of subjects with at least 35% spleen volume reduction in the fedratinib and the BAT arms

# **Secondary Objective(s)**

The secondary objectives are:

- To evaluate the percentage of subjects with at least 50% reduction in myelofibrosis (MF)-associated symptoms as measured by the Myelofibrosis Symptom Assessment Form (MFSAF) (Appendix B)
- To evaluate the percentage of subjects with at least 25% spleen volume reduction (SVR)
- To evaluate the safety of fedratinib
- To evaluate the reduction of spleen size by palpation
- To evaluate durability of spleen response by MRI/CT and by palpation
- To evaluate the durability of symptoms response
- To evaluate spleen and disease progression free survival
- To assess the effectiveness of the risk mitigation strategy for gastrointestinal events and Encephalopathy, including Wernicke's
- To evaluate Health-Related Quality of Life (HRQoL) as measured by the European Organization for Research and Treatment of Cancer Quality of Life C30 (EORTC QLQ-C30) (Appendix C)
- To evaluate Patient-Reported Outcomes (PRO) as measured by the EQ-5D-5L questionnaire (Appendix D)
- To evaluate Overall Survival (OS)

**Study Objectives (Continued)** Table 1:



**Table 2:** Study Endpoints

| Endpoint | Name | Description | <b>Assessment Timeframe</b> |
|---|---|---|---|
| Primary | Spleen volume response rate (RR) | Proportion of subjects who have ≥ 35% SVR at end of cycle 6 | From Screening to the end of Cycle 6 |
| Key<br>Secondary | Symptom response rate (SRR) | Proportion of subjects with ≥ 50% reduction in total symptom scores measured by MFSAF at end of cycle 6 | From C1D1 to the end of Cycle 6 |
| | Spleen volume<br>response rate<br>(RR25) | Proportion of subjects who have ≥ 25% reduction in spleen volume at the end of cycle 6 | From Screening to the end of Cycle 6 |
| Secondary | Safety profile of fedratinib | Incidence and severity of all Grade<br>AEs per NCI CTCAE (Appendix E)<br>Incidence and severity of Grade 3-4<br>AEs as per the NCI CTCAE<br>(Appendix E), including laboratory<br>parameters | From ICF signature up until 30 days after last dose For fedratinib related AEs, anytime until the last study visit |
| | Spleen response rate by palpation (RRP) | Proportion of subjects who have ≥ 50% reduction in spleen size by palpation at end of cycle 6 | From C1D1 to the end of Cycle 6 |
| | Durability of spleen volume response (DR) | Duration of ≥ 35% SVR | From screening to the End of Treatment visit |
| | Durability of<br>spleen response by<br>palpation (DRP) | Duration of $\geq$ 50 % reduction in spleen size by palpation for subjects with a palpable spleen at least 5 cm below the left costal margin (LCM) at baseline | From C1D1 until the 30-day follow-up after last dose visit |
| | Durability of<br>symptoms<br>response (DSR) | Duration of ≥ 50% reduction in total symptom scores measured by MFSAF | From C1D1 until the 30-day follow-up after last dose visit |
| | Spleen and disease<br>progression free<br>survival (SDPFS) | Time from randomization to death due to any reason or disease progression (modified IWG-MRT 2013 including ≥ 25% increase in spleen volume by MRI/CT) | From randomization to<br>the End of Survival<br>Follow-up |

Table 2: Study Endpoints (Continued)

| Endpoint | Name | Description | Assessment Timeframe |
|---|---|---|---|
| Secondary Assessment of effectiveness or risk mitigation strategy for gastrointestina adverse events Encephalopath including Wernicke's HRQoL meast by EORTC QC C30 domains | gastrointestinal<br>adverse events and<br>Encephalopathy,<br>including | Incidence of subjects with a CTCAE Grade ≥3 of nausea, diarrhea, or vomiting, or occurrence of Encephalopathy, including Wernicke's (confirmed by brain MRI or autopsy). Assessment of thiamine levels at screening, on Day 1 of the first 3 cycles and every third cycle thereafter, and at the End of Treatment visit | From ICF signature to<br>the 30-day follow-up<br>after last dose visit |
| | HRQoL measured<br>by EORTC QOL-<br>C30 domains | Mean changes in the HRQoL function<br>and symptom domain scores over the<br>study compared with baseline | From C1D1 to Day 1 of<br>each cycle, at the End of<br>Treatment visit up to the<br>30-day follow-up after<br>last dose visit |
| | PRO measured by EQ-5D-5L | Mean changes in the health utility scores over the study compared with baseline measured by EQ-5D-5L | From C1D1 to Day 1 of<br>each cycle, at the End of<br>Treatment visit up to the<br>30-day follow-up after<br>last dose visit |
| | Overall Survival | Time from randomization to death due to any reason | From randomization to<br>the End of Survival<br>Follow-up |

**Table 2:** Study Endpoints (Continued)

| Endpoint | Name | Description | Assessment Timeframe |
|----------|------|-------------|----------------------|

AEs = adverse events; C1D1 = cycle 1 day 1; CT = computed tomography; CTCAE = Common Terminology Criteria for Adverse Events; EORTC QLQ-C30= European Organization for Research and Treatment of Cancer Quality of Life instrument; HRQoL = Health-related Quality of life; ICF = informed consent form; LCM = left costal margin; MFSAF = Myelofibrosis Symptom Assessment Form; MRI = magnetic resonance imaging;

NCI = National Cancer Institute; PRO = patient-reported outcome;

WE =Wernicke encephalopathy.

# 3. OVERALL STUDY DESIGN

# 3.1. Study Design

The study will be conducted in compliance with the International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

This is a Phase 3 multicenter, open-label, randomized, multinational study in subjects previously treated with ruxolitinib and with Dynamic International Prognostic Scoring System (DIPSS) (Appendix F) intermediate-2 or high risk PMF (Appendix G and Appendix H), post-PV or post-ET MF (Appendix I).

The study will consist of 3 periods: a Screening Period, a Treatment Period including a 30-day follow-up after last dose visit and a survival follow-up period. The overall study design is described in Figure 1, with more detail for each period of the study design found in Section 6.

# **Screening Period**

All enrolled subjects will undergo screening procedures during the screening period which must be completed within 28 days prior to the start of study treatment. This will serve to determine subject eligibility based on all inclusion and exclusion criteria defined in the protocol. For subjects that are receiving ruxolitinib during the screening period or that have potentially reversible laboratory abnormalities (or other criteria that excludes subjects from randomization) detected during screening, the screening period may be extended to 35 days (additional 7 days).

If needed, randomization will be preceded by a taper-off period for previous treatment according to the prescribing information and a washout period for previous treatment in line with the inclusion and exclusion criteria which is to be started at least 14 days before randomization. When screening a subject, it is necessary to account for the required duration of the ruxolitinib washout period of 14 days and the need to perform the MRI or CT scan within 3 days before randomization.

#### Randomization

Upon confirmation of eligibility, subjects will be randomized 2:1 to receive treatment with fedratinib at a dose of 400 mg once daily orally continuously or treatment with BAT.

#### **Treatment Period**

Cycles are defined for administrative purposes as 4-week (28 day) periods irrespective of the assigned treatment arm. Unless otherwise noted, visit windows are  $\pm$  3 days except for MRI/CT scan procedures which have a visit window of  $\pm$  7 days. For the first 3 cycles, site visits will be performed on Day 1 and Day 15 and thereafter on Day 1 for the subsequent cycles. At Cycle 1 Day 8 the site will contact the subject by telephone to assess occurrence and discuss management of nausea, vomiting and diarrhea. Subjects may continue treatment with study treatment until unacceptable toxicity, lack of therapeutic effect, progression of disease according to the IWG-MRT 2013 criteria or until consent is withdrawn.

Subjects may crossover from the BAT arm to the fedratinib arm at any time before the Cycle 6 response assessment in the event of a confirmed progression of splenomegaly (by MRI/CT scan) or after the Cycle 6 response assessment.

Subjects on the BAT arm that discontinue treatment before cycle 6 response assessment without confirmed progression of splenomegaly are allowed to stay on study and eventually cross-over at cycle 6 response assessment.

All subjects will be monitored for adverse events during the study.

All subjects discontinued from protocol-prescribed therapy for any reason will be followed for a period of 30 days following the last dose of study drug to collect safety data.

# **Survival Follow-up Period**

All subjects discontinued from protocol-prescribed therapy for any reason will be followed for survival, subsequent therapies, new malignancy and progression of myelofibrosis to acute myeloid leukemia (AML) every 3 months until death, lost to follow-up, withdrawal of consent for further data collection, or study closure, whichever comes first.

Figure 1: Overall Study Design



AML = acute myeloid leukemia; AE = adverse events; ANC = absolute neutrophil count; DIPSS = Dynamic International Prognostic Scoring System; GI = gastrointestinal; Int = intermediate; LCM = left costal margin; MF = myelofibrosis; MPN = myeloproliferative neoplasm; MRI = magnetic resonance imaging; PB = peripheral blood; PO = oral; QoL/PRO = quality of life/patient-reported outcomes; SVR = spleen volume reduction; WE = Wernicke encephalopathy.

# 3.2. Study Duration for Subjects

The average treatment period for each subject in the fedratinib arm is expected to be approximately 12 months. Subjects receiving BAT may crossover to fedratinib treatment as
specified in Section 6.5. The actual study duration for an individual subject will be dependent upon the actual treatment duration and survival Follow-up duration and is expected not to exceed 5 years. This duration includes at least 36 months for treatment and follow-up, or until death, lost to follow-up, withdrawal of consent for further data collection, or study closure whichever comes first.

#### 3.3. End of Trial

The End of Trial is defined as the date of the last visit of the last subject to complete the Survival Follow-up or the date of receipt of the last data point from the last subject that is required for primary, secondary as prespecified in the protocol, whichever is the later date.

End of trial is expected approximately 3 years after the last subject is randomized.

The trial completes when all key endpoints and objectives of the study have been analyzed. The subjects who remain on active treatment and are continuing to derive benefit may have available to them either a roll-over protocol, or alternative means for providing study drug to them after study closure.

#### 4. STUDY POPULATION

## 4.1. Number of Subjects

The multinational study will enroll approximately 192 subjects previously treated with ruxolitinib (as per the definition below) and with DIPSS-intermediate-2 or high risk PMF, post-PV MF or post-ET MF.

#### 4.2. Inclusion Criteria

Subjects must satisfy the following criteria to be enrolled in the study:

- 1. Subject is at least 18 years of age at the time of signing the informed consent form (ICF)
- 2. Subject has an Eastern Cooperative Oncology Group (ECOG) (Appendix J) Performance Score (PS) of 0, 1 or 2
- 3. Subject has diagnosis of primary myelofibrosis (PMF) according to the 2016 World Health Organization (WHO) criteria (Appendix G and Appendix H), or diagnosis of post-ET or post-PV myelofibrosis according to the IWG-MRT 2007 criteria (Appendix I), confirmed by the most recent local pathology report
- 4. Subject has a DIPSS Risk score of Intermediate-2 or High (Appendix F)
- 5. Subject has a measurable splenomegaly during the screening period as demonstrated by spleen volume of  $\geq 450 \text{ cm}^3$  by MRI or CT-scan (refer to Section 6.1) and by palpable spleen measuring  $\geq 5$  cm below the left costal margin
- 6. Subject has a measurable total symptoms score (≥ 1) as measured by the Myelofibrosis Symptom Assessment Form (MFSAF)
- 7. Subject has been previously exposed to ruxolitinib, and must meet at least one of the following criteria (a and/or b)
  - a. Treatment with ruxolitinib for  $\geq 3$  months with inadequate efficacy response (refractory) defined as < 10% spleen volume reduction by MRI or < 30% decrease from baseline in spleen size by palpation or regrowth (relapsed) to these parameters following an initial response
  - b. Treatment with ruxolitinib for  $\geq 28$  days complicated by any of the following (intolerant):
    - Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months) or
    - Grade  $\geq$  3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while on treatment with ruxolitinib
- 8. Subject must have treatment-related toxicities from prior therapy resolved to Grade 1 or pretreatment baseline before start of last therapy prior to randomization
- 9. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted

- 10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
- 11. A female of childbearing potential (FCBP) must:
  - a. Have 2 negative pregnancy tests as verified by the Investigator during screening prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence\* from heterosexual contact.
  - b. Either commit to true abstinence\* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use and be able to comply with highly effective contraception\*\* without interruption, -14 days prior to starting investigational product, during the study treatment (including dose interruptions), and for 30 days after discontinuation of study treatment.

Note: A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

#### 12. A male subject must:

Practice true abstinence\* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 30 days following investigational product discontinuation, or longer if required for each compound and/or by local regulations, even if he has undergone a successful vasectomy.

- \* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).
- \*\* Agreement to use highly effective methods of contraception that alone or in combination resulting in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly throughout the course of the study. Such methods include: Combined (estrogen and progestogen containing) hormonal contraception: Oral; Intravaginal; Transdermal; Progestogen-only hormonal contraception associated with inhibition of ovulation: Oral; Injectable hormonal contraception; Implantable hormonal contraception; Placement of an intrauterine device; Placement of an intrauterine hormone-releasing system; Bilateral tubal occlusion; Vasectomized partner.

#### 4.3. Exclusion Criteria

The presence of any of the following will exclude a subject from randomization:

- 1. Any of the following laboratory abnormalities:
  - a. Platelets  $< 50 \times 10^9/L$
  - b. Absolute neutrophil count (ANC)  $< 1.0 \times 10^9/L$
  - c. White blood count (WBC)  $> 100 \times 10^9/L$
  - d. Myeloblasts  $\geq 5$  % in peripheral blood
  - e. Estimated glomerular filtration rate < 30 mL/min/1.73 m² (as per the Modification of Diet in Renal Disease [MDRD] formula) (Appendix K)
  - f. Serum amylase or lipase > 1.5 x upper limit of normal (ULN)
  - g. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
  - h. Total bilirubin > 1.5 x ULN, subject's total bilirubin between 1.5 3.0 x ULN are eligible if the direct bilirubin fraction is < 25% of the total bilirubin
- 2. Subject is pregnant or lactating female
- 3. Subject with previous splenectomy
- 4. Subject with previous or planned hematopoietic cell transplant
- 5. Subject with prior history of Encephalopathy, including Wernicke's (WE)
- 6. Subject with signs or symptoms of Encephalopathy, including WE (eg, severe ataxia, ocular paralysis or cerebellar signs)
- 7. Subject with thiamine deficiency, defined as thiamine levels in whole blood below normal range according to the central laboratory and not demonstrated to be corrected prior to randomization
- 8. Subject with concomitant treatment with or use of pharmaceutical, herbal agents or food known to be strong or moderate inducers of Cytochrome P450 3A4 (CYP3A4), or dual CYP2C19 and CYP3A4 inhibitors (refer to Section 8 and Appendix L)
- 9. Subject on any chemotherapy, immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), anagrelide, immunosuppressive therapy, systemic corticosteroids > 10 mg/day prednisone or equivalent. Subjects who have had prior exposure to hydroxyurea (eg, Hydrea) in the past may be enrolled into the study as long as it has not been administered within 14 days prior to randomization
- 10. Subject has received ruxolitinib within 14 days prior to randomization
- 11. Subject with previous exposure to Janus kinase (JAK) inhibitor(s) other than ruxolitinib treatment
- 12. Subject on treatment with aspirin with doses > 150 mg daily
- 13. Subject with major surgery within 28 days prior to randomization

- 14. Subject with diagnosis of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemochromatosis, non-alcoholic steatohepatitis)
- 15. Subject with prior malignancy other than the disease under study unless the subject has not required treatment for the malignancy for at least 3 years prior to randomization. However, subject with the following history/concurrent conditions provided successfully treated may enroll: non-invasive skin cancer, in situ cervical cancer, carcinoma in situ of the breast, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system), or is free of disease and on hormonal treatment only
- 16. Subject with uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4) (Appendix M)
- 17. Subject with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC)
- 18. Subject with serious active infection
- 19. Subject with presence of any significant gastric or other disorder that would inhibit absorption of oral medication
- 20. Subject is unable to swallow capsule
- 21. Subject with any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
- 22. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
- 23. Subject has any condition that confounds the ability to interpret data from the study
- 24. Subject with participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to randomization
- 25. Subject with a life expectancy of less than 6 months

## 5. TABLE OF EVENTS

**Table 3:** Table of Events

| Visits | | Treatment Period <sup>a</sup> | | | | | | | | | | 30-Day | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen-<br>ing | | Cycle | 1 | Cy | vele 2 | Cy | cle 3 b | Cycle 4 | Cycle 5 | Cycle 6 | Cycle ≥ 7 | Response c<br>Assessment | End of<br>Treatment<br>(EOT) | Follow-<br>up after<br>last dose | Survival<br>Follow-up<br>every 3<br>months |
| Days | -28 to -1 | Day 1 | Day 8 | Day 15 | Day 1 | Day 15 | Day 1 | Day 15 | Day 1 | Day 1 | Day 1 | Day 1 | End of C3, 6,<br>12, 18, 24 (±7D) | - | (+ 7 days) | (± 14 days) |
| Informed consent | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Inclusion / Exclusion criteria | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Demographics | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Medical History | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Myelofibrosis disease history | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Prior therapies for disease under study | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | 1 |
| IRT subject registration | X | X | - | - | - | - | - | - | - | - | - | - | - | X | - | - |
| Height | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Treatment | | | | | | | | | | | | | | | | |
| Fedratinib dispensing to subject | - | X | - | - | X | - | X | - | X | X | X | X | - | - | - | - |
| Fedratinib accountability | - | - | - | - | X | - | X | - | X | X | X | X | - | X | - | - |
| Fedratinib administration | - | - Once daily with an evening meal including daily dose of thiamine | | | | | | | | - | - | | | | | |
| Safety assessments | Safety assessments | | | | | | | | | | | | | | | |
| Pregnancy test for FCBP only | X | X | - | - | X | - | X | - | X | X | X | X | - | - | X | - |
| Adverse events | | From ICF signature until 30 days after last dose of study treatment and anytime thereafter if suspected to be related | | | | | | | | | | | | | | |
| Risk mitigation for GI & Encephalopathy including WE | | From ICF signature until 30 days after last dose of study treatment - | | | | | | | | | - | | | | | |
| Prior/concomitant medications | | | | | From | 28 days | prior to | C1D1 u | ntil 30 da | ys after | last dose o | of study trea | itment | | | - |

**Table 3:** Table of Events (Continued)

| | | Treatment Period 30-Day | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen<br>-ing | Cycle 1 | | Cycle 2 | | Cycle 3 b | | Cycle 4 | Cycle 5 | Cycle 6 | Cycle ≥ 7 | Response c<br>Assessment | End of<br>Treatment<br>(EOT) | Follow-<br>up after<br>last dose | Survival<br>Follow-up<br>every 3<br>months | |
| Days | -28 to -1 | Day 1 | Day 8 | Day 15 | Day 1 | Day 15 | Day 1 | Day 15 | Day 1 | Day 1 | Day 1 | Day 1 | End of C3, 6,<br>12, 18, 24 (±7D) | - | (+ 7<br>days) | (± 14 days) |
| Prior/concomitant procedures | | | | | Fron | n 28 days | prior to | C1D1 u | ntil 30 da | ays after | last dose | of study trea | atment | | | - |
| Phone call for management of nausea, vomiting, diarrhea | - | - | X | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Vital signs including weight | X | X | - | - | X | - | X | - | X | X | X | X | - | X | X | - |
| Physical exam | X | X | - | - | X | - | X | - | X | X | X | X | - | X | X | - |
| Transfusion burden assessment | From 84 days prior to C1D1 until 30 days after last dose of study treatment | | | | | | | | | | - | | | | | |
| Local 12-lead ECG | X At any time if clinically indicated | | | | | | | | - | | | | | | | |
| Hematology | X | X | - | X | X | X | X | X | X | X | X | X | - | X | X | - |
| Serum Chemistry | X | X | - | X | X | X | X | X | X | X | X | X | - | X | X | - |
| Lipid panel | X | | | | | | X | | | | X (every 3 <sup>rd</sup> cycle) | | | X | | |
| Urinalysis & Coagulation | X | | | | | | | At a | ny time i | f clinica | lly indicat | ed | | | | - |
| Thiamine (whole blood sample) <sup>d</sup> | X | X | - | - | X | - | X | - | - | - | X (every 3 <sup>rd</sup> cycle) | - | - | X | - | - |
| Cognitive assessments (MMSE) <sup>d</sup> | X | - | - | - | X | - | X | - | - | - | X (every 3rd cycle) | - | - | X | - | - |
| Assessment for survival | - | - | - | - | - | - | - | - | - | - | - | - | - | - | X | X |
| Progression of MF to AML assessment | - | - | - | - | - | - | - | - | - | - | - | - | - | - | X | X |
| Subsequent therapies for disease under study | - | - | - | - | - | - | - | - | - | - | - | - | - | - | X | X |
| ECOG PS | X | X | - | - | X | - | X | - | X | X | X | X | - | X | X | - |

**Table 3:** Table of Events (Continued)

| | | | Treatment Period d | | | | | | | | | 30-Day | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | Screen<br>-ing | | Cycle | 1 | Cy | cle 2 | Cyc | ele 3 <sup>b</sup> | Cycle 4 | Cycle 5 | Cycle 6 | Cycle ≥ 7 | Response <sub>c</sub><br>Assessment | End of<br>Treatment<br>(EOT) | Follow-<br>up after<br>last dose | |
| Days | -28 to -1 | Day 1 | Day 8 | Day 15 | Day 1 | Day 15 | Day 1 | Day 15 | Day 1 | Day 1 | Day 1 | Day 1 | End of C3, 6,<br>12, 18, 24 (±7D) | - | (+ 7<br>days) | (± 14 days) |
| Efficacy Assessments | | | | | | | | | | | | | | | | |
| MRI/CT-Scan <sup>e</sup> | X | - | - | - | - | - | - | - | - | - | - | - | X | X | - | - |
| Spleen size by palpation | Х | X | - | - | Х | - | Х | - | X | X | X | Х | X | X | Х | - |
| MFSAF v.4.0 | X | X | - | - | X | - | X | - | X | X | X | X | X | X | X | - |
| Quality of Life Assessments / P | atient-R | eporte | d Outco | omes (PI | RO) | | | | | | | | | | | |
| EORTC QLQ-C30 V3.0, EQ-<br>5D-5L, | - | X | - | - | X | - | X | - | X | X | X | X | - | X | X | - |
| | | | | | ╙ | | | | | | <u> </u> | | | | oxdot | |
| | | | | | | | <b> </b> | | | | | | | | | |

AML = acute myeloid leukemia; BAT = best available therapy; CT = computed tomography; D = days; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; EORTC = European Organization for Research and Treatment of Cancer; EOT = End of Treatment; FCBP = female of childbearing potential: GI = gastrointestinal; ICF = informed consent form; IRT = Interactive Response Technology; MF = myelofibrosis; MFSAF = Myelofibrosis Symptom Assessment Form; MMSE = Mini-mental state

examination; MRI = magnetic resonance imaging;

PS = Performance Status; WE = Wernicke encephalopathy.

<sup>&</sup>lt;sup>a</sup> A window of ± 3 days is allowed during the Treatment Period.

<sup>&</sup>lt;sup>b</sup> Subjects that discontinue study treatment prior to Cycle 4 or prior to Cycle 7 will complete the response assessments in the End of Treatment visit.

<sup>&</sup>lt;sup>c</sup> Response assessments can be done at the same time as the Day 1 visit of the following Cycle. Response assessments are also performed at the end of every 6th cycle after Cycle 24 for spleen volume by MRI/CT scan, spleen size by palpation and symptoms score.

d And at any time if clinically indicated.

e A window of ± 7 days is allowed for MRI/CT scan procedures. The screening MRI/CT scan needs to be performed within 3 days before randomization. MRI/CT scans may be performed at any time during the study if clinical progression of splenomegaly is suspected.

#### 6. PROCEDURES

Any questions regarding the protocol should be directed to the Celgene-Impact Medical Monitor or designee. All data obtained from these assessments must be recorded in the subject's source documentation. Refer to the eCRF (electronic Case Report Form) completion guidelines for additional information related to data entry requirements. Procedures will be performed as stated in the sections below. Detailed instructions for sample collection, processing, storage, shipping and handling will be contained in a separate laboratory manual provided to the sites. Waivers or deviations to the protocol will not be granted during the conduct of this trial, under any circumstances.

In the event that immediate hematology / biochemistry / urinalysis / coagulation / thiamine values are needed for clinical decisions, local laboratory results may be used pending the outcome of the central laboratory assessment. However, matching samples must always be sent to the central laboratory and clinical decisions and assessments must be reconciled with the results of the central laboratory. The results of these additional analyses will be recorded in the subjects' CRF as applicable as described in Section 10.

Procedures and assessments are described in detail below. The timing of all the below assessments / procedures is specified in the Table of Events, Table 3.

## 6.1. Screening Period

All screening procedures and assessments are performed during a subject's screening period in order to establish eligibility and to document relevant medical and demographic data (eg, medical history and prior/concomitant medications). The written informed consent form must be signed before any study-specific procedures are performed and any samples are collected for study-specific analysis. Subject eligibility is established by the Investigator by confirming all inclusion and exclusion criteria are satisfied. The MRI or CT scan for spleen volume assessment should be performed within 3 days before randomization. Inclusion of a subject can be based on a local MRI or CT scan assessment demonstrating a spleen volume of  $\geq 450 \text{ cm}^3$ . Documentation used to establish eligibility should be forwarded to the Sponsor to ensure documentation is sufficient from a regulatory and quality perspective. The Sponsor may contact the study site for additional information if there is any deficiency in the documentation provided. Failure to satisfy any entry criterion will preclude a subject from receiving the first study treatment dose.

The following will be performed during the 28-day Screening Period as specified in the Table of Events (Table 3) after informed consent has been obtained:

- Interactive Response Technology (IRT) Subject Registration:
  - Registration of the subject into the IRT system.
- Assessment of inclusion/exclusion criteria for study eligibility

Screening evaluations will be performed for all subjects to determine eligibility. Screening laboratory values must demonstrate subject eligibility, but may be repeated within the screening window, if necessary.

#### • Demographics

Information about the subject's demographics (if allowed per local country regulations; including, but not limited to: date of birth, sex, race, and ethnicity).

#### • Medical history (including Disease History)

Relevant medical history, including potential alcohol abuse, and current medical conditions, including MF signs and symptoms, must be recorded on the appropriate Case Report Form (CRF) pages at screening. History of myelofibrosis disease including its prior treatments, response to prior therapy with ruxolitinib and current DIPSS (Dynamic International Prognostic Scoring System) Score, other prior malignancies will also be recorded on the appropriate CRF pages. This may include relevant information related to original MF diagnosis and/or other past malignancies as applicable.

Review of historical bone marrow biopsy information will be used to confirm MPN-associated myelofibrosis diagnosis. The report should come from the most recent local bone marrow biopsy performed and should contain the mutational status of the disease (eg, *JAK2*, *MPL*, and *CALR*).

Information regarding **transfusion history** (at least 84 days prior to and including the randomization date), including pretransfusion hemoglobin (Hgb) levels, number of units transfused and dates of transfusions, will be collected and reported in the appropriate eCRF. Any transfusions given at outside institutions must also be collected.

#### • Pregnancy testing

Pregnancy testing is required for all female subjects of childbearing potential. The Investigator will appraise a female subject as a FCBP according to the definition included in the eligibility criteria (Section 4.2). Justification must be recorded in the eCRF and the source document. Pregnancy testing is not required for non-FCBP subjects. Two urine (or serum) pregnancy tests will be performed to assess subject eligibility during screening with one test within 72 hours prior to the first administration of study treatment, if the initial pregnancy test did not already occur within 72 hours of dosing (negative results required for IP administration).

#### Adverse events

All subjects will be monitored for AEs including AESIs (AE of Special Interest) during the study as described in Section 10.

Information about common side effects already known about fedratinib will be included in the subject informed consent form and should be discussed with the subject as needed during the study. This information can also be found in the IB or will be communicated between IB updates in the form of Investigator notifications.

# • Risk mitigation for Gastrointestinal toxicity & Encephalopathy, including Wernicke's

Refer to Section 7.4 and Section 7.5.

#### • Height

Height will be measured only during the screening period.

#### Symptoms Response Assessment using MFSAF version 4.0

Refer to Section 6.3.1 for more information.

#### Prior/concomitant medications

Information relating to prior/concomitant medications are to be reported on the appropriate eCRF pages. Refer to Section 8 for more information. The details of prior treatment by ruxolitinib with outcomes will be recorded in the subject's eCRF.

#### • Prior/concomitant procedures

Information relating to prior/concomitant procedures are to be reported on the appropriate eCRF pages. Refer to Section 8 for more information.

#### • Physical exam

Information about the physical examination for clinically significant findings including assessment of abnormal eye movements, assessment for cerebellar abnormalities, spleen palpation, as well as spleen size assessment are to be captured in the eCRF.

#### • Vital signs including weight

Information regarding vital signs including seated blood pressure (systolic and diastolic), body temperature, heart rate and weight are measured and reported on the appropriate eCRF.

#### • Electrocardiogram (ECG)

A 12-lead ECG is to be performed locally at the site. The following ECG parameters will be recorded on the respective eCRF(s): Heart rate (HR), PR interval, QRS duration, QT, QTc. The Investigator will review the results and assess as normal, abnormal – not clinically significant, or abnormal – clinically significant, and report the abnormal finding(s) on the appropriate eCRF. If the ECG is abnormal, the Investigator should consult a cardiologist if deemed appropriate. An ECG will be performed at screening and if clinically indicated thereafter.

## • Hematology

This assessment may include the following: red blood cells (RBC) count, hemoglobin, hematocrit, mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), platelet count, white blood cell (WBC) count, RBC morphology, and differential cell count including myeloblasts. Detailed instructions for sample collection, processing, storage, shipping and handling will be contained in a separate laboratory manual provided to the sites.

#### • Serum Chemistry

This assessment may include the following: total bilirubin, direct bilirubin, gamma-glutamyl transferase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT), bicarbonate, alkaline phosphatase (AP), lactate dehydrogenase (LDH) amylase, lipase, total protein, albumin, globulin, sodium, potassium, chloride, calcium, phosphate, magnesium, glucose, urea, creatinine and creatinine clearance as per the Modification of Diet in Renal Disease (MDRD) formula, blood urea nitrogen (BUN) and uric acid. Detailed instructions for sample collection, processing, storage, shipping and handling will be contained in a separate laboratory manual provided to the sites.

#### • Lipid panel

This assessment may include the following: cholesterol, high-density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL), very low-density lipoprotein cholesterol (VLDL) and triglycerides.

#### Coagulation

This assessment may include the following: prothrombin time/international normalized ratio and activated partial thromboplastin time. Coagulation testing will be performed at screening and if clinically indicated thereafter.

#### Urinalysis

This assessment may include the following: macroscopic (eg, color, blood, glucose, ketones, leukocyte esterase, nitrite, pH, protein, specific gravity and bilirubin), microscopic (eg, RBC, WBC, casts, crystals, bacteria and epithelial cells). Urinalysis testing will be performed at screening and if clinically indicated thereafter.

#### • Thiamine level

Information regarding thiamine level in whole blood will be tested according to the Table of Events (Section 5) and as clinically indicated.

#### • Cognitive assessment - Mini-Mental State Examination

Information regarding the cognitive status will be performed using the Mini-Mental State Examination (MMSE): to objectively assess for signs/symptoms of encephalopathy.

If the MMSE-2 SV (standard version) questionnaire (Appendix P) is unavailable at the time of study start, the original version of the MMSE questionnaire may be used. This questionnaire is to be completed as specified in the Table of Events (Table 3) and as clinically indicated.

## • Spleen volume by MRI/CT scan

Spleen volume will be assessed at the study site (MRI or CT Scan if MRI is contraindicated) during screening. The screening MRI/CT scan needs to be performed within 3 days prior to randomization. The locally assessed spleen volume will be recorded in the appropriate CRF pages. The same method MRI or CT scan should be

used consistently throughout the study. MRI/CTs will be reviewed centrally. The central review will be blinded for arm assignment, treatment and dose levels.

#### Spleen size by palpation

Spleen size palpation in cm below left costal margin (LCM) will be assessed at the study site.

#### • Eastern Cooperative Oncology Group (ECOG) performance status

Performance status will be assessed by the Investigator using the ECOG criteria provided in Appendix J.

#### • Biomarker assessments

Blood and saliva (saliva sample taken at screening only) for evaluation of biomarkers, such as, but not limited to, mutational analysis, cytogenetics, signaling pathways, gene expression profiling, inflammatory and fibrogenic circulating proteins, including cytokines, circulating cells such as blasts (CD34+ cells) and immune cells. If collection is required on fedratinib dosing days, samples should be obtained prior to administration of fedratinib.

Evaluation of some of the samples may require blood samples to be collected and processed as multiple samples to allow for the possibility of future analyses.

A blood and saliva sample will be drawn for biomarker assessments.

Specified screening assessments must take place within 28 days after the date of the informed consent form signature. For subjects that are on ruxolitinib at the start of the screening period or who have a laboratory abnormality detected during screening, the screening period may be extended to 35 days to allow for retesting to demonstrate resolution of the laboratory abnormality. In case a subject has a laboratory parameter related to an exclusion criterion that was under the influence of a treatment or medication (eg, platelet transfusion in the last 7 days, granulocyte-colony stimulating factor (G-CSF) in last 14 days) retesting needs to be performed before randomization after an appropriate washout period (refer to Section 4.3).

Subjects who fail screening for study entry may be rescreened if it is reasonable to believe they will meet eligibility criteria during rescreening. If screening assessments are not within the allowed screening period, the rescreened subject must reconsent to participation in the study by signing a new and current informed consent form.

## 6.2. Randomization of a Subject to the Study

All the screening evaluations must be completed, and eligibility criteria must be verified by the responsible Investigator. The appropriate documentation may be reviewed by the Sponsor prior to a subject receiving the first study treatment dose. Information needed to stratify a subject must be available at randomization.

Subjects will be randomized 2:1 to fedratinib or best available therapy (BAT).

Stratification at Randomization will be done according to:

• Spleen size by palpation: < 15 cm below LCM versus ≥ 15 cm below LCM

- Platelets  $\geq 50$  to  $< 100 \times 10^9/L$  versus platelets  $\geq 100 \times 10^9/L$
- Refractory or relapsed to ruxolitinib treatment versus intolerance to ruxolitinib treatment
  - See inclusion criteria #7 (a versus b). In case both apply, the criteria for refractory/relapsed will be used for stratification.

Randomization of the subject (inclusion in the Treatment Period) will occur via Interactive Response Technology (IRT) to enable automated tracking and replenishment of fedratinib study treatment. Specific contact information and instructions will be provided to each study site.

The IRT randomization should be performed as close as possible to the planned first dose of study treatment to avoid enrolling a subject who ultimately does not receive study treatment for any reason. The first dose of study treatment should be administered at the site on the day of randomization but may be delayed for up to 3 days if necessary, for logistical reasons.

If screening assessments are performed within 7 days of the C1D1 date, safety laboratory and physical examinations will not need to be repeated during the C1D1 visit except for hematology laboratory assessments.

The BAT assigned will be documented as study treatment on the appropriate pages of the electronic case report form (eCRF).

#### 6.3. Treatment Period

The following procedures/evaluations will be performed at the frequency specified in the Table of Events (Table 3) during the Treatment Period.

Unless otherwise specified, all study visits during the Treatment Period must occur within  $\pm$  3 days of the scheduled day except for MRI/CT scan procedures which have a visit window of  $\pm$ 7 days. For the first 3 cycles, site visits will be performed on Day 1 and Day 15 and thereafter on Day 1 for the subsequent cycles. At Cycle 1 Day 8 the site will contact the subject by telephone to assess management of nausea, vomiting and diarrhea.

The procedures/evaluations should be performed prior to dosing on the visit day, unless otherwise specified. The following will be performed at treatment visits as specified in the Table of Events (Section 5):

- **Pregnancy testing:** As detailed in Section 6.1
- Prior/concomitant medications and procedures: As detailed in Section 6.1
- Phone call for management of nausea, vomiting, diarrhea: will be assessed and managed by telephone contact
- Vital signs, Physical exam and weight: As detailed in Section 6.1
- Electrocardiogram (ECG): As clinically indicated (detailed in Section 6.1)
- **Hematology:** As detailed in Section 6.1

Before starting each treatment cycle, a hematology lab results including ANC, platelet (PLT) and RBC must be available

- Serum Chemistry: As detailed in Section 6.1
- Lipid panel: As detailed in Section 6.1
- Coagulation: As clinically indicated (detailed in Section 6.1)
- Urinalysis: As clinically indicated (detailed in Section 6.1)
- Thiamine level: As detailed in Section 6.1

As clinically indicated and at C1D1, C2D1, C3D1, C6D1 and every 3<sup>rd</sup> cycle thereafter

#### Transfusion burden assessment

Information regarding RBC and PLT transfusions including pretransfusion Hgb or PLT levels, number of units transfused and dates of transfusions, will be collected and reported in the appropriate eCRF. Information regarding any transfusions given at outside institutions must also be collected.

- Cognitive assessment Mini-Mental State Examination: As detailed in Section 6.1
   As clinically indicated and at C2D1, C3D1, C6D1 and every 3<sup>rd</sup> cycle thereafter
- Response Assessment: As detailed in Section 6.4
- Spleen size by palpation: As detailed in Section 6.1
- Eastern Cooperative Oncology Group (ECOG) performance status: As detailed in Section 6.1

• Administration/accountability of study treatment

Refer to Section 7 for details.

- Adverse events: Refer to Section 6.1
- Risk mitigation for gastrointestinal toxicity & Encephalopathy, including Wernicke's

Refer to Section 7.4 and Section 7.5

#### 6.3.1. Symptoms Response Assessment using MFSAF version 4.0

The MF-related symptoms evaluation will be performed using the MFSAF version 4.0 version using a 7-day recall period (Gwaltney, 2017).

This questionnaire assesses 7 key MF-associated symptoms (night sweats, pruritus, abdominal discomfort, early satiety, pain under ribs on left side, bone or muscle pain, and fatigue). Due to the number of different questionnaires used in clinical trials for patient-reported MF symptoms, this version was developed following harmonization work conducted in collaboration with industry and the FDA with the aim to create a publicly available, consensus-based and harmonized version of MF symptoms

questionnaire (Gwaltney, 2017). The MFSAF version 4.0 was validated and recommended to be used in clinical trials to assess MF symptoms.

The Total Symptom Score is a composite score defined as the sum of each of the 7 symptom scores. To allow indirect comparison with previous MF studies, a modified Total Symptom Score (Mesa, 2013) will also be derived from the 6 symptoms considered (night sweats, pruritus, abdominal discomfort, early satiety, pain under ribs on left side, bone or muscle pain).

A copy of the questionnaire is presented in Appendix B.

MF-related symptoms evaluation will be performed by completing the MFSAF version 4.0 version using a 7-day recall period electronically on a tablet at the site at screening, Day 1 of each treatment cycle, at the EOT and the 30-day follow-up visit after last dose of study treatment. If exceptional circumstances preclude the continued administration of measures using planned modalities, then alternate administration methods may be required.

#### 6.3.2. Health-related Quality of Life Assessments and Patient-Reported Outcomes

Note: All adverse events will be reported by the Investigator via the AE modules in electronic data capture (EDC).

#### 6.3.2.1. EORTC QLQ-C30 questionnaire

HRQoL and its various domains will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life C30 questionnaire (EORTC QLQ-C30) version 3 (Aaronson, 1993). The EORTC QLQ-C30 is a validated questionnaire developed to assess the quality of life of cancer patients. It is the most commonly used PRO instrument in oncology studies. It consists of 30 items classified into 15 domains including 5 functional subscales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning); 3 multi-item symptom subscales (fatigue, nausea/vomiting, and pain); a global QOL subscale; and 6 single items addressing various symptoms and perceived financial impact. All EORTC OLO-C30 items use a 4-point Likert scale (ie, "not at all," "a little," "quite a bit," and "very much"), except the 2 items assessing global QOL (item 29 and item 30), which use a 7-point scale. The EORTC QLQ-C30 uses a recall period of one week (Aaronson, 1993; Hjermstad, 1995; King, 1996; Osoba, 1997; Osoba, 1998). The scale scores are linearly transformed to 0 to 100 scores (Aaronson, 1993). Scores vary from 0 (worst) to 100 (best) for the functional dimensions and GHS, and from 0 (best) to 100 (worst) for the symptom dimensions; higher scores indicate better QoL, better functioning, or more severe symptoms, respectively. A copy of the questionnaire is presented in Appendix C.

#### 6.3.2.2. EQ-5D-5L

Health utilities will be assessed using EQ-5D-5L classifier for 5 levels. The instrument contains 5 items that assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and a visual analog scale (VAS) for global

health. US value set will be used to calculate utility indices for cost-effectiveness modeling.

The EQ-5D-5L is a generic, self-administered preference-based measure of health recently introduced by the EuroQol Group based upon the dimensions of the EQ-5D-3L. It is available in 169 languages, with applications in clinical, cost-effectiveness and population health studies, as well as its routine use by health care systems. The 5-level EQ-5D-5L expands the range of responses in each dimension from 3 to 5 levels (Herdman, 2011). Preliminary studies indicated that prototype 5L versions improved upon the properties of the 3L in terms of reduced ceiling effects, increased reliability, and improved ability to discriminate between different levels of health (Janssen, 2008a; Janssen, 2008b).

The five dimensions covered by the EQ-5D-5L include mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has five levels of "severity" corresponding to "no problems", "some problems", and "extreme problems". The instrument provides a simple descriptive HRQoL profile for each participant. Information relating to EQ-5D health states gathered in the context of multinational trials may be converted into a single summary index using one of the available EQ-5D value sets.

The EQ-5D-5L questionnaire also includes a visual analogue scale which records the respondent's self-rated health on a vertical, 0 to 100 scale where 100 = "Best imaginable health state" and 0 = "Worst imaginable health state". This information can be used as a quantitative measure of health outcome as judged by the individual respondents. A copy of the questionnaire is shown in Appendix D.

The EORTC QLQ-C30, EQ-5D-5L, will be completed electronically on a tablet at the site on Day 1 of each treatment cycle, at the EOT and the 30-day follow-up visit after last dose of study treatment. If exceptional circumstances preclude the continued administration of measures using planned modalities, then alternate administration methods may be required.

All these HRQoL-related assessments should be performed before any other assessments are performed by the Investigator or designee during the visit.





## **6.4.** Response Assessment

Response assessments should occur at the end of C3, C6, C12, C18, C24 and at the end of every sixth (6<sup>th</sup>) cycle as applicable afterwards. The response assessment can be combined with the Day 1 visit of the subsequent cycle or End of Treatment visit. The following assessments will be performed:

- Symptoms response assessment: Refer to Section 6.1
- Spleen volume by MRI/CT scan: Refer to Section 6.1
- Spleen size by palpation: Refer to Section 6.1

In case there are signs of progression of the splenomegaly (eg, by palpation) an MRI/CT scan can be performed to confirm at any time during the study.

If a bone marrow assessment is performed as per standard of care, in addition to the assessments described above, the Investigator will assess response, for example, in terms of complete response (CR), partial response (PR), relapse, cytogenetic and molecular response as per IWG-MRT 2013 (Tefferi, 2013).



#### 6.5. Crossover

Subjects in the BAT arm may crossover to receive fedratinib treatment.

One of the following criteria must be fulfilled:

- 1. Subject has completed the End of Cycle 6 response assessment including MRI/CT scan within 28 days before crossover
- 2. Subject has not completed the End of Cycle 6 response assessment but has demonstrated confirmed progression of splenomegaly.

Confirmed progression of splenomegaly is defined as enlargement of spleen volume by MRI/CT scan (within 28 days before crossover) of  $\geq 25\%$  compared to the subject's baseline as assessed by the central imaging laboratory.

Note: In case of suspected progression of splenomegaly, a response assessment can be performed (refer to the Section 6.4) for confirmation of progression at any time. MRI/CT scans must be sent to the designated central imaging review laboratory and marked for expedited processing.

The presence of any of the following will exclude a subject from crossover to fedratinib treatment:

- 1. Any of the following laboratory abnormalities assessed within 28 days before cross-over:
  - Platelets  $< 25 \times 10^9 / L$  or Platelets  $< 50 \times 10^9 / L$  if associated with major bleeding

- Absolute neutrophil count (ANC)  $< 0.5 \times 10^9/L$
- Myeloblasts  $\geq$  5 % in peripheral blood
- Estimated glomerular filtration rate < 30 mL/min/1.73 m² (as per the Modification of Diet in Renal Disease [MDRD] formula) (Appendix K)
- Serum amylase or lipase > 2.0 x ULN
- Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x ULN
- Total bilirubin > 1.5 x ULN, subject's total bilirubin between 1.5 3.0 x ULN are eligible if the direct bilirubin fraction is < 25% of the total bilirubin
- 2. Subject with signs indicating transformation/progression to blast phase of myelofibrosis
- 3. Subject has received ruxolitinib any other JAK inhibitor or hydroxyurea within 14 days prior to crossover
- 4. Subject with thiamine deficiency, defined as thiamine levels in whole blood below normal range according to the central laboratory and not demonstrated to be corrected prior to crossover
- 5. Subject with signs or symptoms of WE (eg, severe ataxia, ocular paralysis or cerebellar signs) without documented exclusion of WE by thiamine level and brain MRI
- 6. Subject with concomitant treatment with or use of pharmaceutical, herbal agents or food known to be strong inducers of Cytochrome P450 3A4 (CYP3A4), sensitive CYP3A4 substrates with narrow therapeutic range, sensitive Cytochrome P450 2C19 (CYP2C19) substrates with narrow therapeutic range, or sensitive Cytochrome P450 2D6 (CYP2D6) substrates with narrow therapeutic range (refer to Section 7 and Appendix L)
- 7. Subject with serious active infection

Eligibility criteria for crossover must be verified by the responsible Investigator. The appropriate documentation may be reviewed by the Sponsor prior to a subject receiving the first fedratinib dose treatment dose.

If the criteria are met, subjects are eligible for assignment to fedratinib treatment via IRT.

Depending on laboratory results, an adjustment of the fedratinib starting dose (eg, for a low glomerular filtration rate [GFR]) may be required.

After crossover subjects will continue in the study following the schedule of assessments beginning with the C1D1 assessments with the exception of PK samples that will not be collected for subject after crossover.

#### 6.6. End of Treatment Visit

The treatment period will be concluded by an End of Treatment (EOT) visit performed for subjects who are withdrawn from the assigned study treatment (except for those subjects crossing over from the BAT arm to the fedratinib treatment) for any reason as soon as possible after the decision to permanently discontinue treatment has been made.

If clinically justified, a subject that needs to discontinue BAT treatment can stay on "no treatment" or symptom directed treatment, until a crossover as described above or at latest till completion of Cycle 6.

At the time study treatment is discontinued all subjects will undergo the End of Treatment assessment. End of Treatment Visit procedures/assessments may not need to be repeated if previously performed within  $\pm 7$  days of EOT visit. If a subject is discontinued during a regular scheduled visit, all EOT procedures should be completed at that visit.

The following assessments will be performed at the EOT visit as specified in the Table of Events (Section 5):

- IRT subject registration for treatment discontinuation
- Concomitant medications and procedures: As detailed in Section 6.1
- Vital signs, Physical exam and weight: As detailed in Section 6.1
- **Electrocardiogram (ECG):** As clinically indicated (detailed in Section 6.1)
- **Hematology:** As detailed in Section 6.1
- **Serum chemistry:** As detailed in Section 6.1
- **Lipid panel:** As detailed in Section 6.1
- Coagulation: As clinically indicated (detailed in Section 6.1)
- Urinalysis: As clinically indicated (detailed in Section 6.1)
- Thiamine level: As detailed in Section 6.1
- Transfusion burden assessment: As detailed in Section 6.3
- Cognitive assessment Mini-Mental State Examination: As clinical indicated (detailed in Section 6.1)
- **Response Assessment:** As detailed in Section 6.4
- Spleen size by palpation: As detailed in Section 6.1
- Spleen volume by MRI/CT scan: Refer to Section 6.1
- Eastern Cooperative Oncology Group (ECOG) performance status: As detailed in Section 6.1
- Adverse events: Refer to Section 6.1
- Accountability of fedratinib treatment
- Risk mitigation for gastrointestinal toxicity & Encephalopathy, including Wernicke's: Refer to Section 7.4 and Section 7.5.
- Symptoms response assessment: as detailed in Section 6.3

• Health-related Quality of Life Assessments and Patient-Reported Outcomes: as detailed in Section 6.3

## 6.7. 30-Day Follow-up After Last Dose Visit

All subjects will be followed for 30 days after the last dose of study treatment for AE reporting, as well as any SAEs made known to the Investigator at any time thereafter that are suspected of being related to study treatment, as described in Section 10.1.

The following will be performed as specified in the Table of Events (Section 5, Table 3):

- **Pregnancy testing**: As detailed in Section 6.1
- Concomitant medications and procedures: As detailed in Section 6.1
- Vital signs, Physical exam and weight: As detailed in Section 6.1
- Electrocardiogram (ECG): As clinically indicated (detailed in Section 6.1)
- **Hematology:** As detailed in Section 6.1
- **Serum chemistry:** As detailed in Section 6.1
- **Coagulation:** As clinically indicated (detailed in Section 6.1)
- Urinalysis: As clinically indicated (detailed in Section 6.1)
- Thiamine level: As clinically indicated (detailed in Section 6.1)
- Transfusion burden assessment: As detailed in Section 6.3
- **Survival:** Refer to Section 6.8
- Progression of myelofibrosis to acute myeloid leukemia (AML) assessment: Refer to Section 6.8
- Subsequent therapies for disease under study: Refer to Section 6.8
- **Spleen size by palpation:** As detailed in Section 6.1
- Eastern Cooperative Oncology Group (ECOG) performance status: As detailed in Section 6.1
- Adverse events: Refer to Section 6.1
- Risk mitigation for gastrointestinal toxicity & Encephalopathy, including Wernicke's: Refer to Section 7.4 and Section 7.5.
- **Symptoms response:** as detailed in Section 6.3
- Health-related Quality of Life Assessments and Patient-Reported Outcomes: as detailed in Section 6.3

## **6.8.** Survival Follow-up

All subjects discontinued from protocol-prescribed therapy for any reason will be followed for survival, subsequent therapies, new malignancy and progression of myelofibrosis to acute

myeloid leukemia (AML) every 3 months for at least 36 months from the first dose of study medication, or until death, lost to follow-up, withdrawal of consent for further data collection, or study closure, whichever comes first.

A window of  $\pm$  14 days is allowed for post treatment survival follow-up assessments; the visits should be performed every 3 months  $\pm$  14 days and can be done by a documented telephone contact between site and subject.

#### 6.9. Unscheduled Assessments or Visits

Should it become necessary to repeat an evaluation (eg, laboratory tests, vital signs, etc.) outside of scheduled study visits, or to perform additional evaluations than the ones described in the current protocol, the results of these additional evaluations should be recorded in an unscheduled visit CRF pages(s). These evaluations should also appear in the subject's chart and/or other source documentation.

In the event that immediate hematology / biochemistry / urinalysis / coagulation / thiamine values are needed for clinical decisions, local laboratory results may be used pending the outcome of the central laboratory assessment. However, matching samples must always be sent to the central laboratory and clinical decisions and assessments must be reconciled with the results of the central laboratory. The results of these additional analyses will be recorded in the subjects' CRF as applicable as described in Section 10.

#### 7. DESCRIPTION OF STUDY TREATMENT

## 7.1. Description of Investigational Product

The Sponsor will supply fedratinib 100 mg capsules in high density polyethylene (HDPE) bottles for oral administration and will be labeled appropriately as Investigational Product for this study.

The study drug must be kept at the temperature condition as specified on the label. Fedratinib must be stored at temperatures below 30°C.

Other recommended/required concomitant medications per the protocol will be provided by the local site. The Sponsor will not provide these medications.

## 7.2. Best Available Therapy Regimens

BAT will be provided by the local site.

Best available therapy regimen (BAT) may include any Investigator-selected treatment and is not limited to approved JAK inhibitors (used according to the prescribing information), chemotherapy (eg, hydroxyurea), anagrelide, corticosteroid, hematopoietic growth factor, immunomodulating agent, androgens, interferon, and may also include "no treatment" and symptom directed treatment. BAT may not include investigational agents, fedratinib (if approved during the course of the study) and hematopoietic stem cell transplantation.

#### 7.3. Treatment Administration and Schedule

Fedratinib will be dispensed to subjects using the IRT system. The fedratinib dose is 400 mg/day PO (4 x 100 mg capsules) to be self-administered orally once daily continuously on an outpatient basis, preferably together with an evening meal, the same time each day. In case a dose is missed, the next dose should be taken the following day at the same time of day as previously taken before the dose was missed.

A flexible dose modification regimen may be employed to minimize drug toxicity for individual subjects, with possible daily doses of 200 mg, 300 mg, or 400 mg. For subjects with severe impairment of renal function and co-administration of strong or moderate CYP3A4 inhibitors, the fedratinib dose is adjusted (Refer to Section 7.3.2 and Section 7.3.3).

For administrative purposes cycles are defined as 4-week (28-day) periods irrespective of the assigned treatment arm. Subjects may continue treatment with fedratinib or BAT until one of the conditions described in the "Treatment Period" section of Section 3.1 occurs.

Subjects treated on the BAT arm will be treated according to local prescribing information.

#### **7.3.1.** Dose Modification for Toxicity

Management of the BAT will be performed in line with prescribing information and as per the Investigator's discretion as per the local standard of care.

The section below describes the dose management for fedratinib only.

The most common adverse events associated with fedratinib are hematological and gastrointestinal events. Hematological adverse events associated with JAK inhibitors are dose

dependent, mechanism-based and are managed through dose reductions, dose interruptions and transfusions.

The Fedratinib Dose Modification Schedule (Table 4) should only be used for adverse events considered drug-related by the investigator and cannot be attributed to an identifiable cause such as underlying illness or disease progression, other concurrent illness, or concomitant medication.

If a subject experiences a drug toxicity as specified in the table below, the dosing must be interrupted; in some cases (ie, when it is not a liver function test (LFT) abnormality) the dose can be titrated by a 100 mg/day decrement during the study, depending upon the Investigator's judgment, down to a minimum dose of 200 mg/day. For subjects with co-administration of strong or moderate CYP3A4 inhibitors and severe impairment of renal function the fedratinib dose is adjusted (Refer to Section 7.3.2 and Section 7.3.3). In addition, if a subject experiences a dose interruption of fedratinib for more than 28 consecutive days, consultation with the medical monitor is required to determine if study treatment may resume.

If a subject does not tolerate fedratinib therapy after 2 dose level reductions from the starting dose, he/she must be withdrawn from the study treatment. If the toxicity does not resolve in the time period as specified in the table below subjects must be withdrawn from the study treatment. Re-escalation of doses is possible in certain cases. The daily dose of fedratinib cannot exceed 400 mg/day.

**Table 4: Fedratinib Dose Modification Schedule** 

| Adverse Event | Fedratinib<br>Management | Recovery | Fedratinib Dose After<br>Recovery |
|---|---|---|---|
| Hematological | | | |
| Grade 4 or Grade 3<br>thrombocytopenia<br>with major bleeding | Hold fedratinib up to 28 days | Grade ≤ 3 thrombocytopenia without bleeding | Dose decrement by 1 dose level: 100 mg daily decrease |
| Grade 4 neutropenia | Hold fedratinib up to 28 days | Grade ≤ 2 neutropenia | Dose decrement by 1 dose level: 100 mg daily decrease |
| Grade 4 hematological toxicity with dose reduction in subsequent cycle | - | Toxicity resolves for at least 1 cycle | Subsequent upward dose<br>titration possible of 1 dose<br>level (100 mg daily) per cycle<br>as per the Investigator's<br>discretion |
| Recurrence of a Grade<br>4 hematological | | | Subsequent upward dose titration not permitted |
| toxicity | - | - | Fedratinib discontinuation as per the Investigator's discretion |
| Non-hematological | | | |
| Drug-related non-<br>hematological Grade 4<br>or unmanageable<br>Grade 3 toxicity with<br>dose reduction in<br>subsequent cycle | - | - | Subsequent upward dose titration not permitted Fedratinib discontinuation as per the Investigator's discretion |
| Hepatic (LFT abnorm | alities) | | |
| Grade ≥ 3 AST or ALT or total bilirubin | Hold fedratinib Weekly monitoring of LFTs, until resolution After fedratinib resumed, LFT monitoring every 2 weeks for the 3 subsequent cycles at a minimum | Grade ≤ 1 | Fedratinib Hold ≤ 14 days: Dose decrement by 1 dose level: 100 mg daily decrease, Subsequent upward dose titration not permitted Fedratinib Hold > 14 days (AE did not return to Grade ≤ 1): Fedratinib permanently discontinued Grade 4 in the absence of demonstrable cause: permanently discontinue fedratinib |

**Table 4:** Fedratinib Dose Modification Schedule (Continued)

| Adverse Event | Fedratinib<br>Management | Recovery | Fedratinib Dose After<br>Recovery |
|---|---|---|---|
| Recurrence of LFT abnormality (ie, ≥ Grade 3 toxicity) after dose reduction | Discontinue fedratinib permanently | - | - |
| Gastrointestinal | | | |
| Grade 2 nausea, vomiting, diarrhea, or constipation that does not respond to adequate therapeutic or supportive measures within 48 hours | Hold fedratinib<br>up to 14 days | Toxicity resolves to Grade ≤ 1 | Consider resuming the dose at the same level after resolution of adverse event (see section on management of GI toxicity) |
| Grade ≥ 3 or recurrence of Grade 2 nausea vomiting, diarrhea, or constipation that does not respond to adequate therapeutic or supportive measures within 48 hours | Hold fedratinib<br>up to 14 days | Toxicity resolves to Grade ≤ 1 | Consider reducing one dose level after resolution of adverse event (see section on management of GI toxicity below) |
| Other Adverse Events Not Describ | oed Above | | |
| Grade ≥ 3 or recurrence of Grade 2 that does not respond to adequate therapeutic or supportive measures within 48 hours | Hold fedratinib<br>up to 14 days | Toxicity resolves to Grade ≤ 1 | Consider reducing one dose level after resolution of adverse event |
| Grade $\geq 3$ non-hematological toxicity, non-gastrointestinal toxicity or Grade $\geq 2$ peripheral neuropathies | Hold fedratinib<br>up to 14 days | Toxicity resolved to Grade ≤ 1 | Dose decrement by 1 dose level: 100 mg daily decrease |
| In case of a potential case of Encephalopathy, including Wernicke's refer to Section 7.5, Management of Encephalopathy, including Wernicke's | | | |

Encephalopathy, including Wernicke's.

AE = adverse event; ALT = alanine aminotransferase; AST = aspartate aminotransferase; GI = gastrointestinal; LFT = liver function test.

## 7.3.2. Dose Adjustment for Co-administration of Fedratinib with Strong CYP3A4 Inhibitors

Concomitant administration of fedratinib with strong CYP3A4 inhibitors increase fedratinib exposure. Increased fedratinib exposure may increase the risk of AEs. In place of strong CYP3A4 inhibitors, consider alternative therapies that do not strongly inhibit CYP3A4 activity. If strong CYP3A4 inhibitors cannot be replaced, reduce fedratinib dose to 200 mg when administering with strong CYP3A4 inhibitors, (eg, ketoconazole, ritonavir; refer to Appendix L). Additional dose adjustments (decrease or increase of the daily dose) should be made with monitoring of fedratinib-related safety (see Section 7.3.1) and efficacy.

In cases where co-administration with a strong CYP3A4 inhibitor is discontinued, the fedratinib dose should be increased to 300 mg daily during the first two weeks after discontinuation of the

CYP3A4 inhibitor, and then to 400 mg daily thereafter as tolerated. Additional dose adjustments should be made as needed based upon frequent monitoring of safety.

In all the situations above, please contact the Sponsor medical monitor for any question or guidance.

#### 7.3.3. Dose Adjustment for Renal Impairment

No modification of the starting dose is recommended for patients with mild to moderate renal impairment. Due to potential increase of fedratinib exposure, patients with pre-existing moderate renal impairment require more intensive safety monitoring, and if necessary, dose modifications based on adverse reactions.

In subjects that develop severe renal impairment during the study the fedratinib dose should be adjusted by two dose decrement levels (eg, from 400 mg to 200 mg once a day [QD]).

Clinical signs and symptoms for efficacy and fedratinib-related AEs should be monitored and the dose of fedratinib should be further adjusted as necessary.

## 7.4. Overview on Management of Gastrointestinal Adverse Events

Gastrointestinal adverse events, specifically nausea, vomiting and diarrhea, are commonly associated with fedratinib treatment and require multifaceted management using dose adjustment, active treatment or prophylaxis with anti-emetics, and monitoring. GI symptoms generally start in the first treatment cycle but typically improve within 6-8 weeks on fedratinib treatment.

## 7.4.1. Management of Nausea and Vomiting

Management of nausea and vomiting during treatment with fedratinib will be done according to the following steps:

- Subjects will be provided management instructions (including when to contact the study site) before the start of treatment
- In order to mitigate for nausea and vomiting events, it is recommended to take fedratinib with food during an evening meal. Specific instructions for fedratinib administration will be provided for PK sampling days (C1D1, the day before C2D1 and C2D1)
- It is highly recommended to use anti-nausea/vomiting treatment prophylactically according to local practice for the first 8 weeks of treatment (eg, ondansetron). If dimenhydrinate or other muscarinic receptor antagonists are used for nausea and vomiting, administer these agents in the evening to minimize drowsiness and other potential neurological AEs
- Hold / reduce the dose of fedratinib according to Table 4
- Hospitalization may be indicated for Grade 3 or higher nausea or vomiting or events that persist

• For medications that are administered for prophylactic use of nausea and vomiting, if no clinically significant nausea and vomiting occurs during the first 8 weeks of fedratinib treatment, consider weaning the subject off these medications

## 7.4.2. Management of Diarrhea

Management of diarrhea during treatment with fedratinib will be done according to the following steps:

- Subjects should have loperamide available at home and should be provided with diarrhea management instructions (including when to contact the study site) before the start of treatment
- Loperamide should not be given as prevention in case the subject does not experience diarrhea
- Treat with loperamide as per local practice at the onset of diarrhea. Consider starting loperamide at a 4 mg loading dose and then 2 mg after each diarrheal bowel movement without exceeding 16 mg/24 hours
- Dietary modifications including adequate hydration, avoidance of lactose-containing foods and alcohol, small meals with rice, bananas, bread, etc
- Hold / reduce the dose of fedratinib according to Table 4
- Hospitalization may be indicated for Grade 3 or higher persisting diarrhea.
- Management of nausea, vomiting and diarrhea will be assessed during the subject's visit on Day 1 of every following 28-day cycle, at Day 15 of the first three cycles and by a mandatory telephone contact at Day 8 of the first cycle.

## 7.5. Management of Encephalopathy, including Wernicke's

A potential case of Encephalopathy, including Wernicke's is a medical emergency. Screening for Encephalopathy, including Wernicke's and management of cases during treatment with fedratinib will be done according the following steps:

#### 7.5.1. Clinical and Cognitive Assessment

Interval history: including a review of the subject's history for confusion, memory problems, vision problems (eg, double vision) as well as poor nutrition, signs and symptoms of malabsorption, and alcohol use

- Physical examination: including assessment for abnormal eye movements, cerebellar abnormalities and body weight (weight loss compared to previous examination or patient history) during screening and Day 1 of every treatment cycle, at the End of Treatment (EOT), and the 30-Day Follow-up visit
- Mini-Mental State Examination (MMSE): to objectively assess for signs/symptoms of encephalopathy during screening, on Day 1 of Cycles 2 and 3 and every third cycle thereafter, at the End of Treatment Visit and more frequently as clinically indicated

#### 7.5.2. Management of Encephalopathy, including Wernicke's

In case of signs or symptoms that may indicate Encephalopathy, including Wernicke's:

- Hold study medication until Encephalopathy, including Wernicke's is ruled out
- Obtain sample for thiamine level
- Start parenteral thiamine as described in Section 7.5.3 for subjects with thiamine levels < 30 nM/L regardless of thiamine level
- Report the event as an AESI to the Sponsor
- Obtain a neurological consult
- Perform a brain MRI
- If WE is confirmed, discontinue fedratinib permanently
- If WE is ruled out, assess for other causes of encephalopathy and treat accordingly. Once resolved, consider restarting treatment with fedratinib after discussion with study monitor.

#### 7.5.3. Thiamine, Supplementation, Monitoring and Correction

All subjects receiving study medication will receive thiamine supplementation. Start oral thiamine supplementation at a minimum daily dose of 100 mg (or equivalent) at Cycle 1 Day 1. Continue supplementation throughout the treatment period until study medication is discontinued, and through the 30-day follow-up visits.

Thiamine levels (for whole blood) will be monitored in all subjects.

- Thiamine levels are assessed at screening and need to be corrected and retested before starting fedratinib treatment (see inclusion criteria)
- While on treatment with study medication, thiamine levels are assessed in a fasting state at start of Cycles 1, 2, 3 and every third cycle thereafter, at the End of Treatment Visit and as clinically indicated
- In case of documented thiamine deficiency and a subject is receiving thiamine supplementation, while on study:
  - Thiamine levels should be assessed in a fasting state and thiamine supplementation should be given after the blood draw
  - If the subject develops signs or symptoms suggestive of encephalopathy including Wernicke's, please follow instructions in Section 7.5.2
  - For thiamine levels below normal range but > 30 nM/L without signs or symptoms of WE while receiving thiamine supplementation:
    - The site should contact the Medical Monitor regarding the low thiamine level as soon as possible
    - Report the event as an Adverse Event of Special Interest (AESI) to the Sponsor.

- Consider increasing the dose of oral thiamine supplementation to twice the daily dose (if the subject is taking 100 mg, increase to 200 mg)
- o Monitor thiamine level closely (monthly at least) and adjust dose as needed
- For thiamine level < 30 nM/L **without signs or symptoms** of WE while receiving thiamine supplementation:
  - The site should contact the Medical Monitor regarding the low thiamine level as soon as possible
  - Report the event as an Adverse Event of Special Interest (AESI) to the Sponsor.
  - Study medication must be held until thiamine levels are restored to normal range.
  - o Immediate treatment with IV thiamine (stop oral thiamine), at therapeutic dosages eg, 500 mg IV infused over 30 minutes 3 times daily for 2 to 3 days or alternatively IM in equivalent doses according to local standard of care
  - This will be followed by 250 mg to 500 mg IV thiamine infused once a day for 3 to 5 days or alternatively IM in equivalent doses according to local standard of care
  - And then consider increasing the dose of oral thiamine supplementation to twice the previous daily dose (for example if the subject is taking 100 mg, increase the dose to 200 mg)
  - Monitor thiamine levels closely (at least monthly) and adjust the dose as needed
- Thiamine supplementation should be administered as a thiamine only formulation.
- If thiamine levels are low, ensure that magnesium levels are normal or corrected if low

## 7.6. Method of Treatment Assignment

Randomization and treatment assignment will occur at the end of the Screening Period, once all the required screening procedures have been completed and all required data have been submitted to the Sponsor or its authorized representative. Upon receiving acknowledgment of subject's eligibility review from the Sponsor or its authorized representative, the subject can be assigned fedratinib treatment using an IRT built for this study.

Designated research personnel at each investigational site will be assigned unique, password-protected user accounts which give them the authorization to utilize the IRT to enroll subjects.

## 7.7. Packaging and Labeling

Sections 7.7, 7.8 and 7.9, only apply to fedratinib.

The label(s) for fedratinib will include Sponsor name, address and telephone number, the protocol number, fedratinib name, dosage form and strength (where applicable), amount of

fedratinib per container, lot number, expiry date (where applicable), fedratinib identification/kit number, dosing instructions, storage conditions, and required caution statements and/or regulatory statements as applicable. Additional information may be included on the label as applicable per local regulations.

## 7.8. Investigational Product Accountability and Disposal

Sponsor (or designee) will review with the Investigator and relevant site personnel the process for Investigational Product return, disposal, and/or destruction including responsibilities for the site versus Sponsor (or designee).

## 7.9. Investigational Product Compliance

Fedratinib will be administered by the study site personnel in the clinic on PK sampling days. Subjects will self-administer all other fedratinib doses in the treatment period. Study site personnel will review the dosing information with the subject (or legally authorized representative) on scheduled clinic visit days. Subjects (or legally authorized representative) will be asked to bring all unused capsules with them to scheduled clinic visits (ie, prior to the start of the next treatment cycle). Study site personnel will perform a fedratinib administration compliance check and record this information in the subject's source documentation.

Administration of all fedratinib will be recorded including dispensing, dosing and any changes in dosage administration such as interruption or reduction in dosing due to an AE.

#### 8. CONCOMITANT MEDICATIONS AND PROCEDURES

Over the course of this study, additional medications may be required to manage aspects of the disease state of the subjects, including side effects from trial treatments or disease progression. Supportive care, such as anti-emetic medications, may be administered at the discretion of the Investigator.

All prior/concomitant medications including, prescription, over-the-counter, and herbal preparations taken for any indication used from 28 days prior to randomization until 30 days after the last dose of fedratinib/BAT during the study must be reported on the eCRF. The type, dose route, start and end date of administration must be documented on the appropriate pages of the electronic case report form (eCRF).

BAT is regarded to be the study treatment and not a concomitant treatment and will be documented separately on the appropriate pages of the eCRF.

The details of the prior treatment with ruxolitinib and its outcomes will also be recorded in the subject's eCRF regardless of treatment discontinuation/procedure date.

Information regarding transfusion history (at least 84 days prior to and including the randomization date), including pretransfusion hemoglobin (Hgb) levels, number of units transfused and dates of transfusions, will be collected and reported in the appropriate eCRF

For information regarding other drugs that may interact with fedratinib and affect its metabolism, pharmacokinetics, or excretion, please also see the Investigator's Brochure.

#### 8.1. Permitted Concomitant Medications and Procedures

Prophylaxis and/or treatment of gastrointestinal adverse events, specifically nausea, vomiting and diarrhea (eg, loperamide) is an essential part of management of potential fedratinib toxicity. (Refer to Section 7.4).

Subjects are required to take daily thiamine supplementation (Refer to Section 7.5).

Blood product support (RBCs and platelet transfusions) may be administered according to institutional standards.

Subjects may be administered supportive and palliative care (eg, pain control) as clinically indicated throughout the study.

Prior anticancer treatments should be recorded on the appropriate eCRF(s) regardless of treatment discontinuation/procedure date.

For information regarding clinically relevant P450 inducers, inhibitors, substrates, and transporter substrates refer to Section 8.3.

#### **8.2.** Prohibited Concomitant Medications

The following concomitant medications are specifically excluded during the course of the study for subjects randomized to the fedratinib arm or for subjects that crossover to fedratinib treatment:

- Cytotoxic, chemotherapeutic, targeted or investigational agents/therapies
- Immunomodulatory drug therapy (eg, thalidomide)
- Immunosuppressive therapy
- Systemic corticosteroids > 10 mg/day prednisone or equivalent
- Hydroxyurea
- Interferon-alpha
- Anagrelide
- JAK inhibitors other than fedratinib
- Aspirin at doses > 150 mg daily
- Any investigational agent

For information regarding clinically relevant P450 inducers, inhibitors, substrates, and transporter substrates refer to Section 8.3.

For subjects on the BAT arm not crossing over to fedratinib, fedratinib is specifically excluded during the study. Additional treatments might be prohibited according to BAT prescribing information

If a subject requires treatment with any new medications that are specifically excluded, the subject may need to be discontinued from treatment. The Investigator should consult the medical monitor regarding any questions about whether a new medication or dosage of existing medication would require the subject to discontinue from the study.

# 8.3. Clinically Relevant Cytochrome P450 Inducers, Inhibitors, Substrates, and Transporter Substrates

Fedratinib is metabolized by multiple cytochrome P450 enzymes (CYPs) in vitro, with prominent contribution from CYP3A4 and with a lesser contribution from CYP2C19.

#### CYP3A4 inducers and inhibitors

Strong and moderate CYP3A4 inducers (see Appendix L) that may decrease fedratinib plasma concentrations are not permitted while receiving fedratinib.

Strong CYP3A4 inhibitors (see Appendix L) increase fedratinib plasma concentrations. In place of strong CYP3A4 inhibitors, alternative therapies that do not inhibit CYP3A4 need to be considered. If strong CYP3A4 inhibitors cannot be replaced, the strong CYP3A4 inhibitor needs to be used with caution and the fedratinib dose needs to be adjusted (refer to Section 7.3.2).

#### **Dual CYP2C19 and CYP3A4 inhibitors**

Dual inhibitors of CYP2C19 and CYP3A4 (eg, fluconazole, fluvoxamine) that may increase fedratinib plasma concentrations are not permitted while receiving fedratinib.

Sensitive Substrates: Effect of fedratinib on plasma levels of other co-administered drugs (drugs metabolized by CYP3A4, CYP2C19, and CYP2D6):

Co-administration of fedratinib with drugs that are CYP3A4 substrates (eg, midazolam), CYP2C19 substrates (eg, omeprazole), or CYP2D6 substrates (eg, metoprolol) increase the area under the curve from time zero to infinity (AUCinf) of these drugs by 4-, 3-, and 2-fold, respectively, which may increase the risk of adverse reactions of these drugs. Monitor for adverse reactions and adjust the dose of drugs that are CYP3A4, CYP2C19, or CYP2D6 substrates (see Appendix L) as necessary when co-administering with fedratinib.

Transporters: Effect of fedratinib on plasma levels of other co-administered drugs (drugs transported by P-gp, BCRP, MATE-1, MATE-2K, OATP1B1/1B3, and OCT1/2):

Fedratinib can increase plasma levels of drugs that are substrates of transporters, P-gp, BCRP, MATE-1, MATE-2K, OATP1B1/1B3, and OCT1/2. Fedratinib should be used with caution with drugs that are substrates of these transporters (see Appendix L), and dose modifications of substrates of these transporters should be made, as necessary, with monitoring of safety and efficacy.

A list of clinically relevant P450 inducers and inhibitors as well as substrates, and transporter substrates can be found in Appendix L.

#### 9. STATISTICAL CONSIDERATIONS

#### 9.1. Overview

This is a multicenter, open-label, randomized study to evaluate the efficacy and safety of fedratinib compared to best available therapy in subjects previously treated with ruxolitinib and with DIPSS-intermediate-2 or high-risk primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis.

The sections below provide an overview of the proposed statistical considerations and analyses. The final statistical analysis methods will be documented in detail in the statistical analysis plan (SAP).

#### **General Considerations**

A descriptive summary for continuous data will include the number of non-missing observations (n), mean, standard deviation, median, minimum and maximum. In addition, 25% percentile and 75th percentile may be provided if needed.

Categorical data will be summarized using counts (n) and percentages (%). The number of subjects with missing data may be displayed but will not be included in the denominator for the calculation of percentages unless otherwise specified.

Unless otherwise specified, baseline value is defined as the last value or measurement taken prior to the first dose in the study. For crossover subjects, baseline for records after crossover is defined as last value prior to or on the same day of crossover.

For crossover subjects in BAT arm, only data before crossover will be included in the analysis where comparison between fedratinib and BAT is intended. The data after crossover will be summarized separately.

#### **Hierarchical Testing on Key Efficacy Endpoints**

The primary and key secondary efficacy endpoints are listed in Section 2. This study employs multiple testing. A fixed sequence procedure with the following sequence order is planned to maintain a familywise error rate of 2.5% (1-sided):

- 1. Spleen volume response rate by MRI or CT scan  $\geq$  35% reduction (RR),
- 2. Symptoms response rate (SRR),
- 3. Spleen volume response rate by MRI or CT scan  $\geq$  25% reduction (RR25).

## 9.2. Study Population Definitions

**Intent to Treat (ITT) population**: this population will consist of all subjects who were randomized. This is the primary analysis population for efficacy variables. All analyses using this population will be based on the treatment assigned by Interactive Response Technology (IRT).

**Per Protocol population:** this population consists of all randomized subjects who received at least one dose of study medication, had no important violation to the inclusion/exclusion criteria and had no other important protocol deviation that could have an impact on efficacy outcome. A list of important protocol deviations which could have an impact on efficacy outcome will be
detailed in the statistical analysis plan. Subjects in this population will be analyzed according to the actual treatment received. This population will be used as the sensitivity analysis for the primary and selected secondary efficacy variables.

**Symptom evaluable population**: this population is a subset of ITT population subjects who have been treated and have evaluable symptom assessments (ie, non-zero total symptom score) at baseline and at least one post baseline. This population will be used as a sensitivity analysis for symptom response rate.

**Safety population**: this population will consist of all randomized subjects who were administered at least one dose of study medication. This population will be used for the safety analyses as well as for the analyses of exposure and safety data before crossover. All analyses using this population will be based on the treatment received.

**Crossover efficacy population**: this population will consist of all subjects from the BAT arm who crossover to fedratinib arm. This population will be used for the analyses of efficacy data after crossover date.

**Crossover safety population**: this population will consist of all subjects from the BAT arm who crossover to fedratinib arm and received at least one dose of fedratinib. This population will be used for the analyses of exposure and safety data after the crossover date.

**HRQoL-evaluable population**: this population will include all randomized subjects who had an evaluable assessment of a given PRO/HRQoL measure at baseline and at least one evaluable assessment of a given PRO/HRQoL measure post-baseline.



# 9.3. Sample Size Consideration

The primary objective is to compare the spleen volume reduction at the End of Cycle 6 in subjects who received fedratinib and subjects who received BAT. The primary endpoint is spleen volume response rate (RR), which is defined as the proportion of subjects whose spleen volume reduction at the end of Cycle 6 from baseline ≥ 35%.

The hypothesis is following:

$$H_0: RR_{FEDA} \leq RR_{BAT}$$
versus
 $H_a: RR_{FEDA} > RR_{BAT}$ 

In the Jakarta 2 study, the reported RR of fedratinib is approximately 35% for the per protocol population. With the assumption of a 20% drop-out rate, the RR would be 28% based on the ITT population. Assuming a true ITT RR (considering drop-outs) in the BAT arm of 10%, 192 subjects will yield approximately 90% power at a one-sided significance level of 0.025.

For the symptom response rate, the Jakarta 2 study reported 27% for the target population. In the BAT arm, 6% and 15% were reported from the SIMPLIFY-2 and PERSIST-2 trials, respectively

(Harrison, 2018b; Mascarenhas, 2018). Assuming the response rate at end of cycle 6 is 10% in the BAT arm (average of historical information) and 27% in the fedratinib arm, 192 subjects will provide 88% power at a one-sided significance level of 0.025.

## 9.4. Background and Demographic Characteristics

#### 9.4.1. Demographic and Baseline Characteristics

Standard demographic and baseline characteristics (including age and race), medical history, cancer diagnosis and prior anti-cancer therapy will be collected at baseline. Baseline efficacy variables and other prognostic variables will be assessed as well. The details of previous ruxolitinib treatment (eg, dose, best response, duration of response) will be summarized.

These parameters will be summarized on the ITT population and will be analyzed in the treatment group to which they were randomized. Analyses for the safety population will be included if the size of any treatment group in the safety population differs (>10%) from the size of that in the ITT population.

#### 9.4.2. Prior or Concomitant Medications

The prior and concomitant medications will be presented for the ITT population.

Medications will be summarized by treatment group according to the WHO drug dictionary, considering the first digit of the anatomical therapeutic chemical (ATC) class (anatomic category) and the first three digits of the ATC class (therapeutic category). All ATC codes corresponding to a medication will be summarized. Subjects will be counted for each of the ATC categories (anatomic or therapeutic) linked to the medication.

## 9.5. Subject Disposition

Subject disposition (analysis population allocation, entered, discontinued, along with primary reason for discontinuation) will be summarized using frequency and percentage.

# 9.6. Extent of Study Treatment Exposure and Compliance

Extent of exposure will be assessed within the safety population. Summary of dose information will be separated for the fedratinib arm and the BAT arm.

Dose information for fedratinib arm will be assessed by the following variables:

- Duration of treatment exposure is defined as: last fedratinib dose date first fedratinib dose date regardless of unplanned intermittent discontinuations
- The cumulative dose is the sum of all fedratinib doses
- The actual dose intensity is defined as the cumulative dose divided by the duration of fedratinib exposure in terms of the number of weeks on study
- The relative dose intensity is defined as the ratio of the actual dose intensity to the planned dose intensity. The planned dose intensity is defined as the planned fedratinib dose for each cycle divided by planned cycle length in weeks
- Dose reduction and reason for dose reduction

## • Dose interruption / delays

The number of subjects treated, number of cycles administered, duration of dosing (weeks), cumulative dose (mg), dose intensity (mg/week), and relative dose intensity (%) will be summarized. Dose interruption / delays and dose reductions will also be analyzed.

Given determination of BAT for a subject will be made by the Investigator, summary of dose information for BAT arm will be limited to type and frequency of medications in BAT arm. If one medication is prevalent in BAT arm (eg, 50% subjects in BAT arm take the same medication), a detailed summary for that medication will be conducted using the same variables listed above. For crossover subjects, only exposure data prior to crossover will be included.

For subjects in BAT arm who crossover to fedratinib, dose information for fedratinib after crossover will be summarized in the same way as in fedratinib arm, based on crossover safety population.

## 9.7. Efficacy Analysis

## 9.7.1. Spleen Volume Response Rate (35%) by MRI / CT (RR)

The primary analysis for spleen volume response rate by MRI/CT will be based on ITT population. The data cut-off for RR will occur when the last randomized subject has completed 6 cycles of fedratinib or BAT. Subjects with a missing MRI/CT spleen volume at the end of cycle 6, including those who meet the criteria for progression of splenomegaly before end of cycle 6, will be considered non-responders. For crossover subjects, only data before crossover will be included.

A Cochran-Mantel-Haenszel (CMH) test to adjust for planned stratification factors (spleen size by palpation, platelet counts and refractory/relapsed or intolerance to ruxolitinib treatment) will be performed to compare fedratinib to BAT at a one-sided 2.5% alpha level. The RRs and 95% confidence intervals (CI) will be provided for each arm as well as for the difference in RRs and 95% confidence interval of the difference for fedratinib to BAT. In addition, a descriptive summary of spleen volume measurements and percentage change from baseline will be provided.

Sensitivity analyses for RR will be pre-planned and details will be documented in the SAP.

#### 9.7.2. Symptom Response Rate (SRR)

The SRR is a key secondary endpoint and is defined as the proportion of subjects with  $\geq 50\%$  reduction from baseline to the end of Cycle 6 in total symptom score (TSS) measured by MFSAF version 4.0. (Total symptom score is defined in Section 9.9.1). Subjects with a missing TSS at the end of cycle 6 or who had disease progression before the end of the cycle 6 will be considered non-responders. The primary analysis of SRR will be conducted using ITT population with non-zero baseline TSS, and sensitivity analyses will be performed using symptom evaluable population.

For subjects crossing over before the End of Cycle 6 assessment, only data before the crossover date will be included for the comparison with the fedratinib arm.

A CMH test to adjust for planned stratification factors (spleen size by palpation, platelet counts and refractory/relapsed or intolerance to ruxolitinib treatment) will be performed to compare

fedratinib to BAT at a one-sided 2.5% alpha level. The proportions and 95% CIs will be provided for each arm as well as for the difference in proportions and 95% CI of the difference for fedratinib to BAT.

Additional sensitivity analyses will be pre-planned for SRR and will be documented in the SAP.

For crossover subjects, the SRR during the fedratinib period will be summarized separately using the same method as described above. No formal statistical testing will be conducted to compare with BAT. The analysis will be based on the crossover efficacy population with evaluable TSS at the time of crossover.

## 9.7.3. Spleen Volume Response Rate (25%) by MRI / CT (RR25)

The proportion of subjects who have  $\geq 25\%$  reduction in spleen volume at the end of cycle 6 (RR25) is a key secondary endpoint and will be summarized using the same method as RR. Subjects with a missing MRI/CT spleen volume at the end of cycle 6 including those who meet the criteria for progression of splenomegaly before the end of cycle 6 will be considered non-responders. For crossover subjects, only data before crossover will be included.

The analysis will be conducted using ITT and Per Protocol population.

## 9.7.4. Spleen Response Rate by Palpation (RRP)

Spleen response rate by palpation is the proportion of subjects with a spleen response according to the IWG-MRT 2013 (Appendix O) at the end of cycle 6 as compared to baseline. This will be calculated for subjects that have an enlarged spleen ( $\geq 5$  cm below LCM) at baseline. Subjects with a missing spleen size assessment at the end of cycle 6 including those who meet the criteria for progression of splenomegaly before end of cycle 6 will be considered not to be responders. The RR by palpation and 95% CI will be provided for each arm as well as for the difference and 95% CI of the difference for fedratinib to BAT.

The analysis will be conducted based on a subgroup of the ITT population where subjects with baseline spleen size < 5 cm below LCM are excluded (ie, not eligible for spleen response).

## 9.7.5. Durability of Spleen Volume Response by MRI/CT (DR)

Durability of spleen volume response (DR) by MRI/CT is defined as the date from the first documented spleen response (ie,  $\geq$  35% reduction in spleen volume) to the date of subsequent progressive disease (PD) in spleen volume per the IWG-MRT 2013 criteria or death, whichever is earlier. In the absence of an event before the analysis is performed, the DR will be censored at the date of the last valid assessment performed before the analysis performed date.

Duration of spleen volume response by MRI/CT scan will be analyzed using the Kaplan-Meier (K-M) method. Kaplan-Meier estimates of the 25th, 50th, and 75th percentiles and the 95% confidence interval of median will be provided for both fedratinib and BAT arms. Kaplan-Meier curves will be plotted.

The analysis will be conducted based on a subgroup of the ITT population where subjects have achieved  $\geq 35\%$  SVR at any time during treatment. An additional analysis will be performed on a population including subjects who have  $\geq 35\%$  SVR at end of cycle 6 only.

## 9.7.6. Spleen and Disease Progression Free Survival (SDPFS)

Spleen and disease progression free survival is defined as the time from randomization to death due to any reason or disease progression (modified IWG-MRT 2013 including  $\geq$  25% increase in spleen volume by MRI/CT). In the absence of an event before the analysis is performed, the SDPFS will be censored at the date of the last valid assessment.

SDPFS will be analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the 25th, 50th, and 75th percentiles and the 95% confidence interval of median will be provided for both fedratinib and BAT arms. Kaplan-Meier curves will be plotted.

The analysis will be conducted based on ITT population.

#### 9.7.7. Durability of Spleen Response by Palpation (DRP)

Durability of spleen response by palpation (DRP) is defined as time from the date of the first documented palpable spleen response, according to the IWG-MRT 2013 (Appendix O) to the date of the subsequent PD in spleen size according to the IWG-MRT 2013 or death, whichever is earlier. Durability of spleen response by palpation according to the IWG-MRT 2013 criteria will be calculated for subjects that have an enlarged spleen at baseline (≥ 5 cm below LCM), and that have a spleen response by palpation. In the absence of an event before the analysis is performed, the DRP will be censored at the date of the last valid assessment performed before the analysis performed date.

Duration of spleen response by palpation will be analyzed using Kaplan-Meier method (K-M). Kaplan-Meier estimates of the 25th, 50th, and 75th percentiles and the 95% confidence interval of median will be provided for both fedratinib and BAT arms. Kaplan-Meier curves will be plotted.

The analysis will be conducted based on ITT population.

## 9.7.8. Overall Survival

Overall survival (OS) is defined as the time interval from the date of randomization to the date of death due to any cause. In the absence of the confirmation of death before the analysis performed, OS will be censored at the last date of subjects was known to be alive or at the study cut-off date (if applicable), whichever is earlier. OS will be analyzed based on the ITT population using the Kaplan-Meier method. Kaplan-Meier estimates of the 25th, 50th, and 75th percentiles and the 95% confidence intervals of median will be provided for both fedratinib and BAT arms. Kaplan-Meier curves will be plotted based on ITT population.

## 9.7.9. Crossover Efficacy Analysis

For crossover subjects, the visit cycles will be recounted from cycle 1 for fedratinib exposure period. The analyses during the fedratinib period will be summarized separately using the same method as described above. No formal statistical testing will be conducted to compare with BAT.

The analysis will be based on crossover efficacy population.

## 9.8. Safety Analysis

All safety analyses will be conducted based on the safety population or crossover safety population for crossover subjects.

Literature "book" values and normal ranges from local laboratory results will be utilized for this study.

#### 9.8.1. Adverse Events

The type, frequency, seriousness and severity of AEs, and relationship of AEs to study treatment will be summarized.

Adverse events will be analyzed in terms of TEAEs. TEAE is defined as any event that begins or worsens in grade after the start of study medication (or start of fedratinib for crossover subjects) through 30 days after the last dose of study treatment.

Adverse events will be summarized by severity/grade based on the NCI CTCAE. If a subject experiences the same AE multiple times during the treatment, the event will be counted only once by the worst grade / greatest severity.

Treatment emergent adverse events, Grade 3 or higher TEAEs, serious AEs, TEAEs leading to dose reduction, and dose interruption, TEAEs leading to treatment discontinuation, and TEAEs with an outcome of death will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred terms. Adverse events of special interest of fedratinib identified in previous trials in a similar population will be summarized in the same manner. If data warranted, additional analyses on fedratinib safety profile may be performed (eg, incidence of nausea, vomiting and diarrhea in relationship to prophylaxis and treatment, etc.) and will be specified in the statistical analysis plan.

# 9.8.2. Assessment of Risk Mitigation Strategy for Gastrointestinal Adverse Events and Encephalopathy, including Wernicke's

Assessment of risk mitigation strategy will include an analysis of incidence of subjects with a CTCAE Grade ≥3 of nausea, diarrhea, or vomiting, or occurrence of Encephalopathy, including Wernicke's (confirmed by brain MRI or autopsy). Analysis of thiamine levels will be at screening, on Day 1 of the first 3 cycles, every third cycle thereafter, and at the EOT during the study.

## 9.8.3. Laboratory Results

Analysis of laboratory data will be descriptive and conducted on the safety population. Summary of laboratory data (including thiamine levels) and change from baseline will also be performed by subject and by cycle.

Hematological toxicities will be assessed from laboratory parameters. Worst NCI CTCAE grades of leukopenia, neutropenia, thrombocytopenia, and anemia will be calculated according to the NCI common terminology criteria.

Qualitative and quantitative results will be summarized for hematological toxicities. Qualitative data (worst NCI CTCAE grade) will be summarized by cycle and by subject.

## 9.8.4. Electrocardiograms

All ECG data will be provided in a listing.

## 9.8.5. Vital Signs

Vital signs will be summarized based on the number of subjects with at least one potentially clinically significant abnormality (PCSA) occurring during the observation period according to baseline status. The PCSA criteria are provided in Table 5.

Table 5: PCSA Criteria for Vital Signs and Weight

| Parameter | PCSA |
|-------------|-----------------------------------------------------------|
| Heart (bpm) | ≤ 50 bpm and decrease from baseline ≥ 20 bpm |
| | $\geq$ 120 bpm and increase from baseline $\geq$ 20 bpm |
| SBP (mmHg) | $\leq$ 95 mmHg and decrease from baseline $\geq$ 20 mmHg |
| | $\geq$ 160 mmHg and increase from baseline $\geq$ 20 mmHg |
| DBP (mmHg) | ≤ 45 mmHg and decrease from baseline ≥ 10 mmHg |
| | $\geq$ 110 mmHg and increase from baseline $\geq$ 10 mmHg |
| Weight (kg) | ≥ 5 % increase from baseline |
| | ≥ 5 % decrease from baseline |

DBP = diastolic blood pressure; kg = kilograms; mmHg = millimeters of mercury; PCSA = potentially clinically significant abnormalities; SBP = systolic blood pressure.

# 9.9. Patient-reported Outcomes / Health Economics

Patient-Reported Outcomes and Health economics will be assessed using validated instruments (MFSAF version 4.0, EORTC QLQ-C30 version 3.0, EQ-5D-5L and analysis of MFSAF will be based on the ITT population with non-zero baseline TSS, and the analysis of EORTC QLQ-C30, EQ-5D-5L, and data will be based on the HRQoL-evaluable population.

## 9.9.1. Symptoms Response Assessment Using MFSAF V.4.0

The compliance profile over time will be summarized (number and percentage of forms received versus expected, and number of percentage of forms evaluable versus expected). A descriptive summary of each of the individual symptoms at each visit and change from baseline will be provided.

## **Total symptom score (TSS)**

The TSS is defined as the sum of each of the 7 symptom scores (Gwaltney, 2017). To allow indirect comparison with previous MF studies, a modified TSS (Mesa, 2013) will also be derived from the 6 symptoms considered (night sweats, pruritus, abdominal discomfort, early satiety, pain under ribs on left side, bone or muscle pain) and analysis of SRR will be also performed. Fatigue will be assessed as part of the EORTC QLQ-C30.

At each timepoint, the TSS (based on 7 symptoms) and the modified TSS will be calculated. Descriptive summary statistics (size, mean, standard deviation, median, range) will be provided

for baseline scores, postbaseline scores and change from baseline for TSS, modified TSS and symptom scores.

Additional statistical analysis will be provided in a separate HRQoL SAP and reported under a separate specific HRQoL Report.

#### **Durability of symptoms response (DSR)**

The DSR is defined as time from the first documented response in TSS (ie, reduction in TSS ≥ 50%) measured by MFSAF version 4.0 to the first documented TSS reduction < 50%. In the absence of TSS reduction < 50% before the analysis performed, the DSR will be censored at the date of the last valid assessment performed before the analysis performed date. DSR will be analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the 25th, 50th, and 75th percentiles and the 95% confidence intervals of median will be provided. Kaplan-Meier curves will be plotted.

## 9.9.2. EORTC QLQ-C30 Version 3.0

EORTC QLQ-C30 function and symptom domain scores will be calculated at each timepoint according to questionnaire guidelines (Aaronson, 1993). Missing values will be addressed according to questionnaire guidelines. Completion rate will be assessed by treatment arm. Details of data handling including transformation, missing data will be documented in a separate HRQoL SAP and support for further analyses which will be reported under a separate cover.

Descriptive summary statistics (size, mean, standard deviation, median, range) will be provided for EORTC QLQ-C30 function and symptom domain scores at each timepoint.

Changes over the study from baseline will also be reported.

Details of the statistical analysis other than summary statistics will be provided in a separate HRQoL SAP and reported in a separate specific HRQoL Report.

#### 9.9.3. EQ-5D-5L

The EORTC QLQ-C30 and EQ-5D-5L instruments will be scored using guidelines recommended by the EORTC (Fayers, 2001) and the EuroQol Group (2015) (van Reenen, 2015) respectively. The EQ-5D-5L health utility score will be derived according to published guidance (Cheung, 2015; Dolan, 1997). Missing responses for any of the 5 dimensions of the EQ-5D-5L will not be imputed. A higher score represents a better health status.

Descriptive summary statistics (size, mean, standard deviation, median, range) will be provided for health utility scores, and change from baseline will also be reported at each visit.

Additional analyses will be provided in a separate HRQoL/PRO SAP and reported in a separate specific HRQoL.





## 9.11. Interim Analysis

A formal interim analysis is not planned in this study. The primary endpoint will be analyzed at the end of 6 months after the date of first dose of fedratinib or BAT of the last treated subject. A follow up report will be prepared when the whole study is completed.

# 9.12. Other Topics

## 9.12.1. Steering Committee

The conduct of this trial will be overseen by a steering committee (SC), presided over by the coordinating Principal Investigator and if possible the representative Regional Investigators from countries participating in this study.

The SC will serve in an advisory capacity to the Sponsor. Operational details for the SC will be detailed in a separate SC charter.

#### 10. ADVERSE EVENTS

## 10.1. Monitoring, Recording and Reporting of Adverse Events

An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria in Section 10.3), regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE. A diagnosis or syndrome should be recorded on the AE page of the CRF rather than the individual signs or symptoms of the diagnosis or syndrome.

Abuse, withdrawal, sensitivity or toxicity to an investigational product should be reported as an AE. Overdose, accidental or intentional, whether or not it is associated with an AE should be reported on the overdose CRF. Any sequela of an accidental or intentional overdose of an investigational product which meets the definition of an adverse event should be reported as an AE on the CRF. If the sequela of an overdose meets serious criteria, then it must be marked as serious on the CRF. The overdose itself should not be reported as an AE.

Overdose, as defined in this protocol, refers to fedratinib dosing only. On a per dose basis, an overdose is defined as any amount over the protocol-specified dose of fedratinib assigned to a given subject, regardless of any associated adverse events or sequelae. On a schedule or frequency basis, an overdose is defined as anything more frequent than the protocol required schedule or frequency.

omplete data about drug administration, including any overdose, regardless of whether the overdose was accidental or intentional, should be reported in the case report form.

In the event of overdose, the subject should be monitored as appropriate and should receive supportive measures as necessary. There is no known specific antidote for fedratinib overdose. Actual treatment should depend on the severity of the clinical situation and the judgment and experience of the treating physician.

All subjects will be monitored for AEs during the study. Assessments may include monitoring of any or all of the following parameters: the subject's clinical symptoms, laboratory, pathological, radiological or surgical findings, physical examination findings, or findings from other tests and/or procedures.

All AEs will be recorded by the Investigator from the time the subject signs informed consent until 30 days after the last dose of fedratinib or comparator as well as those SAEs made known to the Investigator at any time thereafter that are suspected of being related to fedratinib or comparator. All adverse events (serious/non-serious) will be recorded on the CRF and in the subject's source documents. Refer to Section 10.5 for instructions on how to report SAEs to Drug Safety.

#### 10.2. Evaluation of Adverse Events

A qualified Investigator will evaluate all adverse events as to:

#### 10.2.1. Seriousness

An SAE is any AE occurring at any dose that:

- Results in death;
- Is life-threatening (ie, in the opinion of the Investigator, the subject is at immediate risk of death from the AE);
- Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay);
- Results in persistent or significant disability/incapacity (a substantial disruption of the subject's ability to conduct normal life functions);
- Is a congenital anomaly/birth defect;
- Constitutes an important medical event.

Important medical events are defined as those occurrences that may not be immediately life-threatening or result in death, hospitalization, or disability, but may jeopardize the subject or require medical or surgical intervention to prevent one of the other outcomes listed above. Medical and scientific judgment should be exercised in deciding whether such an AE should be considered serious.

Events **not considered** to be SAEs are hospitalizations for:

- a standard procedure for protocol therapy administration. However, hospitalization or prolonged hospitalization for a complication of therapy administration will be reported as an SAE.
- routine treatment or monitoring of the studied indication not associated with any deterioration in condition.
- the administration of blood or platelet transfusion as routine treatment of studied indication. However, hospitalization or prolonged hospitalization for a complication of such transfusion remains a reportable SAE.
- a procedure for protocol/disease-related investigations (eg, surgery, scans, endoscopy, sampling for laboratory tests, bone marrow sampling). However, hospitalization or prolonged hospitalization for a complication of such procedures remains a reportable SAE.
- hospitalization or prolongation of hospitalization for technical, practical, or social reasons, in absence of an AE.
- a procedure that is planned (ie, planned prior to start of treatment on study); must be documented in the source document and the CRF. Hospitalization or prolonged hospitalization for a complication remains a reportable SAE.

- an elective treatment of or an elective procedure for a pre-existing condition, unrelated to the studied indication, that has not worsened from baseline.
- emergency outpatient treatment or observation that does not result in admission, unless fulfilling other seriousness criteria above.

For each AE, the Investigator will provide information on severity, start and stop dates, relationship to fedratinib or comparator, action taken regarding the fedratinib or comparator, and outcome.

## 10.2.2. Severity/Intensity

For each AE, the Investigator must assess the severity/ intensity of the event.

The severity/intensity of AEs will be graded based upon the subject's symptoms according to the current active minor version of the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0);

https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm#ctc 50

AEs that are not defined in the CTCAE should be evaluated for severity/intensity according to the following scale:

- Grade 1 = Mild transient or mild discomfort; no limitation in activity; no medical intervention/therapy required
- Grade 2 = Moderate mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention/therapy required
- Grade 3 = Severe marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalization is possible
- Grade 4 = Life-threatening extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable
- Grade 5 = Death the event results in death

The term "severe" is often used to describe the intensity of a specific event (as in mild, moderate or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This criterion is not the same as "serious" which is based on subject/event outcome or action criteria associated with events that pose a threat to a subject's life or functioning.

Seriousness, not severity, serves as a guide for defining regulatory obligations.

## 10.2.3. Causality

The Investigator must determine the relationship between the administration of fedratinib or comparator and the occurrence of an AE as Not Suspected or Suspected as defined below:

Not suspected: a causal relationship of the adverse event to fedratinib or

comparator administration is **unlikely or remote**, or other medications, therapeutic interventions, or underlying conditions

provide a sufficient explanation for the observed event.

Suspected: there is a **reasonable possibility** that the administration of

fedratinib or comparator caused the adverse event. 'Reasonable

possibility' means there is evidence to suggest a causal

relationship between fedratinib or comparator and the adverse

event.

Causality should be assessed and provided for each AE based on currently available information. Causality is to be reassessed and provided as additional information becomes available.

If an event is assessed as suspected of being related to a comparator, ancillary or additional fedratinib that has not been manufactured or provided by Celgene-Impact, please provide the name of the manufacturer when reporting the event.

#### **10.2.4. Duration**

For each AE, the Investigator will provide a record of the start and stop dates of the event.

## 10.2.5. Action Taken

The Investigator will report the action taken with fedratinib or comparator as a result of each AE, as applicable (eg, discontinuation, interruption, or dose reduction of IP, as appropriate) and report if concomitant and/or additional treatments were given for the event.

#### **10.2.6.** Outcome

The Investigator will report the outcome of the event for each AE.

All SAEs that have not resolved upon discontinuation of the subject's participation in the study must be followed until recovered (returned to baseline), recovered with sequelae, or death (due to the SAE).

## 10.3. Abnormal Laboratory Values

An abnormal laboratory value is considered to be an AE if the abnormality:

- results in discontinuation from the study;
- requires treatment, modification/interruption of study treatment, or any other therapeutic intervention; or

• is judged to be of significant clinical importance, eg, one that indicates a new disease process and/or organ toxicity or is an exacerbation or worsening of an existing condition

Regardless of severity grade, only laboratory abnormalities that fulfill a seriousness criterion need to be documented as a serious adverse event.

If a laboratory abnormality is one component of a diagnosis or syndrome, then only the diagnosis or syndrome should be recorded as the AE. If the abnormality was not a part of a diagnosis or syndrome, then the laboratory abnormality should be recorded as the AE. If possible, the laboratory abnormality should be recorded as a medical term and not simply as an abnormal laboratory result (eg, record thrombocytopenia rather than decreased platelets).

## 10.4. Pregnancy

All pregnancies or suspected pregnancies occurring in either a female subject of childbearing potential or partner of childbearing potential of a male subject are immediately reportable events.

## **10.4.1.** Females of Childbearing Potential:

Pregnancies and suspected pregnancies (including elevated  $\beta$ -subunit of human chorionic gonadotropin [ $\beta$ hCG] or positive pregnancy test in a female subject of childbearing potential regardless of disease state) occurring while the subject is on fedratinib treatment, or within 30 days of the subject's last dose of fedratinib, are considered immediately reportable events. Investigational Product is to be discontinued immediately and the subject instructed to return any unused portion of the fedratinib to the Investigator. The pregnancy, suspected pregnancy, or positive pregnancy test must be reported to Celgene Drug Safety immediately by email, phone or facsimile, or other appropriate method, using the Pregnancy Initial Report Form, or approved equivalent form.

The female subject may be referred to an obstetrician-gynecologist or another appropriate healthcare professional for further evaluation.

The Investigator will follow the female subject until completion of the pregnancy and must notify Celgene Drug Safety immediately about the outcome of the pregnancy (either normal or abnormal outcome) using the Pregnancy Follow-up Report Form or approved equivalent form.

If the outcome of the pregnancy was abnormal (eg, spontaneous abortion), the Investigator should report the abnormal outcome as an AE. If the abnormal outcome meets any of the serious criteria, it must be reported as an SAE to Celgene Drug Safety within 24 hours of the Investigator's knowledge of the event.

All neonatal deaths that occur within 28 days of birth should be reported, without regard to causality, as an SAE. In addition, any infant death after 28 days that the Investigator suspects is related to the in-utero exposure to the fedratinib should also be reported as an SAE to Celgene Drug Safety within 24 hours of the Investigator's knowledge of the event.

## 10.4.2. Male Subjects

If a female partner of a male subject taking fedratinib becomes pregnant, the male subject taking fedratinib should notify the Investigator, and the pregnant female partner should be advised to call their healthcare provider immediately.

## 10.5. Reporting of Serious Adverse Events

Any AE that meets any seriousness criterion requires reporting as an SAE within 24 hours of the Investigator's knowledge of the event. This instruction pertains to initial SAE reports as well as any follow-up reports.

This requirement applies to all SAEs (regardless of relationship to fedratinib) that occur during the study (from the time the subject signs informed consent until 30 days after the last dose of IP) or any SAE made known to the Investigator at any time thereafter that are suspected of being related to IP. Serious adverse events occurring prior to treatment (after signing the ICF) are to be recorded within the CRF, but do not require reporting to Celgene Drug Safety.

Where required by local legislation, the Investigator is responsible for informing the Institutional Review Board/Ethics Committee (IRB/EC) of the SAE and providing them with all relevant initial and follow-up information about the event. The Investigator must keep copies of all SAE source documents and all correspondence with the IRB/EC.

The SAE is recorded within the CRF, and the data is transmitted electronically to Celgene Drug Safety within 24 hours of the Investigator's knowledge of the event. In the event electronic transmission is not available, a paper SAE Report Form will be completed and sent directly to Celgene Drug Safety, ensuring the event is recorded on the CRF as well.

## 10.5.1. Safety Queries

Queries pertaining to SAEs will be communicated from Celgene Drug Safety to the site via electronic data capture (EDC) or other appropriate method. The response time is expected to be no more than five (5) business days. Urgent queries (eg, missing causality assessment) may be handled by phone.

# **10.6.** Expedited Reporting of Adverse Events

For the purpose of regulatory reporting, Celgene Drug Safety will determine the expectedness of events suspected of being related to fedratinib based on the Investigator Brochure.

In the United States, expedited reports sent to the FDA by the sponsor based on the reasonable possibility threshold are known as "IND safety reports" and will be reported in accordance with 21 CFR 312.32.

For reporting to the FDA, events that are not suspected to be causally related to fedratinib by the sponsor will not be considered adverse reactions. As per FDA regulations, events that are anticipated in the study population, listed in the fedratinib IB Reference Safety Information, will not be considered adverse reactions on individual assessment and will be reviewed on an aggregate basis for assessment of frequency.

For countries within the European Economic Area (EEA), Celgene or its authorized representative will report in an expedited manner to Regulatory Authorities and Ethics

Committees concerned, suspected unexpected serious adverse reactions (SUSARs) with fedratinib in accordance with Directive 2001/20/EC and the Detailed Guidance on collection, verification and presentation of adverse reaction reports arising from clinical trials on investigational products for human use (ENTR/CT3) and also in accordance with country-specific requirements.

For the purpose of regulatory reporting in the EEA, Celgene Drug Safety will determine the expectedness of events suspected of being related to the comparator, based on the UK or EU Summary of Product Characteristics (SmPC).

For the purpose of regulatory reporting in the EEA, Celgene non-investigational medicinal product (when the comparator is a Celgene product such as thalidomide) serious adverse reactions and nonserious adverse reactions will be reported to the Regulatory Authorities, in accordance with Regulation (EC) No. 726/2004 and/or Directive 2001/83/EC as amended, and also in accordance with country-specific requirements for countries within the EEA.

Celgene or its authorized representative shall notify the Investigator of the following information

- Any AE suspected of being related to the use of fedratinib in this study or in other studies that is both serious and unexpected (ie, SUSAR);
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects including reports of mutagenicity, teratogenicity, or carcinogenicity.

Where required by local legislation, the Investigator shall notify his/her IRB/EC promptly of these new serious and unexpected AE(s) or significant risks to subjects.

The Investigator must keep copies of all pertinent safety information on file including correspondence with Celgene and the IRB/EC. (See Section 14.3 for record retention information).

# 10.7. Adverse Events of Special Interest

An adverse event of special interest (AESI) is one of scientific and medical interest specific to understanding of the Investigational Product and may require close monitoring and rapid communication by the Investigator to the Sponsor. AESI (serious and non-serious) are to be recorded within the CRF and the data transmitted electronically to Celgene Drug Safety within 24 hours of the Investigator's knowledge of the event. In the event electronic transmission is not available, a paper SAE Report Form will be completed and sent directly to Celgene Drug Safety, ensuring the event is recorded on the CRF as well. The rapid reporting of AESIs allows ongoing surveillance of these events to characterize and understand them in association with the use of this Investigational Product. Events of special interest may be referred to external experts for review as needed.

The following are considered to be Adverse Events of Special Interest (AESIs):

- Encephalopathy, including Wernicke's (WE) or suspected cases of WE associated with thiamine levels below normal range.
- Thiamine levels below normal range with or without signs or symptoms of WE
- New malignancy after start of study treatment

- Progression of myelofibrosis to acute myeloid leukemia (AML)
- Cardiac failure or cardiomyopathy
- Grade 3 or 4 hyperlipasemia or Grade 3 or 4 hyperamylasemia according to CTCAE criteria, v 5.0 or events of pancreatitis
- Grade 3 or 4 alanine transaminase (ALT), aspartate transaminase (AST), or total bilirubin elevation or events of hepatotoxicity

## 11. DISCONTINUATIONS

#### 11.1. Treatment Discontinuation

The following events are considered sufficient reasons for discontinuing a subject from fedratinib

- Lack of efficacy
- Adverse event
- Progression of disease according to the IWG-MRT 2013 criteria
- Withdrawal by subject
- Death
- Lost to follow-up
- Pregnancy
- Protocol deviation
- Study terminated by Sponsor
- Treatment discontinuation guidance related to the Dose Modification Schedule table (Table 4)
- Other (to be specified on the CRF)

The reason for discontinuation of treatment should be recorded in the CRF and in the source documents. The decision to discontinue a subject from treatment remains the responsibility of the treating physician, which will not be delayed or refused by the Sponsor. However, prior to discontinuing a subject, the Investigator may contact the Medical Monitor and forward appropriate supporting documents for review and discussion.

Subjects that discontinue treatment will complete the 30-Day follow-up visit and enter the Survival Follow-up.

# 11.2. Study Discontinuation

The following events are considered sufficient reasons for discontinuing a subject from the study:

- Screen failure
- Withdrawal by subject
- Death
- Lost to follow-up
- Protocol deviation
- Study terminated by Sponsor
- Other (to be specified on the CRF)

The reason for study discontinuation should be recorded in the CRF and in the source documents.

## 12. EMERGENCY PROCEDURES

## **12.1.** Emergency Contact

In emergency situations, the Investigator should contact the responsible Clinical Research Physician/Medical Monitor or designee by telephone at the number(s) listed on the Emergency Contact Information page of the protocol (after title page).

In the unlikely event that the Clinical Research Physician/Medical Monitor or designee cannot be reached, please contact the global Emergency Call Center by telephone at the number listed on the Emergency Contact Information page of the protocol (after title page). This global Emergency Call Center is available 24 hours a day and 7 days a week. The representatives are responsible for obtaining your call-back information and contacting the on-call Celgene-Impact/contract research organization Medical Monitor, who will then contact you promptly.

Note: The back-up 24-hour global emergency contact call center should only be used if you are not able to reach the Clinical Research Physician(s) or Medical Monitor or designee for emergency calls.

## 12.2. Emergency Identification of Investigational Products

This is an open-label study; therefore, fedratinib will be identified on the package labeling.

## 13. REGULATORY CONSIDERATIONS

#### 13.1. Good Clinical Practice

The procedures set out in this study protocol pertaining to the conduct, evaluation, and documentation of this study are designed to ensure that Celgene-Impact, its authorized representative, and Investigator abide by Good Clinical Practice (GCP), as described in International Counsel on Harmonisation (ICH) Guideline E6 and in accordance with the general ethical principles outlined in the Declaration of Helsinki. The study will receive approval from an IRB/EC prior to commencement. The Investigator will conduct all aspects of this study in accordance with applicable national, state, and local laws of the pertinent regulatory authorities.

## 13.2. Investigator Responsibilities

Investigator responsibilities are set out in the ICH Guideline for Good Clinical Practice and in the local regulations. Celgene-Impact staff or an authorized representative will evaluate and approve all Investigators who in turn will select their staff.

The Investigator should ensure that all persons assisting with the study are adequately informed about the protocol, amendments, study treatments, as well as study-related duties and functions, including obligations of confidentiality of Celgene-Impact information. The Investigator should maintain a list of Sub-investigators and other appropriately qualified persons to whom he or she has delegated significant study-related duties.

The Investigator is responsible for keeping a record of all subjects who sign an informed consent form (ICF) and are screened for entry into the study. Subjects who fail screening must have the reason(s) recorded in the subject's source documents.

The Investigator, or a designated member of the Investigator's staff, must be available during monitoring visits to review data, resolve queries and allow direct access to subject records (eg, medical records, office charts, hospital charts, and study-related charts) for source data verification. The Investigator must ensure timely and accurate completion of CRFs and queries.

The information contained in the protocol and amendments (with the exception of the information provided by Celgene-Impact on public registry websites) is considered Celgene-Impact confidential information. Only information that is previously disclosed by Celgene-Impact on a public registry website may be freely disclosed by the Investigator or its institution, or as outlined in the Clinical Trial Agreement. Celgene-Impact protocol, amendment and IB information is not to be made publicly available (for example on the Investigator's or their institution's website) without express written approval from Celgene-Impact. Information proposed for posting on the Investigator's or their institution's website must be submitted to Celgene-Impact for review and approval, providing at least 5 business days for review.

At the time results of this study are made available to the public, Celgene-Impact will provide Investigators with a summary of the results that is written for the lay person. The Investigator is responsible for sharing these results with the subject and/or their caregiver as agreed by the subject.

## 13.3. Subject Information and Informed Consent

The Investigator must obtain informed consent of a subject and/or a subject's legal representative prior to any study related procedures.

Documentation that informed consent occurred prior to the study subject's entry into the study and of the informed consent process should be recorded in the study subject's source documents including the date. The original ICF signed and dated by the study subject and by the person consenting the study subject prior to the study subject's entry into the study, must be maintained in the Investigator's study files and a copy given to the study subject. In addition, if a protocol is amended and it impacts on the content of the informed consent, the ICF must be revised. Study subjects participating in the study when the amended protocol is implemented must be reconsented with the revised version of the ICF. The revised ICF signed and dated by the study subject and by the person consenting the study subject must be maintained in the Investigator's study files and a copy given to the study subject.

## 13.4. Confidentiality

Celgene-Impact affirms the subject's right to protection against invasion of privacy and to be in compliance with ICH and other local regulations (whichever is most stringent). Celgene-Impact requires the Investigator to permit Celgene-Impact's representatives and, when necessary, representatives from regulatory authorities, to review and/or copy any medical records relevant to the study in accordance with local laws.

Should direct access to medical records require a waiver or authorization separate from the subject's signed ICF, it is the responsibility of the Investigator to obtain such permission in writing from the appropriate individual.

## 13.5. Protocol Amendments

Any amendment to this protocol must be approved by the Celgene-Impact Clinical Research Physician/Medical Monitor. Amendments will be submitted to the IRB/EC for written approval. Written approval must be obtained before implementation of the amended version occurs. The written signed approval from the IRB/EC should specifically reference the Investigator name, protocol number, study title and amendment number(s) that is applicable. Amendments that are administrative in nature do not require IRB/IEC approval but will be submitted to the IRB/IEC for information purposes.

# 13.6. Institutional Review Board/Independent Ethics Committee Review and Approval

Before the start of the study, the study protocol, ICF, and any other appropriate documents will be submitted to the IRB/EC with a cover letter or a form listing the documents submitted, their dates of issue, and the site (or region or area of jurisdiction, as applicable) for which approval is sought. If applicable, the documents will also be submitted to the authorities in accordance with local legal requirements.

Fedratinib can only be supplied to an Investigator by Celgene-Impact or its authorized representative after documentation on all ethical and legal requirements for starting the study has been received by Celgene-Impact or its authorized representative. This documentation must also include a list of the members of the IRB/EC and their occupation and qualifications. If the IRB/EC will not disclose the names, occupations and qualifications of the committee members, it should be asked to issue a statement confirming that the composition of the committee is in accordance with GCP. For example, the IRB General Assurance Number may be accepted as a substitute for this list. Formal approval by the IRB/EC should mention the protocol title, number, amendment number (if applicable), study site (or region or area of jurisdiction, as applicable), and any other documents reviewed. It must mention the date on which the decision was made and must be officially signed by a committee member. Before the first subject is enrolled in the study, all ethical and legal requirements must be met.

The IRB/EC and, if applicable, the authorities, must be informed of all subsequent protocol amendments in accordance with local legal requirements. Amendments must be evaluated to determine whether formal approval must be sought and whether the ICF should also be revised.

The Investigator must keep a record of all communication with the IRB/EC and, if applicable, between a Coordinating Investigator and the IRB/EC. This statement also applies to any communication between the Investigator (or Coordinating Investigator, if applicable) and regulatory authorities.

Any advertisements used to recruit subjects for the study must be reviewed by Celgene-Impact and the IRB/EC prior to use.

# 13.7. Ongoing Information for Institutional Review Board/ Ethics Committee

If required by legislation or the IRB/EC, the Investigator must submit to the IRB/EC:

- Information on serious or unexpected adverse events as soon as possible;
- Periodic reports on the progress of the study;
- Deviations from the protocol or anything that may involve added risk to subjects.

# 13.8. Termination of the Study

Celgene-Impact reserves the right to terminate this study prematurely at any time for reasonable medical or administrative reasons. Any premature discontinuation will be appropriately documented according to local requirements (eg, IRB/EC, regulatory authorities, etc).

In addition, the Investigator or Celgene-Impact has the right to discontinue a single site at any time during the study for medical or administrative reasons such as:

- Unsatisfactory enrollment;
- GCP noncompliance;
- Inaccurate or incomplete data collection;
- Falsification of records:
- Failure to adhere to the study protocol.

#### 14. DATA HANDLING AND RECORDKEEPING

#### 14.1. Data/Documents

The Investigator must ensure that the records and documents pertaining to the conduct of the study and the distribution of the investigational product are complete, accurate, filed and retained. Examples of source documents include: hospital records; clinic and office charts; laboratory notes; memoranda; subject's diaries or evaluation checklists; dispensing records; recorded data from automated instruments; copies or transcriptions certified after verification as being accurate copies; microfiche; x-ray film and reports; and records kept at the pharmacy, and the laboratories, as well as copies of CRFs or CD-ROM.

# 14.2. Data Management

Data will be collected via CRF and entered into the clinical database per Celgene Standard Operating Procedures (SOPs). This data will be electronically verified through use of programmed edit checks specified by the clinical team. Discrepancies in the data will be brought to the attention of the clinical team, and investigational site personnel, if necessary. Resolutions to these issues will be reflected in the database. An audit trail within the system will track all changes made to the data.

## 14.3. Record Retention

Essential documents must be retained by the Investigator according to the period of time outlined in the clinical trial agreement. The Investigator must retain these documents for the time period described above or according to local laws or requirements, whichever is longer. Essential documents include, but are not limited to, the following:

- Signed ICFs for all subjects;
- Subject identification code list, screening log (if applicable), and enrollment log;
- Record of all communications between the Investigator and the IRB/EC;
- Composition of the IRB/EC;
- Record of all communications between the Investigator, Celgene-Impact, and their authorized representative(s);
- List of Sub-investigators and other appropriately qualified persons to whom the Investigator has delegated significant study-related duties, together with their roles in the study, curriculum vitae, and their signatures;
- Copies of CRFs (if paper) and of documentation of corrections for all subjects;
- Fedratinib accountability records;
- Record of any body fluids or tissue samples retained;
- All other source documents (subject records, hospital records, laboratory records, etc.);

• All other documents as listed in Section 8 of the ICH consolidated guideline on GCP (Essential Documents for the Conduct of a Clinical Trial).

The Investigator must notify Celgene-Impact if he/she wishes to assign the essential documents to someone else, remove them to another location or is unable to retain them for a specified period. The Investigator must obtain approval in writing from Celgene-Impact prior to destruction of any records. If the Investigator is unable to meet this obligation, the Investigator must ask Celgene-Impact for permission to make alternative arrangements. Details of these arrangements should be documented.

All study documents should be made available if required by relevant health authorities. Investigator or institution should take measures to prevent accidental or premature destruction of these documents.

## 15. QUALITY CONTROL AND QUALITY ASSURANCE

All aspects of the study will be carefully monitored by Celgene-Impact or its authorized representative for compliance with applicable government regulations with respect to current GCP and SOPs.

## 15.1. Study Monitoring and Source Data Verification

Celgene-Impact ensures that appropriate monitoring procedures are performed before, during and after the study. All aspects of the study are reviewed with the Investigator and the staff at a study initiation visit and/or at an Investigators' Meeting. Prior to enrolling subjects into the study, a Celgene-Impact representative will review the protocol, CRFs, procedures for obtaining informed consent, record keeping, and reporting of AEs/SAEs with the Investigator. Monitoring will include on-site visits with the Investigator and his/her staff as well as any appropriate communications by mail, email, fax, or telephone. During monitoring visits, the facilities, investigational product storage area, CRFs, subject's source documents, and all other study documentation will be inspected/reviewed by the Celgene-Impact representative in accordance with the Study Monitoring Plan.

Accuracy will be checked by performing source data verification that is a direct comparison of the entries made onto the CRFs against the appropriate source documentation. Any resulting discrepancies will be reviewed with the Investigator and/or his/her staff. Any necessary corrections will be made directly to the CRFs or via queries by the Investigator and/or his/her staff. Monitoring procedures require that informed consents, adherence to inclusion/exclusion criteria and documentation of SAEs and their proper recording be verified. Additional monitoring activities may be outlined in a study-specific monitoring plan.

# **15.2.** Audits and Inspections

In addition to the routine monitoring procedures, a Good Clinical Practice Quality Assurance unit exists within Celgene-Impact. Representatives of this unit will conduct audits of clinical research activities in accordance with Celgene SOPs to evaluate compliance with Good Clinical Practice guidelines and regulations.

The Investigator is required to permit direct access to the facilities where the study took place, source documents, CRFs and applicable supporting records of study subject participation for audits and inspections by IRB/ECs, regulatory authorities (eg, FDA, EMA, Health Canada) and company authorized representatives. The Investigator should make every effort to be available for the audits and/or inspections. If the Investigator is contacted by any regulatory authority regarding an inspection, he/she should contact Celgene-Impact immediately.

# **15.3.** Product Quality Complaint

A Product Quality Complaint (PQC) is any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, purity, or performance of any drug product manufactured by or on behalf of Celgene-Impact after it is released for distribution. PQCs may reduce the usability of the product for its intended function or affect performance of the product and therefore pose a significant risk to the subject. Examples of PQCs include (but are not limited to): mixed product, mislabeling, lack of effect,

seal/packaging breach, product missing/short/overage, contamination, suspected falsified, tampered, diverted or stolen material, and general product/packaging damage. If you become aware of a suspected PQC, you are obligated to report the issue immediately.

## 16. PUBLICATIONS

As described in Section 13.2, all protocol- and amendment-related information, with the exception of the information provided by Celgene-Impact on public registry websites, is considered Celgene-Impact confidential information and is not to be used in any publications. Celgene-Impact protocol-related information proposed for use in a publication must be submitted to Celgene-Impact for review and approval and should not be utilized in a publication without express written approval from Celgene-Impact, or as described in the Clinical Trial Agreement.

Celgene-Impact will ensure Celgene-Impact-sponsored studies are considered for publication in the scientific literature in a peer-reviewed journal, irrespective of the results. At a minimum, this applies to results from all Phase 3 clinical studies, and any other study results of significant medical importance. This also includes results relating to investigational medicines whose development programs have been discontinued.

Study results may also be presented at one or more medical congresses and may be used for scientific exchange and teaching purposes. Additionally, this study and its results may be submitted for inclusion in all appropriate health authority study registries, as well as publication on health authority study registry websites, as required by local health authority regulations.

Eligibility for external authorship, as well as selection of first authorship, will be based on several considerations, including, but not limited to, contribution to protocol development, study recruitment, data quality, participation in data analysis, participation in study steering committee (when applicable) and contribution to abstract, presentation and/or publication development.

#### 17. REFERENCES

AHA Medical/Scientific Statement: 1994 Revisions to Classification of Functional Capacity and Objective Assessment of Patients With Diseases of the Heart. Circulation. 1994;90:644-645.

Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 03;85(5):365-76.

Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, et al. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405.



Barosi G, Mesa RA, Thiele J, Cervantes F, Campbell PJ, Verstovsek S, et al. Proposed criteria for the diagnosis of post-polycythemia vera and post-essential thrombocythemia myelofibrosis: a consensus statement from the International Working Group for Myelofibrosis Research and Treatment. Leukemia. 2008 Feb;22(2):437-8.



Campbell PJ, Green AD. Management of polycythemia vera and essential thrombocythemia. Hematology Am Soc Hematol Educ Program. 2005:201-8.

Cervantes F, Dupriez B, Pereira A, Passamonti F, Reilly JT, Morra E, et al. New prognostic scoring system for primary myelofibrosis based on a study of the International Working Group for Myelofibrosis Research and Treatment. Blood. 2009 Mar 26;113(13):2895-901.

Cervantes F, Kiladjian JJ, Niederwieser D, Sirulnik A, Stalbovskaya V, McQuity M, et al. Long-Term Safety, Efficacy, and Survival Findings From Comfort-II, a Phase 3 Study Comparing Ruxolitinib with Best Available Therapy (BAT) for the Treatment of Myelofibrosis (MF). Blood. 2012;120(21):801.

Cheung MC, Hay AE, Crump M, Imrie KR, Song Y, Hassan S, et al. Gemcitabine/dexamethasone/cisplatin vs cytarabine/dexamethasone/cisplatin for relapsed or refractory aggressive-histology lymphoma: cost-utility analysis of NCIC CTG LY.12. J Natl Cancer Inst. 2015 Jul;107(7).

Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108.



EuroQol Research Foundation. EQ-5D-5L User Guide, Ver 2.1. EuroQol Research Foundation [Internet]. 2015 Apr. Available from: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L\_UserGuide\_2015.pdf.

Fayers P. Interpreting quality of life data: population-based reference data for the EORTC QLQ-C30. Eur J Cancer. 2001 Jul;37(11):1331-4.

Gangat N, Caramazza D, Vaidya R, George G, Begna K, Schwager S, et al. DIPSS plus: a refined Dynamic International Prognostic Scoring System for primary myelofibrosis that incorporates prognostic information from karyotype, platelet count, and transfusion status. J Clin Oncol. 2011 Feb 1;29(4):392-7.

Gwaltney C, Paty J, Kwitkowski VE, Mesa RA, Dueck AC, Papadopoulos EJ, et al. Development of a harmonized patient-reported outcome questionnaire to assess myelofibrosis symptoms in clinical trials. Leuk Res. 2017 Aug;59:26-31.



Harrison C, Vannucchi AD. Ruxolitinib: a potent and selective Janus kinase 1 and 2 inhibitor in patients with myelofibrosis. An update for clinicians. Ther Adv Hematol. 2012 Dec;3(6):341-54.

Harrison CN, McLornan DP. Current treatment algorithm for the management of patients with myelofibrosis, JAK inhibitors, and beyond. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):489-97.

Harrison CN, Mesa RA, Jamieson C, Hood J, Bykowski J, Zuccoli G, et al. Case Series of Potential Wernicke's Encephalopathy in Patients Treated with Fedratinib. 2018;130(Suppl 1):4197.

Harrison CN, Vannucchi AM, Platzbecker U, Cervantes F, Gupta V, Lavie D, et al. Momelotinib versus best available therapy in patients with myelofibrosis previously treated with ruxolitinib (SIMPLIFY 2): a randomised, open-label, phase 3 trial. Lancet Haematol. 2018 Feb;5(2):e73-e81.

Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36.

Hjermstad MJ, Fossa SD, Bjordal K, Kaasa S. Test/retest study of the European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire. J Clin Oncol. 1995 May;13(5):1249-54.

Ihle JN, Gilliland DD. Jak2: normal function and role in hematopoietic disorders. Curr Opin Genet Dev. 2007 Feb;17(1):8-14.

Jabbour E, Kantarjian HM, Garcia-Manero G, Quintas-Cardama A, Cardena-Turanzas M, O'Brien S, et al. Outcome Of Patients (pts) With Myelofibrosis (MF) After Ruxolutinib (Rux) Therapy [abstract]. Presented at: 55th Annual Meeting of the American Society of Hematology (ASH): 2013; New Orleans, LA, USA. Abstract No. 1584.

Janssen MF, Birnie E, Bonsel GD. Quantification of the level descriptors for the standard EQ-5D three-level system and a five-level version according to two methods. Qual Life Res. 2008a Apr;17(3):463-73.

Janssen MF, Birnie E, Haagsma JA, Bonsel GD. Comparing the standard EQ-5D three-level system with a five-level version. Value Health. 2008b Mar-Apr;11(2):275-84.

Kantarjian HM, Silver RT, Komrokji RS, Mesa RA, Tacke R, Harrison CN. Ruxolitinib for myelofibrosis--an update of its clinical effects. Clin Lymphoma Myeloma Leuk. 2013 Dec;13(6):638-45.

Keohane C, Radia DH, Harrison CN. Treatment and management of myelofibrosis in the era of JAK inhibitors. Biologics. 2013;7(1):189-98.

King MT. The interpretation of scores from the EORTC quality of life questionnaire QLQ-C30. Qual Life Res. 1996 Dec;5(6):555-67.



Kvasnicka HD. WHO classification of myeloproliferative neoplasms (MPN): A critical update. Curr Hematol Malig Rep. 2013 Dec;8(4):333-41.

Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54.



Mascarenhas J, Hoffman R, Talpaz M, Gerds AT, Stein B, Gupta V, et al. Pacritinib vs Best Available Therapy, Including Ruxolitinib, in Patients With Myelofibrosis: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):652-9.



Mesa RA, Camoriano JK, Geyer SM, Wu W, Kaufmann SH, Rivera CE, et al. A phase II trial of tipifarnib in myelofibrosis: primary, post-polycythemia vera and post-essential thrombocythemia. Leukemia. 2007 Sep;21(9):1964-70.

Mesa RA, Gotlib J, Gupta V, Catalano JV, Deininger MW, Shields AL, et al. Effect of ruxolitinib therapy on myelofibrosis-related symptoms and other patient-reported outcomes in COMFORT-I: a randomized, double-blind, placebo-controlled trial. J Clin Oncol. 2013 Apr 1;31(10):1285-92.



Oh ST, Simonds EF, Jones C, Hale MB, Goltsev Y, Gibbs KD, Jr., et al. Novel mutations in the inhibitory adaptor protein LNK drive JAK-STAT signaling in patients with myeloproliferative neoplasms. Blood. 2010 Aug 12;116(6):988-92.

Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55.

Osoba D, Aaronson N, Zee B, Sprangers M, te Velde A. Modification of the EORTC QLQ-C30 (version 2.0) based on content validity and reliability testing in large samples of patients with cancer. The Study Group on Quality of Life of the EORTC and the Symptom Control and Quality of Life Committees of the NCI of Canada Clinical Trials Group. Qual Life Res. 1997 Mar;6(2):103-8.

Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44.



Passamonti F, Cervantes F, Vannucchi AM, Morra E, Rumi E, Pereira A, et al. A dynamic prognostic model to predict survival in primary myelofibrosis: a study by the IWG-MRT (International Working Group for Myeloproliferative Neoplasms Research and Treatment). Blood. 2010 Mar 04;115(9):1703-8.



Pikman Y, Lee BH, Mercher T, McDowell E, Ebert BL, Gozo M, et al. MPLW515L is a novel somatic activating mutation in myelofibrosis with myeloid metaplasia. PLoS Med. 2006 Jul;3(7):e270.



Swerdlow SH, Editors. WHO classification of tumours of haematopoietic and lymphoid tissues. Lyon, France: IARC Press, 2008.

Tefferi A. Primary myelofibrosis: 2017 update on diagnosis, risk-stratification, and management. Am J Hematol. 2016 Dec;91(12):1262-71.

Tefferi A. The recent advances in classic BCR-ABL-negative myeloproliferative disorders. Clin Adv Hematol Oncol. 2007;5:113-

Tefferi A, Cervantes F, Mesa R, Passamonti F, Verstovsek S, Vannucchi AM, et al. Revised response criteria for myelofibrosis: International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus report. Blood. 22 Aug 2013;122(8):1395-8.



van Reenen M, Janssen B. [Internet]. EQ-5D-5L user guide: basic information on how to use the EQ-5D-5L instrument. Version 2.1. Rotterdam (Netherlands): EuroQol Research Foundation;

April 2015. [cited 2018 Mmm dd]. Available from: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L UserGuide 2015.pdf

Vannucchi AM, Harrison CN. Emerging treatments for classical myeloproliferative neoplasms. Blood. 2017 Feb 9;129(6):693-703.

Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, et al. A double-blind, placebo-controlled trial of ruxolitinib for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):799-807.



## 18. APPENDICES

## APPENDIX A. TABLE OF ABBREVIATIONS AND SPECIAL TERMS

| Abbreviation or<br>Specialist Term | Explanation |
|---|---|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AML | Acute myeloid leukemia |
| ANC | Absolute neutrophil count |
| AST | Aspartate aminotransferase |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the curve |
| BAT | Best available therapy |
| BM | Bone marrow |
| BUN | Blood urea nitrogen |
| CALR | Calreticulin |
| CI | Confidence interval |
| CRF | Case report form |
| CSR | Clinical Study report |
| CT | Computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CYP2C19 | Cytochrome P450 2C19 |
| CYP3A4 | Cytochrome P450 3A4 |
| CYP2D6 | Cytochrome P450 2D6 |
| DIPSS | Dynamic International Prognostic Scoring System |
| DR | Duration of spleen volume response |
| DRP | Duration of spleen response by palpation |
| DSR | Duration of symptoms response |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |

| Abbreviation or<br>Specialist Term | Explanation |
|---|---|
| EEA | European Economic Area |
| EORTC | European Organization for Research and Treatment of Cancer |
| EMA | European Medicine Agency |
| EOT | End of treatment |
| ET | Essential thrombocythemia |
| EU | European Union |
| FCBP | Female of childbearing potential |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte-colony stimulating factor |
| GI | Gastrointestinal |
| GVHD | Graft-versus-host-disease |
| Hgb | Haemoglobin |
| HIV | Human immunodeficiency virus |
| HRQoL | Health-related Quality of Life |
| IB | Investigator Brochure |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| IL- | Interleukin- |
| IPSS | International Prognostic Scoring System |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technology |
| IWG-MRT | International Working Group-Myeloproliferative Neoplasms Research and Treatment |
| JAK | Janus kinase |
| K-M | Kaplan-Meier |
| LCM | Left costal margin |
| LDH | Lactate dehydrogenase |
| LFT | Liver function test |
| MDRD | Modification of Diet in Renal Disease |
| MedDRA | Medical Dictionary for Regulatory Activities |

| Abbreviation or<br>Specialist Term | Explanation |
|---|---|
| MF | Myelofibrosis (in terms of this protocol, myeloproliferative neoplasm associated myelofibrosis) |
| MFSAF | Myelofibrosis Symptom Assessment Form |
| MMSE | Mini-Mental State Examination |
| MPL | Myeloproliferative leukemia virus |
| MPN | Myeloproliferative neoplasms |
| MRI | Magnetic resonance imaging |
| MTD | Maximum tolerated dose |
| NCI | National Cancer Institute |
| OS | Overall survival |
| PB | Peripheral blood |
| PD | progressive disease |
| PD-L1 | Program death-ligand 1 |
| PK | Pharmacokinetics |
| PLT | Platelet |
| PMF | Primary myelofibrosis |
| PQC | Product Quality Complaint |
| PRO | Patient-reported outcomes |
| PS | Performance Status |
| PV | Polycythemia vera |
| QD | Once a day |
| QoL | Quality of Life |
| RBC | Red blood cell |
| RR | Response rate |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SC | Steering committee |
| SCT | Stem-cell transplantation |
| SDPFS | Spleen and disease progression free survival |
| SOP | Standard Operating Procedure |
| SRR | Symptom response rate |
| STAT | Signal transducers and activators of transcription |
| Abbreviation or<br>Specialist Term | Explanation | | |
|---|---|--|--|
| SUSAR | Suspected unexpected serious adverse reaction | | |
| SVR | Spleen volume reduction | | |
| TEAE | Treatment Emergent Adverse Event | | |
| TGF-β | Transforming growth factor-β | | |
| T <sub>max</sub> | Time to maximum plasma concentration | | |
| TNF-a | Tumor necrosis factor-a | | |
| TSS | Total Symptom Score | | |
| ULN | Upper limit of normal | | |
| US | United States | | |
| VAS | Visual analog scale | | |
| WBC | White blood cell | | |
| WE | Wernicke Encephalopathy | | |
| WHO | World Health Organization | | |

## APPENDIX B. MYELOFIBROSIS SYMPTOM ASSESSMENT FORM (MFSAF) VERSION 4.0

Myelofibrosis Symptom Assessment Form version 4.0 7-Day Recall (MFSAF v4.0 7-Day Recall)

Instructions (to be modified based on data collection mode): The following questions refer to symptoms that you may experience as a result of your myelofibrosis. Please read through and complete the questions on the following screens. There are no right or wrong answers. Please select the answer that best applies to you.

| Ite | ms: | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. | During the pa | st 7 da | ys, hov | wseve: | re was | yourv | vorst fa | atigue ( | (weari | ness, t | tiredness)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 2. | During the pa | st 7 da | ys, hov | wseve: | re were | your | worst 1 | nights | weats | (or fee | eling hot or flushed)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 3. | During the pa | st 7 da | ys, hov | wseve: | re was | yourv | vorst it | ching' | ? | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 4. | During the par<br>bloating)? | st 7 da | ys, hov | wseve: | re was | yourv | vorst a | bdomi | naldis | comf | ort (feeling pressure or |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 5. | During the pa | st 7 da | ys, hov | wseve: | re was | the wo | rst pai | n unde | eryou | rribso | on your left side? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 6. | During the pa | st 7 da | ys, wh | at was | the wo | rst fee | ling o | ffullne | ess you | ı had a | after beginning to eat? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Absent | | | | | | | | | | Worst Imaginable |
| 7. | During the pa | st 7 da | ys, hov | wseve: | re was | yourv | vorst b | one pa | in (no | tjoint | or arthritis pain)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |

MYELOFIBROSIS SYMPTOM ASSESSMENT FORM VERSION 4.07-DAY RECALL (MFSAF v4.07-DAY RECALL)

© 2010-2016 MAYO CLINIC. ALL RIGHTS RESERVED.

Source: (Gwaltney, 2017).

Absent

Worst Imaginable

## APPENDIX C. QUALITY OF LIFE ASSESSMENT: EORTC QLQ-C30 QUESTIONNAIRE

#### EORTC QLQ-C30 (version 3)

Your birthdate (Day, Month, Year):

Please fill in your initials:

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers. The information that you provide will remain strictly confidential.

| Too | Today's date (Day, Month, Year): 31 🗆 🗆 🗆 🗆 🗆 | | | | |
|---|---|---|---|---|---|
| | | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 1. | Do you have any trouble doing strenuous activities,<br>like carrying a heavy shopping bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2. | Do you have any trouble taking a <u>long</u> walk? | 1 | 2 | 3 | 4 |
| 3. | Do you have any trouble taking a $\underline{short}$ walk outside of the house? | 1 | 2 | 3 | 4 |
| 4. | Do you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| 5. | Do you need help with eating, dressing, washing yourself or using the toilet? | 1 | 2 | 3 | 4 |
| Dι | ıring the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 6. | Were you limited in doing either your work or other daily activities? | 1 | 2 | 3 | 4 |
| 7. | Were you limited in pursuing your hobbies or other leisure time activities? | 1 | 2 | 3 | 4 |
| 8. | Were you short of breath? | 1 | 2 | 3 | 4 |
| 9. | Have you had pain? | 1 | 2 | 3 | 4 |
| 10. | Did you need to rest? | 1 | 2 | 3 | 4 |

Please go on to the next page

11. Have you had trouble sleeping?

12. Have you felt weak?

15. Have you vomited?

13. Have you lacked appetite?

14. Have you felt nauseated?

16. Have you been constipated?

3

3

3

3

3

2

2

2

4

4

4

4

4

| During the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|
| 17. Have you had diarrhea? | 1 | 2 | 3 | 4 |
| 18. Were you tired? | 1 | 2 | 3 | 4 |
| 19. Did pain interfere with your daily activities? | 1 | 2 | 3 | 4 |
| 20. Have you had difficulty in concentrating on things,<br>like reading a newspaper or watching television? | 1 | 2 | 3 | 4 |
| 21. Did you feel tense? | 1 | 2 | 3 | 4 |
| 22. Did you worry? | 1 | 2 | 3 | 4 |
| 23. Did you feel irritable? | 1 | 2 | 3 | 4 |
| 24. Did you feel depressed? | 1 | 2 | 3 | 4 |
| 25. Have you had difficulty remembering things? | 1 | 2 | 3 | 4 |
| 26. Has your physical condition or medical treatment interfered with your <u>family</u> life? | 1 | 2 | 3 | 4 |
| 27. Has your physical condition or medical treatment<br>interfered with your <u>social</u> activities? | 1 | 2 | 3 | 4 |
| 28. Has your physical condition or medical treatment<br>caused you financial difficulties? | 1 | 2 | 3 | 4 |

#### For the following questions please circle the number between 1 and 7 that best applies to you

| 29. | How wo | uld you rate | e your over | all <u>health</u> dur | ing the past | week? | |
|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ver | y poor | | | | | | Excellent |
| 30 | Hanrina | uld von rat | a vour over | all quality of | life during | the nact wee | st-7 |
| 50. | 110W W0 | uiu you rau | e your over | an <u>quanty or</u> | me during | ine past wee | in.: |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ver | y poor | | | | | | Excellent |
| Sour | ce: (Aaı | ronson, 19 | 993) | | | | |

## APPENDIX D. PATIENT-REPORTED OUTCOMES: EQ-5D-5L QUESTIONNAIRE

| Under each heading, please tick the ONE box that best describes | your health TODAY. |
|---|---|
| MOBILITY | |
| I have no problems in walking about | |
| I have slight problems in walking about | |
| I have moderate problems in walking about | |
| I have severe problems in walking about | |
| I am unable to walk about | |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | |
| I have extreme pain or discomfort | |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | |

- · We would like to know how good or bad your health is TODAY.
- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- . Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =



# APPENDIX E. NATIONAL CANCER INSTITUTE (NCI) COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (CTCAE) VERSION 5.0

Currently active version of NCI CTCAE, Version 5.0:

https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm#ctc 50

## APPENDIX F. DYNAMIC INTERNATIONAL PROGNOSTIC SCORING SYSTEM (DIPSS)

#### **DIPSS Risk Score**

| | | Value | |
|---------------------------------|------|-------|------|
| Prognostic variable | 0 | 1 | 2 |
| Age, years | ≤ 65 | > 65 | |
| White blood cell count, x 109/L | ≤ 25 | > 25 | |
| Hemoglobin, g/dL | ≥ 10 | | < 10 |
| Peripheral blood blast, % | < 1 | ≥ 1 | |
| Constitutional symptoms, Y/N | N | Y | |

The risk category is obtained by adding up the values of each prognostic variable.

Risk categories are defined as low: 0; intermediate-1: 1 or 2; intermediate-2: 3 or 4; and high: 5 or 6.

Constitutional symptoms are defined as >10% weight loss in 6 months, night sweats, unexplained fever higher than 37.5°C.

Sources: (Passamonti, 2010).

## APPENDIX G. IWG-MRT: INTERNATIONAL WORKING GROUP-MYELOPROLIFERATIVE NEOPLASMS RESEARCH AND TREATMENT (IWG-MRT)

Proposed nomenclature by the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT)

de novo presenting disease

Primary myelofibrosis (PMF)

Myelofibrosis transformation from prior polycythemia vera

(PV) or essential thrombocythemia (ET)

Post PV myelofibrosis (post-PV MF)

Post ET myelofibrosis (post-ET MF)

Transformation to acute leukemia

Primary myelofibrosis in blast phase (PMF-BP)

Post PV/ET MF in blast phase

Source: (Mesa, 2007).

# APPENDIX H. 2016 WORLD HEALTH ORGANIZATION (WHO) DIAGNOSTIC CRITERIA FOR PRIMARY MYELOFIBROSIS (PMF)

2016 WHO diagnostic criteria for prePMF and overt PMF

| PrePMF <sup>a</sup> | Overt PMF <sup>b</sup> |
|---|---|
| Major criteria | |
| 1. Megakaryocytic proliferation and atypia, without reticulin fibrosis > grade 1*, accompanied by increased age-adjusted BM cellularity, granulocytic proliferation, and often decreased erythropoiesis | <ol> <li>Presence of megakaryocytic proliferation and atypia,<br/>accompanied by either reticulin and/or collagen fibrosis<br/>grades 2 or 3*</li> </ol> |
| 2. Not meeting the WHO criteria for BCR-ABL1 <sup>+</sup> CML, PV, ET, myelodysplastic syndromes, or other myeloid neoplasms | 2. Not meeting WHO criteria for ET, PV, BCR-ABL1 <sup>+</sup> CML, myelodysplastic syndromes, or other myeloid neoplasms |
| 3. Presence of JAK2, CALR, or MPL mutation or in the absence of these mutations, presence of another clonal marker <sup>c</sup> , or absence of minor reactive BM reticulin fibrosis <sup>d</sup> | 3. Presence of JAK2, CALR, or MPL mutation or in the absence of these mutations, presence of another clonal marker <sup>c</sup> , or absence of reactive myelofibrosis <sup>d</sup> |
| Minor criteria | |
| Presence of at least 1 of the following, confirmed in 2 consecutive determinations: | Presence of at least 1 of the following, confirmed in 2 consecutive determinations: |
| a. Anemia not attributed to a comorbid condition | a. Anemia not attributed to a comorbid condition |
| b. Leukocytosis ≥ 11 x 10°/L | b. Leukocytosis ≥ 11 x 10 <sup>9</sup> /L |
| c. Palpable splenomegaly | c. Palpable splenomegaly |
| d. LDH increased to above upper normal limit of institutional reference range | d. LDH increased to above upper normal limit of institutional reference range |
| | e. Leukoerythroblastosis |

<sup>\*</sup> More than 25% above mean normal predicted value.

<sup>&</sup>lt;sup>a</sup> Diagnosis of prePMF requires meeting all 3 major criteria, and at least 1 minor criterion.

<sup>&</sup>lt;sup>b</sup> Diagnosis of overt PMF requires meeting all 3 major criteria, and at least 1 minor criterion.

<sup>&</sup>lt;sup>c</sup> In the absence of any of the 3 major clonal mutations, the search for the most frequent accompanying mutations (eg, ASXL1, EZH2, TET2, IDH1/IDH2, SRSF2, SF3B1) are of help in determining the clonal nature of the disease.

d Minor (grade 1) reticulin fibrosis secondary to infection, autoimmune disorder or other chronic inflammatory conditions, hairy cell leukemia or other lymphoid neoplasm, metastatic malignancy, or toxic (chronic) myelopathies.

## Grading of myelofibrosis

## Myelofibrosis grading

| MF-0 | Scattered linear reticulin with no intersections (crossovers) corresponding to normal BM |
|---|---|
| MF-1 | Loose network of reticulin with many intersections, especially in perivascular areas |
| MF-2 | Diffuse and dense increase in reticulin with extensive intersections, occasionally with focal bundles of thick fibers mostly consistent with collagen, and/or focal osteosclerosis* |
| MF-3 | Diffuse and dense increase in reticulin with extensive intersections and coarse bundles of thick fibers consistent with collagen, usually associated with osteosclerosis* |

Semiquantitative grading of BM fibrosis (MF) with minor modifications concerning collagen and osteosclerosis. Fiber density should be assessed only in hematopoietic areas.

Source: (Arber, 2016).

<sup>\*</sup>In grades MF-2 or MF-3 an additional trichrome stain is recommended.

## APPENDIX I. PROPOSED CRITERIA FOR THE DIAGNOSIS OF POST-POLYCYTHEMIA VERA AND POST-ESSENTIAL THROMBOCYTHEMIA MYELOFIBROSIS

International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) recommended criteria for post-PV MF and post-ET MF

| Criteria for post-polycythemia vera myelofibrosis | Criteria for post-essential thrombocythemia myelofibrosis |
|---|---|
| Required criteria: | |
| 1. Documentation of a previous diagnosis of polycythemia vera as defined by the WHO criteria | 1. Documentation of a previous diagnosis of essential thrombocythemia as defined by the WHO criteria |
| 2. Bone marrow fibrosis grade 2–3 (on 0–3 scale) or grade 3–4 (on 0–4 scale) <sup>a</sup> | 2. Bone marrow fibrosis grade 2–3 (on 0–3 scale) <sup>3</sup> or grade 3–4 (on 0–4 scale) <sup>a</sup> |
| Additional criteria (two are required): | |
| 1. Anemia <sup>b</sup> or sustained loss of requirement of either phlebotomy (in absence of cytoreductive therapy) or cytoreductive treatment for erythrocytosis | 1. Anemia <sup>b</sup> and a $\geq$ 2 mgml-1 decrease from baseline hemoglobin level |
| 2. A leukoerythroblastic peripheral blood picture | 2. A leukoerythroblastic peripheral blood picture |
| 3. Increasing splenomegaly defined as either an increase in palpable splenomegaly of $\geq 5$ cm (distance of the tip of the spleen from the left costal margin) or the appearance of a newly palpable splenomegaly | 3. Increasing splenomegaly defined as either an increase in palpable splenomegaly of $\geq 5$ cm (distance of the tip of the spleen from the left costal margin) or the appearance of a newly palpable splenomegaly |
| 4. Development of $\geq 1$ of three constitutional symptoms: $> 10\%$ weight loss in 6 months, night sweats, unexplained fever ( $> 37.5$ °C) | 4. Increased LDH (above reference level) |
| | 5. Development of $\geq$ 1 of three constitutional symptoms: $>$ 10% weight loss in 6 months, night sweats, unexplained fever ( $>$ 37.5°C) |

<sup>&</sup>lt;sup>a</sup> Grade 2–3 according to the European classification: <sup>3</sup> diffuse, often coarse fiber network with no evidence of collagenization (negative trichrome stain) or diffuse, coarse fiber network with areas of collagenization (positive trichrome stain). Grade 3–4 according to the standard classification: <sup>4</sup> diffuse and dense increase in reticulin with extensive intersections, occasionally with only focal bundles of collagen and/or focal osteosclerosis or diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis.

<sup>&</sup>lt;sup>b</sup> Below the reference range for appropriate age, sex, gender and altitude considerations. Source: (Barosi, 2008).

#### APPENDIX J. ECOG PERFORMANCE STATUS SCALE

The ECOG Performance Status Scale is used to score a subject's quality of life through evaluation, by a health professional, of daily activities and how those activities are affected by the disease of the subject.

| Score | Description |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work. |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead |

Source: (Oken, 1982).

## APPENDIX K. ESTIMATION OF THE GLOMERULAR FILTRATION RATE BY THE MDRD FORMULA

#### **GFR** Estimation

GFR is estimated using the MDRD formula below:

GFR (mL/min/1.73 m<sup>2</sup>) = 175 x (Scr)<sup>-1.154</sup> x (age)<sup>-0.203</sup> x 1.212 (if African American) x 0.742 (if female)

Where Scr (standardized serum creatinine) = mg/dL; age = years

Source: (Levey, 2006).

## APPENDIX L. CLINICALLY RELEVANT P450 INDUCERS, INHIBITORS, SUBSTRATES, AND TRANSPORTER SUBSTRATES

A list of clinically relevant P450 inducers and inhibitors as well as substrates, and transporter substrates can be found in this appendix. This is not an exhaustive list. It is periodically updated at the following link:

https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm

#### Examples of clinical inducers for P450-mediated metabolisms

| Strong CYP3A inducers | Moderate CYP3A inducers |
|---|---|
| carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort | bosentan, efavirenz, etravirine, modafinil |

#### Examples of clinical inhibitors for P450-mediated metabolisms

| Strong CYP3A inhibitors | Dual CYP2C19 and CYP3A4 inhibitors |
|---|---|
| boceprevir, cobicistat, conivaptan, danoprevir and ritonavir, elvitegravir and ritonavir, grapefruit juice, indinavir and ritonavir, itraconazole, ketoconazole, lopinavir and ritonavir, paritaprevir and ritonavir and (ombitasvir and/or dasabuvir), posaconazole, ritonavir, saquinavir and ritonavir, telaprevir, tipranavir and ritonavir, troleandomycin, voriconazole | fluconazole, fluvoxamine |
| clarithromycin, diltiazem, idelalisib, nefazodone, nelfinavir | |

## Examples of clinical substrates for P450-mediated metabolism

| | Sensitive substrates | Substrates with narrow therapeutic range |
|---|---|---|
| CYP2C19 | S-mephenytoin, omeprazole | S-mephenytoin |
| CYP2D6 | atomoxetine, dextromethorphan, eliglustat, nebivolol, nortriptyline, perphenazine, tolterodine, venlafaxine | desipramine |
| CYP3A | alfentanil, avanafil, buspirone, conivaptan, darifenacin, darunavir, ebastine, everolimus, ibrutinib, lomitapide, lovastatin, midazolam, naloxegol, nisoldipine, saquinavir, simvastatin, sirolimus, tacrolimus, tipranavir, triazolam, vardenafil | Alfentanil, cyclosporin, diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus |
| | budesonide, dasatinib, dronedarone, eletriptan, eplerenone, felodipine, indinavir, lurasidone, maraviroc, quetiapine, sildenafil, ticagrelor, tolvaptan | |

## **Examples of clinical substrates for transporters**

| Transporter | Substrate |
|---|---|
| P-gp | dabigatran, digoxin, fexofenadine |
| BCRP | rosuvastatin, sulfasalazine |
| OATP1B1<br>OATP1B3 | asunaprevir, atorvastatin, bosentan, cerivastatin, danoprevir, docetaxel, fexofenadine, glyburide, nateglinide, paclitaxel, pitavastatin, pravastatin, repaglinide, rosuvastatin, simvastatin acid |
| MATE1,<br>MATE-2K,<br>OCT2 | dofetilide, metformin |

## APPENDIX M. NEW YORK HEART ASSOCIATION CLASSIFICATION FOR CONGESTIVE HEART FAILURE

#### **Classification of Heart Failure**

| Class | Functional Capacity |
|---|---|
| Class I | Subjects with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain. |
| Class II | Subjects with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain. |
| Class III | Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. |
| Class IV | Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased. |

Source: AHA Medical/Scientific Statement (1994).



# APPENDIX O. REVISED RESPONSE CRITERIA FOR MYELOFIBROSIS: INTERNATIONAL WORKING GROUP-MYELOPROLIFERATIVE NEOPLASMS RESEARCH AND TREATMENT (IWG-MRT) AND EUROPEAN LEUKEMIANET (ELN) CONSENSUS REPORT (2013)

| Response<br>Categories | Required Criteria (For All Response Categories, Benefit Must Last For ≥ 12 Weeks To Qualify As A Response) |
|---|---|
| CR | Bone marrow:* Age-adjusted normocellularity; $< 5\%$ blasts; $\le$ grade 1 MF $\dagger$ and Peripheral blood: Hemoglobin $\ge 100$ g/L and $<$ UNL; neutrophil count $\ge 1$ x $10^9$ /L and $<$ UNL; Platelet count $\ge 100$ x $10^9$ /L and $<$ UNL; $< 2\%$ immature myeloid cells $\ddagger$ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH |
| PR | Peripheral blood: Hemoglobin $\geq 100$ g/L and $<$ UNL; neutrophil count $\geq 1$ x $10^9$ /L and $<$ UNL; platelet count $\geq 100$ x $10^9$ /L and $<$ UNL; $<$ 2% immature myeloid cells‡ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH or Bone marrow:* Age-adjusted normocellularity; $<$ 5% blasts; $\leq$ grade 1 MF†, and peripheral blood: Hemoglobin $\geq 85$ but $<$ 100 g/L and $<$ UNL; neutrophil count $\geq 1$ x $10^9$ /L and $<$ UNL; platelet count $\geq 50$ , but $<$ 100 x $10^9$ /L and $<$ UNL; $<$ 2% immature myeloid cells‡ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH |
| Clinical improvement (CI) | The achievement of anemia, spleen or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia§ |
| Anemia<br>response | Transfusion-independent patients: $a \ge 20$ g/L increase in hemoglobin level Transfusion-dependent patients: becoming transfusion-independent { |
| Spleen response | A baseline splenomegaly that is palpable at 5-10 cm, below the LCM, becomes not palpable** or A baseline splenomegaly that is palpable at $> 10$ cm, below the LCM, decreases by $\geq 50\%$ ** A baseline splenomegaly that is palpable at $< 5$ cm, below the LCM, is not eligible for spleen response A spleen response requires confirmation by MRI or computed tomography showing $\geq 35\%$ spleen volume reduction |
| Symptoms<br>response# | $A \geq 50\%$ reduction in the MPN-SAF TSS†† |
| Progressive<br>disease‡‡ | Appearance of a new splenomegaly that is palpable at least 5 cm below the LCM or A $\geq$ 100% increase in palpable distance, below LCM, for baseline splenomegaly of 5-10 cm or A 50% increase in palpable distance, below LCM, for baseline splenomegaly of $>$ 10 cm or Leukemic transformation confirmed by a bone marrow blast count of $\geq$ 20% or A peripheral blood blast content of $\geq$ 20% associated with an absolute blast count of $\geq$ 1 x 10(9)/L that lasts for at least 2 weeks |
| Stable disease | Belonging to none of the above-listed response categories |
| Relapse | No longer meeting criteria for at least CI after achieving CR, PR, or CI, or Loss of anemia response persisting for at least 1 month or Loss of spleen response persisting for at least 1 month |

EMH, extramedullary hematopoiesis (no evidence of EMH implies the absence of pathology- or imaging study-proven non-hepatosplenic EMH); LCM, left costal margin; UNL, upper normal limit.

- \* Baseline and posttreatment bone marrow slides are to be interpreted at one sitting by a central review process. Cytogenetic and molecular responses are not required for CR assignment.
- † Grading of MF is according to the European classification Thiele et al. European consensus on grading bone marrow fibrosis and assessment of cellularity. Haematologica. 2005;90:1128.
- ‡ Immature myeloid cells constitute blasts + promyelocytes + myelocytes + metamyelocytes + nucleated red blood cells. In splenectomized patients, < 5% immature myeloid cells is allowed.
- § Increase in severity of anemia constitutes the occurrence of new transfusion dependency or a  $\geq$  20 g/L decrease in hemoglobin level from pretreatment baseline that lasts for at least 12 weeks. Increase in severity of thrombocytopenia or neutropenia is defined as a 2-grade decline, from pretreatment baseline, in platelet count or absolute neutrophil count, according to the CTCAE version 4.0. In addition, assignment to CI requires a minimum platelet count of  $\geq$  25 000 x 10(9)/L and absolute neutrophil count of  $\geq$  0.5 x 10(9)/L.
- Applicable only to patients with baseline hemoglobin of < 100 g/L. In patients not meeting the strict criteria for transfusion dependency at the time of randomization, but have received transfusions within the previous month, the pretransfusion hemoglobin level should be used as the baseline.
- { Transfusion dependency before randomization is defined as transfusions of at least 6 units of packed red blood cells (PRBC), in the 12 weeks prior to study randomization, for a hemoglobin level of < 85 g/L, in the absence of bleeding or treatment-induced anemia. In addition, the most recent transfusion episode must have occurred in the 28 days prior to randomization. Response in transfusion-dependent patients requires absence of any PRBC transfusions during any consecutive "rolling" 12-week interval during the treatment phase, capped by a hemoglobin level of  $\ge 85$  g/L.
- # In splenectomized patients, palpable hepatomegaly is substituted with the same measurement strategy.
- \*\*Spleen or liver responses must be confirmed by imaging studies where  $a \ge 35\%$  reduction in spleen volume, as assessed by MRI or CT, is required. Furthermore,  $a \ge 35\%$  volume reduction in the spleen or liver, by MRI or CT, constitutes a response regardless of what is reported with physical examination.
- †† Symptoms are evaluated by the MPN-SAF TSS.17 The MPN-SAF TSS is assessed by the patients themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). Symptoms response requires ≥ 50% reduction in the MPN-SAF TSS.
- ‡‡ Progressive disease assignment for splenomegaly requires confirmation by MRI or computed tomography showing a ≥ 25% increase in spleen volume from baseline. Baseline values for both physical examination and imaging studies refer to pretreatment baseline and not to posttreatment measurements.

Source: (Tefferi, 2013).

## APPENDIX P. MINI-MENTAL STATE EXAMINATION-2

| MMQE. | Date of examination | | Б | aminer | | |
|---|---|---|---|---|---|---|
| MINIOF | Name | | | Age | Sex | |
| standard Version | Years of school com | pleted | Purpose of exi | am | | |
| Blue Form | Assessment of level | | | | | |
| | Alert/ | Drowsy | Stuporous | Comatose/ | | |
| | Responsive | | | Unresponsive | | |
| in parentheses. Admi- | in boldface type should be ro<br>nistration should be conduct<br>he response is incorrect or 1<br>Now I'd like to ask y | ed privately<br>if the respon | and in the examin<br>se is correct. Begir | ee's primary languag<br>1 by introducing the 1 | <ol> <li>Unless other</li> </ol> | appear<br>erwise |
| | | | RESP | PONSE | SCC | |
| REGISTRATION | | | | | (circle | e one) |
| MLK [pause], ŠENSII<br>Repeat up to 3 times,<br>MILI<br>SEN | SIBLE | se]. Now re | em back after is | back to me. | _ 0<br>_ 0 | 1 1 1 |
| | ORE<br>ds in mind. I am going to a | sk vou to s | av them again in | a few minutes. | _ 0 | |
| | | on you to o | ay alom again in | a 1011 11111111111111111111111111111111 | | |
| DRIENTATION TO | | | | | | |
| /hat day is today? V | | | | | 0 | 4 |
| year | | - | | | 0 | 1 |
| | son? | _ | | | _ 0 | 1 |
| | of the year? | - | | | _ 0 | 1 |
| date | | _ | | | _ 0 | 1 |
| DRIENTATION TO | D PLACE* | | | | | |
| here are we now? | | | | | | |
| state | e (or province)? | _ | | | _ 0 | 1 |
| | nty (or city/town)? | | | | _ 0 | 1 |
| city/ | <b>ftown</b> (or part of city/neighbo | rhood)? | | | _ 0 | 1 |
| | ding (name or type)? | - | | | 0 | 1 |
| | r of the building<br>m number or address)? | | | | _ 0 | 1 |
| | that are appropriate for the setting | and increasin | gly precise may be su | bstituted and noted. | | |
| RECALL. | | | | | | |
| | ee words I asked you to re | member? [[ | Oo not offer any hir | nts.] | | |
| MIL | | | , | | 0 | 1 |
| | NSIBLE | · · | | | . 0 | 1 |
| | ORE | - | | | . 0 | 1 |
| | If administering the MMSE-2:S<br>the space provided at the top o | f page 2 and | continue with admi | nistration. total rav | | . points) |
| | orida Ave. • Lutz, FL 33549 | | | | | |
| (MSE copyright © 1975, 1998, 2 | 2001 and MMSE-2 copyright © 2010 by Mi | niMental, LLC. All I<br>ted in blue and bur | rights reserved. Published 2<br>mundy ink on white paper. At | 2001, 2010 by PAR. May not be<br>ny other version is unauthorized | reproducéd in whole | e or in part |
| ny form or by any means without<br>8765432 | t written permission of 1945. This form is prin | Reorder #F | | | | in the U.S. |

| | MMSE-2:B total raw scor | | | |
|---|---|---|---|---|
| ATTENTION AND CALC | III ATION [Serial 7e] | | | e. points) |
| | The state of the s | subtracting 7 from each answer until I tell y | | positio |
| What is 100 take away 7? | [93] | | 0 | 1 |
| f needed, say: Keep going. | [86] | | 1000 | 1 |
| f needed, say: Keep going. | [79] | | | 1 |
| f needed, say: Keep going. | [72] | | | 1 |
| f needed, say: Keep going. | [65] | | . 0 | 1 |
| core I point for each correct ar<br>even if the previous answer was | | ered correct if it is 7 less than the previous answe | er, | |
| NAMING | | | | |
| What is this? [Point to eye.] | | | 0 | 1 |
| What is this? [Point to ear.] | | | 0 | 1 |
| REPETITION | | | | |
| | | ady? IT IS A LOVELY, SUNNY DAY BUT TO<br>acord response verbatim. Repeat up to one ti | | |
| IT IS A LOVELY, SUNNY D. | AY BUT TOO WARM. | Market and the second s | | 1 |
| | at these pictures and po | o something. [Show examinee the geometric | ; | |
| and their point to the triangl | | | | |
| | Correct response | Observed response | | |
| | 0 | | 0 | 1 |
| | Ш | | 0 | 1 |
| | Δ | | 0 | 1 |
| READING | | | | |
| Show examinee the word stir | nulus page.] Please do v | what this says to do. | | |
| CLOSE YOU | JR EYES | | _ 0 | 1 |
| WRITING | | | | |
| Please write a sentence. [/f e | xaminee does not respo | e and provide a pen or pencil.]<br>nd, say: Write about where you live.]<br>ns a subject and a verb. Ignore errors in gramman | 0 | 1 |
| DRAWING | | | | |
| Display the intersecting penta | | rn and provide a pen or pencil.] Please copy<br>sided figures that intersect to form a 4-sided figur | | 1 |
| | | MMS<br>total ray | SE-2:SV<br>w score | |

Confidential and Proprietary

2 WARNING! PHOTOCOPYING OR DUPLICATION OF THIS FORM WITHOUT PERMISSION IS A VIOLATION OF COPYRIGHT LAWS.







## **CLOSE YOUR EYES**





## Celgene Signing Page

This is a representation of an electronic record that was signed electronically in Livelink. This page is the manifestation of the electronic signature(s) used in compliance with the organizations electronic signature policies and procedures.

EDMS Doc. Number: 25557463 - 23009667